| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE: |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 1 OF 33 |
| Active | Informed Vital Core, Pulse Rate Clinical Study Protocol | IVC-400-006 | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| March 31, 2023 | Chris Joslin | Mark Whitehouse | |

## Informed Vital Core Pulse Rate Clinical Study Protocol

IVC-400-006 Rev. 1

Mindset Medical, LLC

| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE: |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 2 OF 33 |
| Active | Informed Vital Core, Pulse Rate Clinical Study Protocol | IVC-400-006 | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| March 31, 2023 | Chris Joslin | Mark Whitehouse | |

## A Multi-Center Prospective Open Label Study of a Web-based Application for Pulse Rate in Adult Patients

Original date: March 31, 2023

Principal Investigator: Daniel Lubelski, M.D.

| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE: |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 3 OF 33 |
| Active | Informed Vital Core, Pulse Rate Clinical Study Protocol | IVC-400-006 | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| March 31, 2023 | Chris Joslin | Mark Whitehouse | |

#### PROTOCOL APPROVAL FORM

Protocol Number: IVC-400-006

Study Title: A Multi-Center Prospective Open Label Study of a Web-based Application for Pulse Rate in Adult Patients

Version Number: Version 1.0 dated March 31, 2023.

This study protocol was subjected to critical review. The information it contains is consistent with Mindset Medical, LLC's current knowledge of the risks and benefits of the investigational technology, as well as with the moral, ethical, and scientific principles governing clinical research as set out in the *Declaration of Helsinki*, as amended in 2000 and clarified in 2004, and the guidelines on *Good Clinical Practice*.

The study protocol has been reviewed and approved by the following:

| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE: |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 4 OF 33 |
| Active | Informed Vital Core, Pulse Rate Clinical Study Protocol | IVC-400-006 | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| March 31, 2023 | Chris Joslin | Mark Whitehouse | |

| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE: |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 5 OF 33 |
| Active | Informed Vital Core, Pulse Rate Clinical Study Protocol | IVC-400-006 | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| March 31, 2023 | Chris Joslin | Mark Whitehouse | |

#### **Investigator's Agreement**

I have read the protocol version 1.0 dated March 31, 2023 and agree to conduct the study as outlined.

The information contained in this document and all information provided to me related to this protocol are the confidential and proprietary information of Mindset Medical (Sponsor), and except as may be required by federal, state, or local laws or regulations, may not be disclosed to others without prior permission of Sponsor. However, the Principal Investigator at each site may disclose such information to supervised individuals working on the study, provided such individuals agree to be bound to maintain the confidentiality of such information.

I agree to abide by the above Confidentiality Statement.

I agree to conduct the study according to this protocol. Any changes in procedure will only be made if necessary to protect study subjects' safety, rights, or welfare.

I agree to comply with the current *International Conference on Harmonization Tripartite Guideline on Good Clinical Practice* and applicable U.S. FDA regulations including 21 CFR 50, 54, and 56.

I agree to conduct the study in person or to supervise the study.

I agree to ensure that all individuals who assist me in the conduct of the study have access to the study protocol and any amendments and am aware of their obligations under this protocol.

| Printed Name of Investigator |
|------------------------------|
| Signature of Investigator |
| Date |

| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE: |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 6 OF 33 |
| Active | Informed Vital Core, Pulse Rate Clinical Study Protocol | IVC-400-006 | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| March 31, 2023 | Chris Joslin | Mark Whitehouse | |

## **Summary of Changes**

| Original | Amendment Change | Reason for Change |
|------------------|------------------|-------------------|
| Original release | N/A | N/A |

| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE: |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 7 OF 33 |
| Active | Informed Vital Core, Pulse Rate Clinical Study Protocol | IVC-400-006 | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| March 31, 2023 | Chris Joslin | Mark Whitehouse | |

## Contents

| PROTOCOL SYNOPSIS | 10 |
|--------------------------------------|----|
| STUDY OBJECTIVES | 12 |
| STUDY HYPOTHESIS | 13 |
| STUDY ENDPOINTS | 13 |
| Primary Endpoint | |
| BACKGROUND | 13 |
| STUDY DESIGN | 15 |
| NUMBER OF SITES | 15 |
| NUMBER OF SUBJECTS | 16 |
| STUDY DURATION | 16 |
| SCHEDULE OF ASSESSMENTS | 17 |
| ELIGIBILITY | 18 |
| Inclusion CriteriaExclusion Criteria | |
| SUBJECT IDENTIFICATION | 18 |
| STUDY EXECUTION | 19 |
| Enrollment | |
| Pre-intervention screening | |

| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE: |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 8 OF 33 |
| Active | Informed Vital Core, Pulse Rate Clinical Study Protocol | IVC-400-006 | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | · |
| March 31, 2023 | Chris Joslin | Mark Whitehouse | |

| ADVERSE EVENTS | 21 |
|---|---|
| Definitions | 21 |
| Required Reporting Timelines per Regulatory Guidance | |
| WITHDRAWAL AND LOST TO FOLLOW UP | |
| STATISTICAL METHODS | 23 |
| Sample Size | |
| Statistical Analysis | 23 |
| Analysis of the primary endpoint | |
| DATA MANAGEMENT | 24 |
| ELECTRONIC CASE REPORT FORMS (ECRFS) AND SOURCE DOCUMENTATION | 24 |
| Access to Source Data and Monitoring | 24 |
| Archiving Study Records | 25 |
| ETHICAL, LEGAL, AND ADMINISTRATIVE ASPECTS | 26 |
| Sponsor Responsibilities | |
| Investigator Responsibilities | |
| GOOD CLINICAL PRACTICE | 26 |
| PROTOCOL APPROVAL AND AMENDMENT | |
| Protocol Approval and Amendment | |
| TERMINATION OF THE STUDY | |
| TERMINATION OF THE STUDY | |
| TERMINATION OF THE STUDY CONFIDENTIALITY PUBLICATION SITE TRAINING | |
| TERMINATION OF THE STUDY CONFIDENTIALITY PUBLICATION SITE TRAINING REQUIRED REPORTS. | |
| TERMINATION OF THE STUDY CONFIDENTIALITY PUBLICATION SITE TRAINING | |
| TERMINATION OF THE STUDY CONFIDENTIALITY PUBLICATION SITE TRAINING REQUIRED REPORTS. | |

| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE: |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 9 OF 33 |
| Active | Informed Vital Core, Pulse Rate Clinical Study Protocol | IVC-400-006 | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| March 31, 2023 | Chris Joslin | Mark Whitehouse | |

| TABLE OF COMMON ACRONYMS | 32 |
|--------------------------|----|
| REFERENCES | 33 |

| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE: |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 10 OF 33 |
| Active | Informed Vital Core, Pulse Rate Clinical Study Protocol | IVC-400-006 | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| March 31, 2023 | Chris Joslin | Mark Whitehouse | |

## **Protocol Synopsis**



| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE: |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 11 OF 33 |
| Active | Informed Vital Core, Pulse Rate Clinical Study Protocol | IVC-400-006 | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| March 31, 2023 | Chris Joslin | Mark Whitehouse | |

| Study hypothesis | PR will be collected simultaneously with the IVC App and reference device |
|---|---|
| Intervention model | Single Group Assignment |
| Masking | None (open label) |
| Investigational device | Informed Vital Core Application (IVC App) by Mindset Medical, LLC |
| Reference device | |
| Primary objective | The primary objective of the study is to establish that pulse rate (PR) measured with the IVC App are accurate with the reference |
| Primary endpoint | |
| Study design | The study will recruit subjects from clinics, hospitals, and the general public. |

| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE: |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 12 OF 33 |
| Active | Informed Vital Core, Pulse Rate Clinical Study Protocol | IVC-400-006 | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| March 31, 2023 | Chris Joslin | Mark Whitehouse | |

| Patient population | Inclusion Criteria |
|---|---|
| | Subjects 22 -85 years of age |
| | Subjects willing to sign the Informed Consent Form and comply with the protocol |
| | Exclusion Criteria |
| | Subjects required to wear mask or bandage that obstructs forehead, cheeks, or chin |
| | <ul> <li>Refusal to remove makeup, sunscreen, lotion, clothing, or items obstructing the face for the duration of measurement</li> </ul> |
| | <ul> <li>Presence of facial tattoos, large birthmarks, or other skin alterations (scars, hemangiomas, vitiligo) on upper cheeks (cheekbone) or forehead of the subject</li> </ul> |
| | Condition that does not allow the subject to remain still for 60 seconds at a time |
| | Subjects with cardiac arrhythmia |
| | Any known medical condition which may result in an inaccurate measurement using the reference device |
| | Subjects with the inability to complete an ECG |
| Sample size | |
| Study visits | Screening/Baseline |
| Study duration | One day |

This multi-center prospective open label study is designed to evaluate the accuracy of Informed Vital Core Application (IVC App), a web-based application designed for measurements of vital signs including pulse rate. It is hypothesized that the accuracy of the IVC App is non-inferior to the FDA-cleared/approved vital sign monitoring device (reference device).

## **Study Objectives**

| The primary objective of the study is to establish that pulse rate (PR) measured with the IVC App are accurate |
|---|
| measured with the reference . |

| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE: |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 13 OF 33 |
| Active | Informed Vital Core, Pulse Rate Clinical Study Protocol | IVC-400-006 | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| March 31, 2023 | Chris Joslin | Mark Whitehouse | |

## **Study Hypothesis**

## **Study Endpoints**

#### **Primary Endpoint**

## Background

Vital sign measurement is a core process in delivering healthcare. Pulse rate is one of the most frequently measured vital signs in inpatient as well as outpatient encounters. Currently, pulse rate may have to be measured several times in a day.



| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE: |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 14 OF 33 |
| Active | Informed Vital Core, Pulse Rate Clinical Study Protocol | IVC-400-006 | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| March 31, 2023 | Chris Joslin | Mark Whitehouse | |



Mindset Medical will conduct a clinical study to evaluate the accuracy of measurement for pulse rate using the IVC App, compared to appropriate reference devices. The study will recruit subjects from clinics, hospitals, and the general public.

| INFORMED MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE: |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 15 OF 33 |
| Active | Informed Vital Core, Pulse Rate Clinical Study Protocol | IVC-400-006 | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| March 31, 2023 | Chris Joslin | Mark Whitehouse | |

| Study Design |
|---|
| This is a multi-center prospective open label study where the same subjects are assigned the IVC Application and the |
| The study will recruit subjects from clinics, hospitals, and the general public. |
| All subjects will be called to beyo facial accomment and undersative DD measurements using the IVC Ann |
| All subjects will be asked to have facial assessment conducted and undergo two PR measurements using the IVC App. . |
| The PR obtained by the IVC App will be compared to the HR obtained by the |

Subjects will visit the clinic only once for the vital signs assessments unless a technical fallback session is required.

#### **Number of Sites**

The study will be conducted in up to ten (10) investigational sites in the United States. Enrollment will be competitive and each site will not enroll more than 25% of the total patient population without the written consent of the sponsor.

| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE: |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 16 OF 33 |
| Active | Informed Vital Core, Pulse Rate Clinical Study Protocol | IVC-400-006 | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| March 31, 2023 | Chris Joslin | Mark Whitehouse | |

## Number of Subjects

## **Study Duration**

Study assessment is one day.

| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE: |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 17 OF 33 |
| Active | Informed Vital Core, Pulse Rate Clinical Study Protocol | IVC-400-006 | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| March 31, 2023 | Chris Joslin | Mark Whitehouse | |

## Schedule of Assessments

Table 2- Schedule of Assessments

| | Screening /Baseline |
|------------------------------------|---------------------|
| | Day 1 |
| Study Visit/Day | Visit 1 |
| Informed Consent | X |
| Eligibility | X |
| Demographics | X |
| Fitzpatrick Scale Assignment** | X |
| Medical History | X |
| Concomitant Medication | X |
| Adverse Event Form (If applicable) | X |
| Pulse Rate (IVC)* | X |

| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE: |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 18 OF 33 |
| Active | Informed Vital Core, Pulse Rate Clinical Study Protocol | IVC-400-006 | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| March 31, 2023 | Chris Joslin | Mark Whitehouse | |

#### Eligibility

#### **Inclusion Criteria**

- Subjects 22 85 years of age
- Subjects willing to sign the Informed Consent Form and comply with the protocol

#### **Exclusion Criteria**

- Subjects required to wear mask or bandage that obstructs forehead, cheeks, or chin
- Refusal to remove makeup, sunscreen, lotion, clothing, or items obstructing the face for the duration of measurement
- Presence of facial tattoos, large birthmarks, or other skin alterations (scars, hemangiomas, vitiligo) on upper cheeks (cheekbone) or forehead of the subject
- Condition that does not allow the subject to remain still for 60 seconds at a time
- Subjects with cardiac arrhythmia
- Any known medical condition which may result in an inaccurate measurement using the reference device
- Subjects with the inability to complete an ECG

#### **Subject Identification**

Subjects will be enrolled per the inclusion and exclusion criteria. Written informed consent, including Health Insurance Portability and Accountability Act (HIPAA) authorization, must be obtained prior to initiation of any study-specific investigative procedures. Eligible subjects will be enrolled and given a 6-digit identification code that consists of the three-digit site code, followed by a three-digit subject ID beginning with 001 and assigned sequentially (e.g., 301 001; site 301 and the first subject screened 001).

| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE: |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 19 OF 33 |
| Active | Informed Vital Core, Pulse Rate Clinical Study Protocol | IVC-400-006 | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| March 31, 2023 | Chris Joslin | Mark Whitehouse | |

### **Study Execution**

#### Enrollment

Subjects that meet the protocol qualifications and provide written informed consent shall be offered enrollment in the study. Concomitant study enrollment may be allowed with approval of the Sponsor. Study subjects may be enrolled in this study only once. A subject will be considered enrolled when the subject has signed the Informed Consent Form (ICF).

#### Pre-intervention screening

#### **Review of Eligibility Criteria**

Review the list of inclusion and exclusion criteria to ensure the subject is eligible to participate.

#### **Informed Consent**

Prior to conducting any study-specific tests or procedures required in this protocol, the Investigator or designee will obtain informed consent in writing from all subjects prior to any screening or study procedures. The Investigator will follow a standard process for obtaining consent that complies with all applicable regulatory requirements.

If the ICF is amended during the study, the investigator must follow all applicable regulatory requirements pertaining to approval of the amended ICF by the IEC/IRB and use of the amended form. Ongoing subjects will be required to re-confirm consent by signing the amended form.

The original and any amended signed and dated ICFs must be retained at the study site, and a copy of the signed and dated ICFs must be given to the subject. During the study, the subject will be informed if information becomes available that may be relevant to the subject's willingness to participate in the study.

| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE: |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 20 OF 33 |
| Active | Informed Vital Core, Pulse Rate Clinical Study Protocol | IVC-400-006 | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| March 31, 2023 | Chris Joslin | Mark Whitehouse | |

The subject will be informed of procedures to protect subject privacy. Under U.S. federal law (the Privacy Rule) any protected health information (PHI) that is created or obtained during this study cannot be used or disclosed without permission. Informed consent on data processing will be obtained in writing directly from the subject before recording of any data. Authorization to use and disclose PHI will be obtained in writing directly from the subject before recording of any data. Recorded data will be pseudonymized before transferring to authorized individuals. The investigator will maintain source documents that link unique subject numbers with subject names.

#### **Study Procedure**

- Review the subject's medical history and concomitant medications and document on the appropriate Electronic Case Report Form (eCRF).
- Assign the Fitzpatrick Scale Category. Fitzpatrick category assignment must be completed by an Investigator.
- Record the subject's demographics on the appropriate eCRF.
- Record any adverse events, protocol deviations, device failures.
- Complete subject disposition eCRF.

| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE: |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 21 OF 33 |
| Active | Informed Vital Core, Pulse Rate Clinical Study Protocol | IVC-400-006 | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| March 31, 2023 | Chris Joslin | Mark Whitehouse | |

#### **Adverse Events**

#### **Definitions**

An **Adverse Event (AE)** is any untoward event that occurs after device implantation, any condition that increases in severity or frequency after device implantation, or any medical condition present at or before implantation that worsens after device implantation. All adverse events should be reported whether or not their occurrence has a causal relationship with the administration of the study material.

A **Serious Adverse Event (SAE)** is defined as any experience that:

- Is fatal or life-threatening
- Is permanently incapacitating or disabling
- Requires or prolongs in-patient hospitalization
- Results in a congenital anomaly or birth defect
- Results in permanent disability or incapacity
- Necessitates medical or surgical intervention to preclude a permanent disability or incapacity

Adverse events are not anticipated in this clinical study, since the study involves collection of pulse rate data using a remote software application and heart rate using an ECG device for a short period of time at the clinical study sites.

An **Unanticipated Adverse Device Effect (UADE)** is "any serious" adverse effect on health or safety or any life-threatening problem or death caused by, or associated with a device, if that effect, problem, or death was not previously identified in any nature, severity, or degree of incidence in the investigational plan or any other unanticipated serious problem associated with a device that relates to the rights, safety, and welfare of subjects.

| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE: |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 22 OF 33 |
| Active | Informed Vital Core, Pulse Rate Clinical Study Protocol | IVC-400-006 | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| March 31, 2023 | Chris Joslin | Mark Whitehouse | |

A record of each AE, including details of the nature, onset, duration, severity, relationship to the device will be recorded. AEs, should they occur, will be summarized and presented at each annual renewal for all subjects participating in the study. SAEs and UADEs should be reported to the FDA under the MDR reporting requirements and to the manufacturer.

#### Required Reporting Timelines per Regulatory Guidance

Required reporting time limit for the Sponsor is the number of days between the company's first knowledge of a reportable event (i.e., the receipt of information by any employee of the company) and the date the Food and Drug Administration (FDA) must be notified. Day one begins the day after the company receives information which reasonably suggests that a reportable event has occurred. Device related death, serious injury, or malfunction must be reported to FDA within 30 calendar days (no allowances are made for weekends or holidays).

However, if the event necessitates a correction or removal action, to prevent an unreasonable risk of substantial harm to the public health, then a report must be submitted within five (5) workdays, notwithstanding days including Saturdays, Sundays, and scheduled federal holidays.

#### Withdrawal and Lost to Follow Up

Subjects have the right to withdraw from the study at any time for any reason. The Investigator, acting in the subject's best interests, also has the right to withdraw subjects from the study. Since this study is a one-time assessment, early withdrawal is unlikely. However, it is possible for a subject withdrawal after signing consent and prior to study procedures. In all cases, the reason(s) for withdrawal must be recorded on the eCRF.

While adverse events are not anticipated in this clinical study, if the reason for removal of a subject from the study is an adverse event, the event will be recorded on the appropriate eCRF(s) and will be reported to Mindset Medical per the AE reporting guidelines (Required Reporting Timelines per Regulatory Guidance). All efforts will be made to follow the subject until the condition resolves, or the Investigator determines that the subject's health has returned to an acceptable state.

| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE: |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 23 OF 33 |
| Active | Informed Vital Core, Pulse Rate Clinical Study Protocol | IVC-400-006 | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| March 31, 2023 | Chris Joslin | Mark Whitehouse | |

#### Statistical Methods

#### Sample Size

#### **Inclusion of Incompetent Subjects**

Subjects who lack the capacity to provide written informed consent shall not be enrolled in this study.

#### **Statistical Analysis**

Detailed methodology for descriptive and inferential statistical analyses of the data collected in this study will be documented in the Statistical Analysis Plan (SAP). Analysis populations will be defined in the SAP and any methodology to be used for missing data. The SAP will be prepared and agreed upon by signature and date by the Sponsor prior to database lock. In addition to the SAP, other graphical representations of the results may be produced after review of the data (post hoc). Any major modifications of the definition of the endpoints or analysis will be reflected in a protocol amendment.

The SAP will define how missing data will be handled, where applicable, including the use of imputation or sensitivity analyses.

#### Analysis of the primary endpoint

The Intent-to-Capture (ITC) population will be defined as all consented subjects who passed screening and completed at least one data collection session without withdrawing.

The Per Protocol analysis group for the primary endpoint will consist of subjects from whom PR measurements from the IVC App and HR from the lateral ways were collected during the same window.

| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE: |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 24 OF 33 |
| Active | Informed Vital Core, Pulse Rate Clinical Study Protocol | IVC-400-006 | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| March 31, 2023 | Chris Joslin | Mark Whitehouse | |

The reference device Rhythm Analysis will be performed on the ECG rhythm strip using the procedure described in the Rhythm Analysis

D 1 14

#### Data Management

Procedure IVC-400-006i.

Data will be reviewed throughout the study to identify any missing data, errors in data entry, or inconsistencies in the data provided. A query process will be used to resolve any discrepancies identified during the data review process and follow a Data Management Plan (DMP) that will be prepared and agreed upon by signature and date by the Sponsor prior to database lock.

#### Electronic Case Report Forms (eCRFs) and Source Documentation

All data obtained during the study should be entered on the eCRFs promptly. All source documents from which eCRF entries are derived should be placed in the subject's medical records. The eCRFs for each subject may be checked against source documents at the study site by the clinical site monitor.

#### Access to Source Data and Monitoring

During the course of the study, a representative of the Sponsor or a designated representative, i.e., a Clinical Research Associate (CRA) or monitor, may make site visits as frequently as necessary to review protocol compliance, compare eCRFs and individual subjects' medical records, assess clinical supply inventory as appropriate, and ensure that the study is being conducted in accordance with pertinent regulatory requirements. eCRF entries will be verified with source documentation. The review of medical records will be performed in a manner to ensure that subject confidentiality is maintained.

| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE: |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 25 OF 33 |
| Active | Informed Vital Core, Pulse Rate Clinical Study Protocol | IVC-400-006 | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| March 31, 2023 | Chris Joslin | Mark Whitehouse | |

It is the Investigator's obligation to ensure that documentation of all relevant data such as medical history, concomitant diseases, date of study enrollment, visit dates, results of examinations, administrations of medication(s), and AEs are correctly entered in the subject's file.

Checking of the eCRFs for completeness and clarity, and cross-checking with source documents in the presence of the Investigator or designee, will be required to monitor the progress of the study. Moreover, regulatory authorities, IRB/REB, and/or the Sponsor's Clinical Quality Assurance group, or designee, may wish to carry out such source data checks and/or on-site audit inspections. Direct access to source data will be required for these inspections and audits; they will be carried out giving due consideration to data protection and medical confidentiality. The Investigator agrees to give the auditor access to all relevant documents for review. The same procedure applies in the case of an inspection by the regulatory authorities. Access to the eCRF will be password controlled and will conform with 21 CFR Part 11.

After every on-site audit, the Investigator will receive an audit confirmation by the auditor. This must be filed together with the study documentation and be made available to the regulatory authorities in case of supervision. At the end of the study, audit certificates will be included in the final report.

The Sponsor or designated representatives will affirm and uphold the principle of the subject's right to protection against the invasion of privacy. Throughout the study, all data will only be identified by subject number. Anonymity of the data will be maintained in all data analyses.

#### **Archiving Study Records**

Study records are to be maintained for a period defined by the laws and regulations of the participating country. For this study, a minimum of 2 years is required after the latter of the following two dates: the date the investigation was terminated or completed or the date the records are no longer required for purposes of supporting an FDA approval application.

| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE: |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 26 OF 33 |
| Active | Informed Vital Core, Pulse Rate Clinical Study Protocol | IVC-400-006 | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| March 31, 2023 | Chris Joslin | Mark Whitehouse | |

Copies of all case report forms completed on subjects will be retained in individual subject files by the Investigator in a secure location.

#### ETHICAL, LEGAL, AND ADMINISTRATIVE ASPECTS

#### **Sponsor Responsibilities**

The Sponsor or their designee will conduct a remote or in-person site visit to verify the qualification of each Investigator, inspect the site facilities, and inform the Investigator of responsibilities and the procedures for ensuring adequate and correct documentation.

#### **Investigator Responsibilities**

The Investigator is required to prepare and maintain adequate and accurate case histories designed to record all observations and other data pertinent to the study for each study subject. All information recorded on the eCRFs must be consistent with the subjects' source documentation, i.e., medical records.

#### **Good Clinical Practice**

The procedures set out in this study protocol are designated to ensure that the Sponsor and the Investigator abide by the principles of the Good Clinical Practice (GCP) guidelines of the International Conference on Harmonization (ICH) and of the Declaration of Helsinki (2000 with clarification in 2004 and as amended thereto). The study also will be carried out in keeping with local legal requirements, as appropriate.

#### **Protocol Approval and Amendment**

Before the start of the study, the study protocol and/or other relevant documents will be approved by the IRB/REB or other Competent Regulatory Authorities in accordance with local legal requirements. The Sponsor must ensure that all ethical and legal requirements have been met before the first subject is enrolled in the study.

| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE: |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 27 OF 33 |
| Active | Informed Vital Core, Pulse Rate Clinical Study Protocol | IVC-400-006 | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| March 31, 2023 | Chris Joslin | Mark Whitehouse | |

The protocol is to be followed exactly. To alter the protocol, amendments must be written, receive approval from the appropriate personnel, and receive IRB or other Competent Regulatory Authorities approval prior to implementation, as appropriate. If preliminary or interim review indicates that modification should be made in the experimental design, study parameters, subject selection, etc., these changes will be made after appropriate amendment(s) to this protocol with the mutual approval of the Sponsor and the Investigator. Any protocol change that may significantly affect the safety of study subjects must also be submitted for review and approval by the IRB prior to implementation.

Administrative changes not affecting the subject risk/benefit may be made without the need for a formal amendment. All amendments will be distributed to all protocol recipients, with appropriate instructions.

#### Termination of the Study

If the Investigator or Sponsor becomes aware of conditions or events that suggest a possible study-related hazard to subjects if the study continues, they may recommend to the Sponsor that the study be terminated after appropriate consultation between the relevant parties. The decision to terminate the study remains with the Sponsor. The study may also be terminated early at the Sponsor's discretion in the absence of such a finding. All enrolled subjects to that point will be notified of the study termination and reassured regarding depersonalization of any accrued specimens.

Conditions that may warrant termination by the Sponsor may include, but are not limited to, the discovery that in the opinion of the Sponsor, the study poses an unexpected, significant, or unacceptable risk to the subjects enrolled in the study. Additionally, a decision on the part of the Sponsor to suspend or discontinue development of the investigational device may be made.

#### Confidentiality

All study findings and documents will be regarded as confidential. The Investigator and members of his/her staff must not disclose such information without prior written approval from the Sponsor.

| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE: |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 28 OF 33 |
| Active | Informed Vital Core, Pulse Rate Clinical Study Protocol | IVC-400-006 | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| March 31, 2023 | Chris Joslin | Mark Whitehouse | |

The anonymity of participating study subjects must be maintained. Subjects will be identified on eCRFs and other documents submitted to the Sponsor by their subject number, not by name. Documents not to be submitted to the Sponsor that identify the subject (e.g., the signed informed consent) must be maintained in confidence by the Investigator.

#### **Publication**

At the conclusion of the study, publication of the primary study outcomes may be prepared for publication in a reputable scientific journal. The publication of the principal results from any single center or other collaborative experience within the study is not allowed until the preparation and publication of the primary study outcomes. Publication of the study results with the assent of the Sponsor and Investigators should not be delayed for more than 12 months after completion of the study.

#### **Site Training**

All Investigators and appropriate study staff will be required to participate in an on-site or web-based training (or initiation if appropriate) to provide orientation and training regarding the applicable study-specific procedures, protocol, and eCRFs.

| INFORMED MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE: |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 29 OF 33 |
| Active | Informed Vital Core, Pulse Rate Clinical Study Protocol | IVC-400-006 | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| March 31, 2023 | Chris Joslin | Mark Whitehouse | |

#### **Required Reports**

**Table 3- Reporting Requirements** 

| Event | Report to | Timing of Report |
|---|---|---|
| Study-related<br>AEs/SAEs/UADEs | Sponsor | Within 24 hours of the study site becoming aware of such events |
| Withdraw of IRB approval | Sponsor | Within 5 working days |
| Any deviation from the protocol to protect the life or physical well-being of a subject in an emergency situation | Sponsor and IRB | As soon as possible, but in no event later than 5 working days after the emergency occurred |
| Any study-specific procedure(s) being performed without prior written informed consent being obtained | Sponsor and IRB | Within 5 working days of the study-specific procedure(s) being performed |

#### **Product Complaints**

Any alleged deficiency related to the identity, quality, purity, durability, reliability, safety, effectiveness, or performance of a Mindset Medical product (IVC Application) shall be reported by the site to the IRB (if required) as soon as possible and to Mindset Medical via email within 3 working days after the deficiency was identified.

| INFORMED MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE: |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 30 OF 33 |
| Active | Informed Vital Core, Pulse Rate Clinical Study Protocol | IVC-400-006 | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | · |
| March 31, 2023 | Chris Joslin | Mark Whitehouse | |

The site shall record the following on the product complaint form for each complaint:

- Date of complaint
- Description of the complaint, and
- Any associated adverse event(s), if applicable.

The product, along with associated components/accessories, associated with the complaint shall be returned per Sponsor instructions as soon as possible.

#### **Contact Information**



| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE: |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 31 OF 33 |
| Active | Informed Vital Core, Pulse Rate Clinical Study Protocol | IVC-400-006 | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| March 31, 2023 | Chris Joslin | Mark Whitehouse | |

## Device Regulatory Approval/Clearance



Per FDA Guidance document, Information Sheet Guidance For IRBs, Clinical Investigators, and Sponsors Significant Risk and Nonsignificant Risk Medical Device Studies, NSR device studies do not have to have an IDE application approved by FDA. However, an IRB's NSR determination of this study is required.

| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE: |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 32 OF 33 |
| Active | Informed Vital Core, Pulse Rate Clinical Study Protocol | IVC-400-006 | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| March 31, 2023 | Chris Joslin | Mark Whitehouse | |

## Table of Common Acronyms

| | Table of Common Acronyms |
|---|---|
| AE | Adverse Event |
| BPM | Beats per Minute |
| DMP | Data Management Plan |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Report Form |
| HIPAA | Health Information Portability and Accountability Act |
| HTTPS | Hypertext Transfer Protocol Secure |
| HR | Heart Rate |
| ICH-GCP | International Conference of Harmonization Good Clinical Practice |
| ITC | Intent to Capture |
| IVC | Informed Vital Core app |
| NSR | Non-Significant Risk |
| PPG | Photoplethysmography |

| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE: |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 33 OF 33 |
| Active | Informed Vital Core, Pulse Rate Clinical Study Protocol | IVC-400-006 | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| March 31, 2023 | Chris Joslin | Mark Whitehouse | |

| Table of Common Acronyms | |
|--------------------------|-------------------------------------|
| PR | Pulse Rate |
| RGB | Red, Green, Blue |
| RMS | Root Mean Square |
| ROI | Region of Interest |
| rPPG | Remote Photoplethysmography |
| RSA encryption | Rivest-Shamir-Adleman encryption |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SMS | Short Message Service |
| URL | Uniform Resource Locator |
| UADE | Unanticipated Adverse Device Effect |

## References

FDA Guidance Document, Information Sheet Guidance For IRBs, Clinical Investigators, and Sponsors Significant Risk and Nonsignificant Risk Medical Device Studies, January 2006

| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE: |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 1 OF 25 |
| Active | Informed Vital Core –Clinical Study Instruction Guide: Pulse Rate | IVC-400-006g | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| April 5, 2023 | Chris Joslin | Mark Whitehouse | |

# Informed Vital Core Clinical Study Instruction Guide: Pulse Rate

| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE: |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 2 OF 25 |
| Active | Informed Vital Core –Clinical Study Instruction Guide:<br>Pulse Rate | IVC-400-006g | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| April 5, 2023 | Chris Joslin | Mark Whitehouse | |

## **Table of Contents**

| 1. | INTRODUCTION | 3 |
|---|---|---|
| 2. | CLINICAL STUDY MATERIALS AND EQUIPMENT | 3 |
| 3. | EQUIPMENT/ITEMS NEEDEDSTUDY ENVIRONMENT REQUIREMENTS | 3 |
| | 3.1. Warnings | 4 |
| 4. | VERIFY ECG SETTINGS | 5 |
| 5. | ECG PREPARATION | 9 |
| 6. | SENDING THE IVC APP | 12 |
| 7. | PREPARING THE IVC APP FOR PR MEASUREMENT | 14 |
| 8. | UPLOADING THE ECG DATA FROM THE THUMB DRIVE | 17 |
| 9. | VERIFY XML FILES ARE IN GOOGLE DRIVE | 22 |
| ΑP | PENDIX A – CLOCK SYNCHRONIZATION BETWEEN ECG AND IVC APP MOBILE PHONE | 24 |

| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE: |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 3 OF 25 |
| Active | Informed Vital Core –Clinical Study Instruction Guide: Pulse Rate | IVC-400-006g | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| April 5, 2023 | Chris Joslin | Mark Whitehouse | |

## Informed Vital Core Instructions IVC-PR-CLINICAL-STUDY Pulse Rate PRO

#### 1. Introduction

The instruction guide details the equipment used and the steps necessary to conduct the Informed Vital Core Pulse Rate Clinical Study IVC-400-006 comparing pulse rate (PR) measurements using the Informed Vital Core Application (IVC App) and a heart rate (HR) measured by an ECG device.

#### 2. Clinical Study Materials and Equipment

Mindset Medical (Sponsor) will provide the following materials:

- One mobile phone to run the Informed Vital Core Application, equipped with Google Voice phone number, Google Drive, and Gmail address (IVC Mobile Phone)
- Edan SE-301 ECG device with patient cable
- ECG Power Cord
- Spare disposable tab electrodes (one-time use per subject)
- Alcohol wipes
- Thumb drive
- USB-C to USB-A cable
- Make-up removal wipes
- Informed Vital Core PRO (IVC-PR-CLINICAL-STUDY)
- Phone Stand
- Phone Charger

#### 3. Study Environment Requirements

The study environment has the following requirements:

- Quiet room
- Comfortable chair
- Table at normal height (i.e., office desk or kitchen table)
- Wi-fi access
- Normal lighting with face being uniformly lit
  - Ensure there are no shadows, dark spots, or bright spots on the subject's face
  - No movement in the background behind the subjects
  - No varied lighting from windows, computer screens, or TV on the subject's face or behind the subject.
| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE: |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 4 OF 25 |
| Active | Informed Vital Core –Clinical Study Instruction Guide:<br>Pulse Rate | IVC-400-006g | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| April 5, 2023 | Chris Joslin | Mark Whitehouse | |

#### 3.1. Warnings

- The subject's face must be well illuminated with no shadows, including shadows cast from eyeglasses on the cheeks, no dark spots or bright spots falling across their face. Ensure the lighting direction is in front of the subject.
- Do not place subjects in front of windows or open spaces that would allow for bright light to shine from behind the subject, lowering the quality of the lighting on the face.
- Subjects should have no movement in background no TVs, people walking behind, flashing lights or shadows, or moving fans.
- No hats, do-rags, or masks should be worn by the subject. The forehead, cheeks, and chin need to be visible.
- Heavy bangs and hair should be pulled away from the subject's face.
- Ensure the subject does not have any makeup, lotion, sunscreen, etc. on their cheeks, forehead, and chin. Clean, bare skin on the subject's face is required and makeup removal wipes may be used to remove anything on the cheeks, forehead, or chin.
- The subject must remain still during the 60-second measurement session.
  - No talking
  - No movement of the head, mouth, leg, or arms to which ECG electrodes are attached.
- Ensure that the disposable ECG tabs and electrodes are securely adhered to the subject. You may need
  to use medical tape to properly secure the electrodes to the subject and ensure the disposable tabs are
  not pulling away from the skin.
  - The disposable tabs are to be used once per subject and then discarded.
  - Excessive hair may need to be shaved away from the subject's skin to ensure adherence with the disposable electrodes.

| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE: |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 5 OF 25 |
| Active | Informed Vital Core –Clinical Study Instruction Guide:<br>Pulse Rate | IVC-400-006g | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| April 5, 2023 | Chris Joslin | Mark Whitehouse | |

## 4. Verify ECG Settings



| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE: |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 6 OF 25 |
| Active | Informed Vital Core –Clinical Study Instruction Guide:<br>Pulse Rate | IVC-400-006g | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| April 5, 2023 | Chris Joslin | Mark Whitehouse | |



| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE: |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 7 OF 25 |
| Active | Informed Vital Core –Clinical Study Instruction Guide:<br>Pulse Rate | IVC-400-006g | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| April 5, 2023 | Chris Joslin | Mark Whitehouse | |



| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE: |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 8 OF 25 |
| Active | Informed Vital Core –Clinical Study Instruction Guide: Pulse Rate | IVC-400-006g | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| April 5, 2023 | Chris Joslin | Mark Whitehouse | |



| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE: |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 9 OF 25 |
| Active | Informed Vital Core –Clinical Study Instruction Guide: Pulse Rate | IVC-400-006g | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| April 5, 2023 | Chris Joslin | Mark Whitehouse | |

### 5. ECG Preparation



| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE: |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 10 OF 25 |
| Active | Informed Vital Core –Clinical Study Instruction Guide:<br>Pulse Rate | IVC-400-006g | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| April 5, 2023 | Chris Joslin | Mark Whitehouse | |

| | · |
|---|---|
| Step | Task |
| 6. | Take an alcohol swab and clean both forearms (middle) and the left leg above the ankle. Shave hair from electrode sites, if necessary. Excessive hair prevents a good connection. Dry the skin with a gauze pad to increase capillary blood flow to the tissues and to remove the dead, dry skin cells and oils. |
| 7. | Place a disposable tab electrode on the cleaned forearms and above the left ankle. Fully attach the alligator clips to the electrodes. • RA white (inside right arm) • LA black (inside left arm) • LL red (above the inside left ankle) |
| | ① Left Forearm ② Right Forearm ③ Left Ankle |
| | Ensure that all alligator clips are completely attached to the respective disposable electrode tab and that all tabs are securely fixed to the respective part of the body. NOTE: you can use medical adhesive tape to secure the alligator clips and disposable taps if necessary. |
| | Right arm alligator clip |
| | Left arm alligator clip |

| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE: |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 11 OF 25 |
| Active | Informed Vital Core –Clinical Study Instruction Guide: Pulse Rate | IVC-400-006g | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| April 5, 2023 | Chris Joslin | Mark Whitehouse | |



| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE: |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 12 OF 25 |
| Active | Informed Vital Core –Clinical Study Instruction Guide:<br>Pulse Rate | IVC-400-006g | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| April 5, 2023 | Chris Joslin | Mark Whitehouse | |

### 6. Sending the IVC App



| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE: |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 13 OF 25 |
| Active | Informed Vital Core –Clinical Study Instruction Guide:<br>Pulse Rate | IVC-400-006g | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| April 5, 2023 | Chris Joslin | Mark Whitehouse | |



| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE: |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 14 OF 25 |
| Active | Informed Vital Core –Clinical Study Instruction Guide: Pulse Rate | IVC-400-006g | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| April 5, 2023 | Chris Joslin | Mark Whitehouse | |

# 7. Preparing the IVC App for PR Measurement

| Step | Task |
|---|---|
| 1. | Ensure the subject has been sitting comfortably for 5 minutes, positioned behind a table of normal height with their back pressed against the seat rest, their feet flat on the floor, legs uncrossed, and their face uniformly lit with the light in front of the subject. |
| 2. | Tap on the Google Voice App on the mobile phone. |
| 3. | Tap the link contained in the SMS Message. Contained to the Contained of the SMS Message Contained of the Contained of t |
| 4. | When the Chrome mobile web browser is opened, tap and enter 01/01/2000 into the DOB confirmation field. |
| 5. | Tap the Continue button. Tap the Start button. |
| ٥. | Tap the Start button. |

| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE: |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 15 OF 25 |
| Active | Informed Vital Core –Clinical Study Instruction Guide:<br>Pulse Rate | IVC-400-006g | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| April 5, 2023 | Chris Joslin | Mark Whitehouse | |



| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE: |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 16 OF 25 |
| Active | Informed Vital Core –Clinical Study Instruction Guide:<br>Pulse Rate | IVC-400-006g | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| April 5, 2023 | Chris Joslin | Mark Whitehouse | |



10. When the IVC App measurement session is complete, a pulse rate measurement is displayed.

| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE: |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 17 OF 25 |
| Active | Informed Vital Core –Clinical Study Instruction Guide:<br>Pulse Rate | IVC-400-006g | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| April 5, 2023 | Chris Joslin | Mark Whitehouse | |



### 8. Uploading the ECG Data from the Thumb Drive

| Step | Task |
|---|---|
| 1. | Remove the thumb drive from the back of the ECG machine and insert the USB-A to USB-C adapter |
| | (USB-A side). |
| 2. | Insert the USB-C side of the USB-A to USB-C adapter into the mobile phone. |

| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE: |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 18 OF 25 |
| Active | Informed Vital Core –Clinical Study Instruction Guide: Pulse Rate | IVC-400-006g | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| April 5, 2023 | Chris Joslin | Mark Whitehouse | |



| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE: |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 19 OF 25 |
| Active | Informed Vital Core –Clinical Study Instruction Guide: Pulse Rate | IVC-400-006g | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| April 5, 2023 | Chris Joslin | Mark Whitehouse | |



| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE: |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 20 OF 25 |
| Active | Informed Vital Core –Clinical Study Instruction Guide:<br>Pulse Rate | IVC-400-006g | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| April 5, 2023 | Chris Joslin | Mark Whitehouse | |



| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE: |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 21 OF 25 |
| Active | Informed Vital Core –Clinical Study Instruction Guide: Pulse Rate | IVC-400-006g | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| April 5, 2023 | Chris Joslin | Mark Whitehouse | |



| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE: |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 22 OF 25 |
| Active | Informed Vital Core –Clinical Study Instruction Guide: Pulse Rate | IVC-400-006g | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| April 5, 2023 | Chris Joslin | Mark Whitehouse | |



# 9. Verify XML Files are in Google Drive

| Step | Task |
|---|---|
| 1. | In a web-browser on your laptop, go to <a href="https://drive.google.com">https://drive.google.com</a> . |
| 2. | Click on the G-Suite account associated with your clinical site (i.e., 301, 302). |

| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE: |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 23 OF 25 |
| Active | Informed Vital Core –Clinical Study Instruction Guide:<br>Pulse Rate | IVC-400-006g | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| April 5, 2023 | Chris Joslin | Mark Whitehouse | |



| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE: |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 24 OF 25 |
| Active | Informed Vital Core –Clinical Study Instruction Guide: Pulse Rate | IVC-400-006g | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| April 5, 2023 | Chris Joslin | Mark Whitehouse | |

### Appendix A – Clock Synchronization between ECG and IVC App Mobile Phone



| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE: |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 25 OF 25 |
| Active | Informed Vital Core –Clinical Study Instruction Guide: Pulse Rate | IVC-400-006g | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| April 5, 2023 | Chris Joslin | Mark Whitehouse | |



1

| Visit | |
|------------------------------|-------------------------------------------|
| Visit Name: | |
| Visit Date: | |
| Informed Consent | |
| Informed Consent date: | |
| Protocol Version Date: | Please Select |
| Demographics | |
| Date of Birth: | |
| Age: | year(s) |
| Sex: | Female Male |
| Ethnicity: | Not Hispanic or Latino |
| | Hispanic or Latino Unknown |
| Race (check all that apply): | American Indian or Alaska Native |
| | Asian |
| | Black or African American |
| | Native Hawaiian or Other Pacific Islander |
| | White |
| | Other |
| Other Specify: | |

Version: 1.0.0.0

dsg<sub>edc</sub>.

2



| Visit |
|---|
| Visit Name: |
| Visit Date: |
| Inclusion/Exclusion |
| Did the subject meet all the inclusion and none of the exclusion criteria? Yes No |
| Inclusion Criteria |
| Subjects 22 - 85 years of age: Yes No |
| Subjects willing to sign the Informed Consent Form and comply with the protocol: Yes No |
| Exclusion Criteria |
| Subjects required to wear mask or bandage that obstructs forehead, cheeks, or chin: Yes No |
| Refusal to remove makeup, sunscreen, lotion, clothing, or items obstructing the face Yes No for the duration of readings: |
| Presence of facial tattoos, large birthmarks, or other skin alterations (scars, hemangiomas, vitiligo) on upper cheeks (cheekbone) or forehead of the subject: |
| Condition that does not allow the subject to remain still for 60 seconds at a time: Yes No |
| Subjects with cardiac arrhythmia: Yes No |
| Any known medical condition which may result in an inaccurate measurement using the reference device: |
| Subjects with the inability to complete an ECG: Yes No |

| | Protocol Number: | Site Number: | Subject ID: | eCRF: |
|---------|------------------|--------------|-------------|-------|
| dsgedet | | | | 3 |

| Visit | |
|---|---|
| Visit Name: | |
| Visit Date: | |
| Fitzpatrick Scale Assignment | |
| Skin Type: | 1 - Pale White Skin |
| | 2 - White Skin |
| | 3 - Light Brown Skin |
| | 4 - Moderate Brown Skin |
| | 5 - Dark Brown Skin |
| | 6 - Deeply Pigmented Dark Brown to Black Skin |
| Physical Traits | |
| Is the subject wearing Glasses? | Yes No |
| Does the subject have facial hair? | Yes No |

Protocol Number: Site Number: Subject ID: eCRF:



| Visit | |
|-----------------------------------------------|--------|
| VISIL | |
| Visit Name: | |
| Visit Date: | |
| Cardiac Medical History | |
| Coronary Artery Disease? | Yes No |
| Congestive Heart Failure: | Yes No |
| Peripheral Arterial Disease: | Yes No |
| ESRD (End-Stage Renal Disease): | Yes No |
| Hemodialysis: | Yes No |
| Diabetes: | Yes No |
| HTN (Hypertension): | Yes No |
| History of Myocardial Infraction: | Yes No |
| Valvular Heart Disease: | Yes No |
| Cardiac Pacemaker: | Yes No |
| Pulmonary Embolism: | Yes No |
| Metastatic Cancer: | Yes No |
| Peripheral Vascular Disease: | Yes No |
| COPD (Chronic Obstructive Pulmonary Disease): | Yes No |
| Emphysema: | Yes No |
| History of DVT (Deep Vein Thrombosis): | Yes No |
| Other Heart disease: | Yes No |
| Specify: | |



| Visit | |
|-------------------------|----------------|
| Visit Name: | |
| Visit Date: | |
| Medical History | |
| Any chronic conditions? | Yes No |
| Diagnosis: | |
| Start Date: | |
| Ongoing: | |
| End Date: | Yes No |
| Elid Date. | |
| Diagnosis: | |
| Diagnosis. | |
| Start Date: | |
| Ongoing: | Yes No |
| End Date: | |
| Diagnosis: | |
| Start Date: | |
| Ongoing: | Yes No |
| End Date: | |
| Diagnosis: | |
| Diagliosis. | |
| Start Date: | |
| Ongoing: | Yes No |
| End Date: | |
| | aCRE Number: 5 |

Subject ID:

eCRF:

5



| Diagnosis: | |
|-------------|--------|
| Start Date: | |
| Ongoing: | Yes No |
| End Date: | |
| Diagnosis: | |
| Start Date: | |
| Start Date: | |
| Ongoing: | Yes No |
| End Date: | |
| Diagnosis: | |
| Start Date: | |
| Ongoing: | |
| | Yes No |
| End Date: | |
| Diagnosis: | |
| Start Date: | |
| Ongoing: | Yes No |
| End Date: | |
| Diagnosis: | |
| _ | |
| Start Date: | |

| dsg <sub>edc</sub> , | Protocol Number: | Site Number: | Subject ID: | eCRF:<br>5 |
|---|---|---|---|---|
| | Ongoing: Yes | No | | |
| | End Date: | | | |
| | Diagnosis: | | | |
| | Start Date: | | | |

Ongoing: Yes No

End Date:

| Protocol | Number: | Site | Number: |
|----------|---------|------|---------|

dsg<sub>edc</sub>.

Subject ID:

eCRF:

6

| Visit | |
|-----------------------------------|--------|
| Visit Name: | |
| Visit Date: | |
| Pulse Rate | |
| Informed Vital Core Pulse Rate 1 | |
| Was pulse rate taken by IVC? | Yes No |
| Reason Not Done: | |
| Date Performed: | |
| Informed Vital Core Pulse Rate 1: | bpm |
| Informed Vital Core Pulse Rate 2 | |
| Was pulse rate taken by IVC? | Yes No |
| Reason Not Done: | |
| Date Performed: | |
| Informed Vital Core Pulse Rate 2: | bpm |

dsg<sub>edc</sub>,

7

| Visit | |
|----------------------------------|--------|
| Visit Name: | |
| Visit Date: | |
| Electrocardiogram | |
| ECG 1 | |
| Was ECG performed? | Yes No |
| Reason Not Performed: | |
| Date Performed: | |
| Have you uploaded the ECG Strip? | Yes No |
| Reason ECG Not Uploaded: | |
| ECG 2 | |
| Was ECG performed? | Yes No |
| Reason Not Performed: | |
| Date Performed: | |
| Have you uploaded the ECG Strip? | Yes No |
| Reason ECG Not Uploaded: | |



eCRF: 7.1

| Visit | |
|-----------------------------|---------------------|
| Visit Name: | |
| Visit Date: | |
| Electrocardiogram | |
| ECG 1 | |
| Was Rhythm strip received? | Yes No |
| Date Analyzed: | |
| | Not able to Analyze |
| Reason not able to Analyze: | |
| ECG Pulse Rate: | bpm |
| ECG 2 | |
| Was Rhythm strip received? | Yes No |
| Date Analyzed: | |
| | Not able to Analyze |
| Reason not able to Analyze: | |
| ECG Pulse Rate: | bpm |

Subject ID:

eCRF:

100



| Adverse Events | |
|------------------------------------------|---------------|
| Adverse Event: | |
| Start Date: | |
| Ongoing? | Yes No |
| End Date: | |
| Severity: | Please Select |
| Serious: | Yes No |
| Serious Adverse Event | |
| Life threatening: | Yes No |
| Significant Disability: | Yes No |
| Hospitalization: | Yes No |
| Date of Admission: | |
| Date of Discharge: | |
| Congenital Anomaly or Birth Defect: | Yes No |
| Other Medically Important Event: | Yes No |
| Death: | Yes No |
| Date of Death: | |
| Relationship to Study Procedure: | Please Select |
| Action Taken with Study Procedure: | Please Select |
| Other Action Taken: | |
| Any Unanticipated Adverse Device Effect: | Yes No |
| Outcome: | Please Select |
| Caused Study Discontinuation: | Yes No |

eCRF Number: 100



| Concomitant Medication | |
|---------------------------|---------------|
| Medication: | Please Select |
| Other Medication Specify: | |
| Indication: | Please Select |
| Indication Specify: | |
| Start Date: | |
| End Date: | |
| Ongoing: | Yes No |
| Dose: | |
| Dose Unit: | Please Select |
| Frequency: | Please Select |
| Route: | Please Select |



| Technical Fallback | |
|-----------------------------------------------|---------------|
| How many technical fall backs were performed? | Please Select |
| Technical Fallback session 1 | |
| Technical Fallback Session 1 Reason: | Please Select |
| Date of Fallback Session: | |
| Specify, Details 1: | |
| Technical Fallback session 2 | |
| Technical Fallback Session 2 Reason: | Please Select |
| Date of Fallback Session: | |
| Specify, Details 2: | |
| Technical Fallback session 3 | |
| Technical Fallback Session 3 Reason: | Please Select |
| Date of Fallback Session: | |
| Specify, Details 3: | |

| Protocol Number: | Site Number: | Subject ID: | eCRF: |
|------------------|--------------|-------------|-------|
| | | | 400 |

| Device Failure |
|------------------|
| Date of Failure: |
| Time of Failure: |
| Notes: |

dsg<sub>edc</sub>.
| rotocol Number: | Site Number: | Subject ID: |
|-----------------|--------------|-------------|

eCRF: 500

| dsg <sub>edc</sub> . |
|----------------------|
|----------------------|

| Protocol Deviation | |
|---------------------------------|---------------|
| Date of Deviation: | |
| Type of Deviation: | Please Select |
| Other, Specify: | |
| Brief Description of Deviation: | |

Version: 1.0.0.0

| Protocol Number: | Site Number: | Subject ID: | eCRF: |
|------------------|--------------|-------------|-------|
| | | | 600 |

| End of Study | |
|-------------------------------------|---------------|
| Completion or Discontinuation Date: | |
| Status: | Please Select |
| Comments: | |

Version: 1.0.0.0

eCRF Number: 600

dsg<sub>edc</sub>.

700



| Investigator Signature | |
|---|---|
| I have reviewed the case report form pages and confirm that, to this subject. | the best of my knowledge, they accurately reflect the study information obtained for |
| Investigator's Signature: | |
| Date of Signature: | |
| Time of Signature: | |

Version: 1.0.0.0







## About Advarra's IRB Roster/ Membership List

Advarra maintains one roster and follows specific regulations and policies to determine how each individual panel that reviews research will be comprised. Each convened IRB meeting that reviews research will include:

- No fewer than 5 voting members and no more than 9 voting members
- At least 1 scientific member for meetings reviewing US based research, and 2 scientific members for meetings reviewing Canadian research
- At least 1 non-scientific member
- Both men and women
- At least 1 person who is not otherwise affiliated with Advarra
  - o These individuals may be referred to as "unaffiliated" or "community" members
  - These members are identified in the list below with the letter "N" in the "Affiliated?" column



## Additional Information about IRB Review of Canadian Research

In addition to the requirements above, meetings where Canadian research is reviewed will include:

- At least 1 member knowledgeable in ethics
- At least 1 member knowledgeable in Canadian laws relevant to the biomedical research to be approved

All IRB members can review US based research. Members eligible to review Canada-based research are identified below with the letter "Y" in the "Reviews CAN Research?" column. Additionally, whether these members are deemed to be knowledgeable in ethics and/or knowledgeable in Canadian laws relevant to the biomedical research to be approved will be identified in the "CAN: Knowledgeable in ethics and/or law?" column.

#### About the IRB

Advarra is organized and operates in compliance with the US and Canadian regulations and policies governing research with human subjects, as applicable.

- Advarra's IRB is registered with <u>FDA and</u> OHRP.
- Advarra's voluntary Federal wide Assurance (FWA) has been approved by <u>OHRP</u>.
  - IRB Organization (IORG) Number: 0000635
  - FWA Number: 00023875
  - IRB Registration Number: 00000971
- Advarra is fully accredited by the <u>Association for the Accreditation of Human</u> <u>Research Protection Programs (AAHRPP)</u>

| Name | Credentials | Role | Primary Expertise | Affiliated? | Chair? | Reviews<br>CAN<br>Research? | CAN:<br>Knowledgeable in<br>ethics and/or law? |
|---|---|---|---|---|---|---|---|
| Altier, Sarah | EdD | Non-Scientist | Educator | N | | N | |
| Ambrosini, Daniel | BA, LLB, MSc, PhD | Other Scientist | Psychiatry/ Legal | N | | Y | Ethics, Law |
| Aramburu Alegria,<br>Christine | PhD, RN | Other Scientist | Nursing/ Social Psychology/<br>Transgender Issues | N | | N | |







| Name | Credentials | Role | Primary Expertise | Affiliated? | Chair? | Reviews<br>CAN<br>Research? | CAN:<br>Knowledgeable in<br>ethics and/or law? |
|---|---|---|---|---|---|---|---|
| Astein, Diego | MD | Physician<br>Scientist | Radiology | Y | Chair | Y | Ethics |
| Baird, Kristin | MD | Physician<br>Scientist | Oncology/ Pediatrician/<br>Hematology | N | | N | |
| Benedict, Wendy | BA | Non-Scientist | Social Worker | N | | N | |
| Bergstrom, Steven | MD | Physician<br>Scientist | Oncology/ Pediatrician/<br>Hematology | N | | N | |
| Berlin, Suzanne | DO | Physician<br>Scientist | Oncology/ Women's Cancers | N | | N | |
| Bernstein, Erica | PharmD, BCPS | Other Scientist | Pharmacology | N | | N | |
| Berry, Donna | PhD, RN, AOCN,<br>FAAN | Other Scientist | Nursing/ Oncology | N | | N | |
| Block, Michelle | MS, BS, RAC, CIP | Non-Scientist | Regulatory/DoD Regulated Research | Υ | | Υ | |
| Blum, Robert | PharmD | Other Scientist | Pharmacology | N | Chair | N | |
| Booker, Burthia | PhD | Other Scientist | Biomedical Sciences | N | | N | |
| Borgatta, Lynn | MD, MPH | Physician<br>Scientist | Obstetrics/ Gynecology | N | | Υ | |
| Bottorff, Michael | PharmD | Other Scientist | Pharmacology | N | | N | |
| Braun, Peter | MD | Physician<br>Scientist | Internal Medicine/ Infectious<br>Disease | N | | N | |
| Brock, Jennifer | RN | Other Scientist | Nursing/ Oncology | N | | N | |
| Brown, Janice | RPh, MLS | Non-Scientist | Educator/ Librarian | N | | N | |
| Brzozowski, Jane | MS, BS | Non-Scientist | Patient Advocacy | N | | N | |
| Burkey, Madison | BSN, RN, OCN | Other Scientist | Nursing/ Oncology | Υ | | Υ | |
| Byers, Derek | MD, PhD, FCCP | Physician<br>Scientist | Internal Medicine/<br>Immunology | N | | N | |
| Campbell, Laura | MD | Physician<br>Scientist | Oncology/ Hematology/<br>Pediatrics/ Bioethics | N | | N | |
| Carr, Raymond | RPh | Other Scientist | Pharmacist | N | | N | |
| Casabar, Ed | PharmD, BCPS,<br>AQ-ID | Other Scientist | Pharmacology | N | | N | |







| Name | Credentials | Role | Primary Expertise | Affiliated? | Chair? | Reviews<br>CAN<br>Research? | CAN:<br>Knowledgeable in<br>ethics and/or law? |
|---|---|---|---|---|---|---|---|
| Cavagnaro, Joy | PhD, DABT, RAC | Other Scientist | Toxicology/ Regulatory Affairs<br>Consultant | N | | N | |
| Chukwu, Bernadette | PharmD | Other Scientist | Pharmacovigilance/ Drug<br>Safety | Y | | N | |
| Cooper, Kindra | JD | Non-Scientist | Legal | N | | N | |
| Cooper, Phyllis | RN, BSN, OCN,<br>CCRP | Other Scientist | Nursing/ Oncology | N | | N | |
| Cosentino, Lidia | PhD | Other Scientist | Biology/ Protocol development | N | | Y | |
| Cram, Gary | AS | Non-Scientist | Ethics | N | | N | |
| Cullity, Connie | MD, MPH | Physician<br>Scientist | FDA Regulations | Y | | N | |
| Cummings, Theresa | RN, MS | Other Scientist | Nursing/ Public Health | N | | N | |
| Davidson, Barbara | MS, RN, MSN,<br>CCRC | Other Scientist | Community Health Nursing | Y | | Y | |
| Davidson, Susan | MD | Physician<br>Scientist | Infectious Disease/<br>Homeostasis | N | | N | |
| Davis, Hannah | BS, MS | Other Scientist | Biology / Biomedical | Υ | | N | |
| Desai, Pankaj | PhD | Other Scientist | Biopharmaceutics/<br>Pharmacokinetics | N | | N | |
| Dorsch, Kimberly | BS | Other Scientist | Stem Cell/ Tissue Research | N | | N | |
| Drada, Denisse | | Non-Scientist | Regulatory | Υ | | Υ | |
| Duhon, Bryson | PharmD, BCPS | Other Scientist | Pharmacology | N | | N | |
| Dyson, Maynard | MD, MA, CIP | Physician<br>Scientist | Pediatrician/ Pulmonology | N | | N | |
| Ebert, Susan | MS, CIP | Non-Scientist | Regulatory | Υ | Sr. Chair<br>Dir. | N | |
| Fernicola, Daniel | MD, FACC | Physician<br>Scientist | Cardiology | N | | N | |
| Ferrell, David | ThB, BA, MA | Non-Scientist | Religion / Ethics | N | | Υ | Ethics |
| Fittizzi, Cheryl | RN, CIM, CIP | Other Scientist | Nursing/ Emergency Trauma/<br>Public Health | N | | N | |
| Fitzgerald, Michael | PhD | Other Scientist | Social Psychology | N | | N | |
| - | | | | | | | |





| Name | Credentials | Role | Primary Expertise | Affiliated? | Chair? | Reviews<br>CAN<br>Research? | CAN:<br>Knowledgeable in<br>ethics and/or law? |
|---|---|---|---|---|---|---|---|
| Fleck, David | PhD | Other Scientist | Psychiatry/ Behavioral<br>Neuroscience | N | | N | |
| Flowers, Janelle | MEd | Non-Scientist | Guidance Counselor | N | | N | |
| Foster, Joyce | MS | Non-Scientist | Family Therapy | N | | N | |
| Garrick, Tania | RN, BScN, MA | Other Scientist | Nursing | N | | Υ | |
| Gelinas, Luke | PhD, MAR, AB | Non-Scientist | Ethics | Y | Sr. Chair<br>Dir. | Y | Ethics |
| Georgiadis, Nina | MD | Physician<br>Scientist | Neonatal Intensive Care | N | | Υ | |
| Gill, Cyrus | RN, MS, CCRA | Other Scientist | Nursing/ Phase I | N | | N | |
| Ginnings, Susan | RPh | Other Scientist | Pharmacist | N | | N | |
| Gold, Herschel | BA, LLB | Non-scientist | Legal | N | | Υ | Ethics, Law |
| Goldman, Ran | MD, MHA, FRCPC | Physician<br>Scientist | Pediatrician | N | Chair | Υ | Ethics |
| Gonzales, Yury | MD, FACP | Physician<br>Scientist | Internal Medicine | N | | Υ | |
| Gordner, Linda | BA | Non-Scientist | Special Education | N | | Υ | |
| Gottke, Melissa | BA | Non-Scientist | Regulatory | Υ | | Υ | |
| Gray, Vernon | PhD | Non-Scientist | County Government<br>Administrator | N | | N | |
| Grimes, Brittany | MS | Non-Scientist | Regulatory | Υ | | Υ | |
| Groisman, Iris | PhD | Other Scientist | Biochemistry/ Radiobiology/<br>Pharmacogenetics | N | | Y | Ethics |
| Group, Melinda | BS, RPh | Other Scientist | Pharmacist/ Hospital<br>Research | N | | N | |
| Groza, Florina | MSc | Other Scientist | Biochemistry | Υ | | Υ | |
| Haffizulla, Farzanna | MD, FACP,<br>FAMWA | Physician<br>Scientist | Internal Medicine | N | | N | |
| Hensler, Carolyn | BS | Non-Scientist | Regulatory | N | | N | |
| Henson, Tricia | BA, RN | Other Scientist | Nursing Sciences | Υ | | Υ | |
| Hewes, Julia | MPH, BSN, RN,<br>OCN | Other Scientist | Nursing/ Oncology | N | | N | |







| Name | Credentials | Role | Primary Expertise | Affiliated? | Chair? | Reviews<br>CAN<br>Research? | CAN:<br>Knowledgeable in<br>ethics and/or law? |
|---|---|---|---|---|---|---|---|
| Hierholzer, Robert | MD | Physician<br>Scientist | Psychiatrist | N | | N | |
| Higley, Amanda | PhD, CIP | Other Scientist | Psychology | Υ | Chair | N | |
| Hill, Margaret | RN, MS | Other Scientist | Nursing/ Oncology/ Clinical<br>Trials Research | N | | N | |
| Hiller, David | BSN, RN, AEMT,<br>CIP | Other Scientist | Regulatory Critical Care<br>Nursing | Y | Chair | N | |
| Horton, Alicia | JD, MPH | Non-Scientist | Legal/ Public Health | N | | N | |
| Hoshower, Jason | BS, CIP | Non-Scientist | Regulatory | Υ | | Υ | |
| Houser, Patricia | MD | Physician<br>Scientist | Family Medicine | N | | N | |
| Hsiao, Karin | BS, MS, MBA | Other Scientist | Biomedical Engineering/<br>Device | N | | N | |
| Jacobsen, Eric | MD | Physician<br>Scientist | Oncology/ Lymphoma | N | | N | |
| Johnson, Dena | BS, MEd, CCRP,<br>CIP | Non-Scientist | Regulatory | Y | Chair | N | |
| Jordan, William | DO | Physician<br>Scientist | Oncology/ Medical | N | | N | |
| Kaul, Neha | MA, MS, BSc | Other Scientist | Social and Behavioral<br>Research; Regulatory;<br>Bioethics/Ethics; Molecular<br>Biology | Y | | N | |
| Keely, Levering | BSN, MPA | Other Scientist | Nursing/ Device specialist | N | | N | |
| Kim, James | MD, MBA | Physician<br>Scientist | General Practice/ Non-<br>Cancer Pain Management | N | | Y | |
| Kirk, Julia | BA, CIP | Non-Scientist | Regulatory | Y | | Υ | |
| Klaff, Ali | BSCIP | Non-Scientist | Regulatory | Υ | | Υ | |
| Knopman, David | MD | Physician<br>Scientist | Alzheimer/ Neurology | N | | N | |
| Kopec, Frederick | JD | Non-Scientist | Legal | N | Chair | N | |
| Kronish, Daniel | MD | Physician<br>Scientist | Oncology/ Pediatrician | Y | Chair | Y | |





| Name | Credentials | Role | Primary Expertise | Affiliated? | Chair? | Reviews<br>CAN<br>Research? | CAN:<br>Knowledgeable in<br>ethics and/or law? |
|---|---|---|---|---|---|---|---|
| Kuebler, Philip | MD, PhD, BS | Physician<br>Scientist | Internal Medicine/ Oncology/<br>Hematology | N | | N | |
| Kuzmanovic, Dario | BA, MHSc, CRA,<br>CHRC | Non-Scientist | Bioethics | N | | Y | Ethics, Law |
| Kysela, Kathleen | CIP | Non-Scientist | Regulatory | Υ | | Υ | |
| LaCount, Peter | MHS, MEd | Non-Scientist | Compliance Director | N | | N | |
| Lawrence, Janice | PhD, MA, BA, BPE | Other Scientist | Physical Ed/ Life Coach | N | | Υ | |
| Leduc, Lucie | LLM | Non-Scientist | Legal/ Ethics | N | | Υ | Ethics, Law |
| Leo, Jessica | AA, CIP | Non-Scientist | Regulatory | Υ | | Υ | |
| Letko, Erik | MD | Physician<br>Scientist | Ophthalmology/ Surgery | N | | N | |
| Lettman, Robert | BA, MBA, JD, PA | Non-Scientist | Legal | N | | N | |
| Lind, Alecia | BS, CIP | Non-Scientist | Regulatory | Υ | | Y | |
| Longstaff, Holly | PhD | Non-Scientist | Ethics | N | | Υ | Ethics |
| Lopez, Bennie | MBA | Non-Scientist | Educator | N | | N | |
| Lossada, Mery | MD, PA | Physician<br>Scientist | Psychiatry/ Neurology | N | | N | |
| Maloof, Damiana | MSN, RN, OCN | Other Scientist | Nursing/ Oncology | N | | N | |
| Martin, Christopher | PharmD, MS | Other Scientist | Pharmacology | N | Chair | N | |
| McPhillips, Joseph | PhD | Other Scientist | Clinical Research Consultant | N | | N | |
| Mensah, Sharon | MS | Other Scientist | Biological Sciences/ Clinical<br>Research | N | | N | |
| Mihalov, Linda | MD, FACOG | Physician<br>Scientist | Oncology/ Gynecology | N | | N | |
| Mitchell, Cameron | BA | Non-Scientist | Regulatory | Υ | | Υ | |
| Morse, Linda | RN, MSN, OCN | Other Scientist | Nursing/ Oncology | N | | N | |
| Mueller, Lava | MEd, MDiv | Non-scientist | Chaplain | N | | N | |
| Munk, Gary | PhD, MS, BS | Other Scientist | Virology/ Biosafety | N | | N | |
| Nattrass, Susan | OC, PhD, CBDT | Other Scientist | Osteoporosis and Women's<br>Health | N | | Y | |
| Neff, Robert | BS | Non-Scientist | Mobile Medical | N | | N | |
| Nolan, Joseph | PhD, MS, MA, BA,<br>BS | Other Scientist | Statistics | N | | N | |

CAN Office: 372 Hollandview Trail, Suite 300, Aurora, Ontario, Canada L4G 0A5





| Name | Credentials | Role | Primary Expertise | Affiliated? | Chair? | Reviews<br>CAN<br>Research? | CAN:<br>Knowledgeable in<br>ethics and/or law? |
|---|---|---|---|---|---|---|---|
| Noss, Michael | MD | Physician<br>Scientist | Family Medicine | N | | N | |
| O'Connell, Mary | | Non-Scientist | Regulatory | N | | N | |
| Odor, Erin | MA, CIP | Non-Scientist | Regulatory | Υ | Chair | N | |
| O'Leary, Maura | MD | Physician<br>Scientist | Oncology/ Pediatrician/<br>Hematology | N | | N | |
| Oliver, Ayesha | BS | Non-Scientist | Regulatory | Υ | | Υ | |
| Ott, Carl | MD, MPH | Physician<br>Scientist | Internal Medicine | N | | N | |
| Parker, R. Lamar | MD, FACOG, CPI | Physician<br>Scientist | Obstetrics/ Gynecology | N | | N | |
| Patrick, Kyle | DO | Physician<br>Scientist | Medical Research | N | | N | |
| Pettey, Cheri | MA, BA | Non-Scientist | Bioethics/ Philosophy | Υ | Chair | N | |
| Pfeiffer, Matthew | PhD | Other Scientist | Pharmacology/ Toxicology | N | | N | |
| Popovici-Toma, Dan | MD | Physician<br>Scientist | Medical Advisor | N | | Y | Ethics |
| Povar, Gail | MD, MPH, FACP | Physician<br>Scientist | Internal Medicine | N | Chair | N | |
| Psenicka, Eva | BSc | Non-Scientist | Physiology/ Regulatory | N | | Υ | |
| Ramjiawan, Bram | PhD | Other Scientist | Pharmacology | N | | Υ | |
| Randolph, Robert | DMin | Non-Scientist | Chaplain | N | | N | |
| Razzetti, Albert | MD | Physician<br>Scientist | Internal Medicine/<br>Pulmonology | N | | N | |
| Reddish, Mitchell | PhD | Non-Scientist | Professor/ Religious Studies/<br>Ethicist | N | | N | |
| Renner, Laura | BA | Non-Scientist | Regulatory | Υ | | N | |
| Rewers, Mae, Edna | MS, JD, MBA | Non-Scientist | Legal/ Healthcare/ Research<br>Compliance | N | | N | |
| Reynolds, Deborah | RN, OCN | Other Scientist | Nursing/ Oncology | N | | N | |
| Robinson, Deana | MPH, BS, LPN,<br>CPhT | Other Scientist | Clinical Research LPN | Y | | Y | |







| Name | Credentials | Role | Primary Expertise | Affiliated? | Chair? | Reviews<br>CAN<br>Research? | CAN:<br>Knowledgeable in<br>ethics and/or law? |
|---|---|---|---|---|---|---|---|
| Robinson, Richard | MD | Physician<br>Scientist | Medical Oncology/ Internal<br>Medicine | N | | N | |
| Romain, Michael | MD | Physician<br>Scientist | Internal Medicine | N | | N | |
| Romanchuk, Robert | BSHS, CIP,<br>CCRCP | Other Scientist | Clinical Research<br>Administration/ Respiratory<br>Therapy | N | | Y | |
| Rush, Jason | BS, CIP | Non-Scientist | Regulatory | Υ | | N | |
| Ruwart, Mary | PhD, BS | Other Scientist | Biophysics/ Biochemistry | N | | N | |
| Ryan, Laurajo | PharmD, MSc,<br>BCPS | Other Scientist | Pharmacology | N | | N | |
| Sadorra, Carol | PhD | Non-Scientist | Regulatory | Υ | | Υ | |
| Salama, Suzette | BPharm, MSc, PhD | Other Scientist | Ethicist/ Pharmacology | N | | Y | Ethics, Law |
| Saylor, Brenda | RN, BSN, ARM | Other Scientist | Community Health Nursing | Υ | | Υ | |
| Selsky, Clifford | PhD, MD | Physician<br>Scientist | Pediatrics, Hematology<br>Oncology | N | | N | |
| Sever, John | MD, PhD | Physician<br>Scientist | Pediatrician/ Infectious<br>Diseases | N | | N | |
| Shachar, Carmel | JD, MPH | Non-Scientist | Legal | N | | N | |
| Shafer, Michaela | PhD, RN | Other Scientist | Biomedical Research/<br>Nursing | N | | N | |
| Sheedy, Carmen | BA | Non-Scientist | Regulatory | Υ | | Υ | |
| Shulman, Mitchell | MDCM, FRCPC,<br>CSPQ | Physician<br>Scientist | Emergency Medicine | N | | Y | |
| Siegmann, Glenn | MS, RPh | Other Scientist | Pharmacist | N | | N | |
| Singh, Sukhbir | MD, MBA | Physician<br>Scientist | Psychiatry Research | Y | Chair | N | |
| Skroback, Judith | BM | Other Scientist | Devices | Y | | Υ | |
| Somerstein, Shari | RPh | Other Scientist | Pharmacist | N | | N | |
| Sommer, Dane | DMin, MDiv, BCC | Non-Scientist | Ministry | N | | N | |
| Spaulding, Trevor | BA, CIP | Non-Scientist | Regulatory | Υ | | Υ | |
| Stoltz, Randall | MD, CPI | Physician<br>Scientist | Phase I Research/<br>Cardiovascular | N | | N | |





| Name | Credentials | Role | Primary Expertise | Affiliated? | Chair? | Reviews<br>CAN<br>Research? | CAN:<br>Knowledgeable in<br>ethics and/or law? |
|---|---|---|---|---|---|---|---|
| Stone, Kurt | DD | Non-Scientist | Ministry | N | | N | |
| Strull, William | MD | Physician<br>Scientist | Internal Medicine | N | | N | |
| Taucher, Kate | PharmD, MHA,<br>BCOP | Other Scientist | Pharmacology | N | | N | |
| Teal, Marilyn | PharmD, BS | Other Scientist | Pharmacology | N | | Y | Ethics |
| Tillman, Beverly | RN, MSN | Other Scientist | Public Health | N | | N | |
| Tkaczuk, Katherine | MD | Physician<br>Scientist | Oncology/ Hematology | N | | N | |
| Vanderwel, Marianne | MEng, MSc | Other Scientist | Quality Assurance/ Research Ethics | N | | Y | Ethics, Law |
| Vernon, Kim | JD | Non-Scientist | Legal/ Prisoner Advocate | N | | N | |
| Walker, Christina | MD | Physician<br>Scientist | Family Medicine | N | | N | |
| Way, Cynthia | CIP | Non-Scientist | Regulatory/ Phase I<br>Research | N | | N | |
| Wells, Christine | MD | Physician<br>Scientist | Neurology/ Patient Advocate | N | | Y | Ethics |
| Westby, Christian | PhD | Other Scientist | Physiology | Υ | Chair | N | |
| Wood, Leslie | BA | Non-scientist | Communications | N | | Υ | Ethics |
| Wright-Moore,<br>Conschetta | RN, MPH | Other Scientist | Nursing/ Clinical Research | Y | | Y | |







# **Changes from All Member Roster Dated 03/01/2023**

| Member Name | Change | Date Change Made |
|---|---|---|
| Lauren Hartsmith | Removed | 04/01/2023 |
| Laura Campbell | Added | 04/11/2023 |
| Robert Romanchuk | Changed to Unaffiliated; removed Chair indication | 05/15/2023 |
| Neha Kaul | Added | 05/17/2023 |
| Mary Ruwart | Removed Chair indication | 05/19/2023 |









# About Advarra's IRB Roster/ Membership List

Advarra maintains one roster and follows specific regulations and policies to determine how each individual panel that reviews research will be comprised. Each convened IRB meeting that reviews research will include:

- No fewer than 5 voting members and no more than 9 voting members
- At least 1 scientific member for meetings reviewing US based research, and 2 scientific members for meetings reviewing Canadian research
- At least 1 non-scientific member
- Both men and women
- At least 1 person who is not otherwise affiliated with Advarra
  - o These individuals may be referred to as "unaffiliated" or "community" members
  - These members are identified in the list below with the letter "N" in the "Affiliated?" column



#### Additional Information about IRB Review of Canadian Research

In addition to the requirements above, meetings where Canadian research is reviewed will include:

- At least 1 member knowledgeable in ethics
- · At least 1 member knowledgeable in Canadian laws relevant to the biomedical research to be approved

All IRB members can review US based research. Members eligible to review Canada-based research are identified below with the letter "Y" in the "Reviews CAN Research?" column. Additionally, whether these members are deemed to be knowledgeable in ethics and/or knowledgeable in Canadian laws relevant to the biomedical research to be approved will be identified in the "CAN: Knowledgeable in ethics and/or law?" column.

#### About the IRB

Advarra is organized and operates in compliance with the US and Canadian regulations and policies governing research with human subjects, as applicable.

- Advarra's IRB is registered with <u>FDA and</u> OHRP.
- Advarra's voluntary Federal wide Assurance (FWA) has been approved by <u>OHRP</u>.
  - IRB Organization (IORG) Number: 0000635
  - o FWA Number: 00023875
  - IRB Registration Number: 00000971
- Advarra is fully accredited by the <u>Association for the Accreditation of Human</u> Research Protection Programs (AAHRPP)

| Name | Credentials | Role | Primary Expertise | Affiliated? | Chair? | Reviews<br>CAN<br>Research? | CAN:<br>Knowledgeable in<br>ethics and/or law? |
|---|---|---|---|---|---|---|---|
| Altier, Sarah | EdD | Non-Scientist | Educator | N | | N | |
| Ambrosini, Daniel | BA, LLB, MSc, PhD | Other Scientist | Psychiatry/ Legal | N | | Y | Ethics, Law |
| Aramburu Alegria, | PhD, RN | Other Scientist | Nursing/ Social Psychology/ | N | | N | |
| Christine | | | Transgender Issues | | | | |







| Name | Credentials | Role | Primary Expertise | Affiliated? | Chair? | Reviews<br>CAN<br>Research? | CAN:<br>Knowledgeable in<br>ethics and/or law? |
|---|---|---|---|---|---|---|---|
| Astein, Diego | MD | Physician<br>Scientist | Radiology | Y | Chair | Y | Ethics |
| Baird, Kristin | MD | Physician<br>Scientist | Oncology/ Pediatrician/<br>Hematology | N | | N | |
| Benedict, Wendy | BA | Non-Scientist | Social Worker | N | | N | |
| Bergstrom, Steven | MD | Physician<br>Scientist | Oncology/ Pediatrician/<br>Hematology | N | | N | |
| Berlin, Suzanne | DO | Physician<br>Scientist | Oncology/ Women's Cancers | N | | N | |
| Bernstein, Erica | PharmD, BCPS | Other Scientist | Pharmacology | N | | N | |
| Berry, Donna | PhD, RN, AOCN,<br>FAAN | Other Scientist | Nursing/ Oncology | N | | N | |
| Block, Michelle | MS, BS, RAC, CIP | Non-Scientist | Regulatory/DoD Regulated Research | Υ | | Υ | |
| Blum, Robert | PharmD | Other Scientist | Pharmacology | N | Chair | N | |
| Booker, Burthia | PhD | Other Scientist | Biomedical Sciences | N | | N | |
| Borgatta, Lynn | MD, MPH | Physician<br>Scientist | Obstetrics/ Gynecology | N | | Υ | |
| Bottorff, Michael | PharmD | Other Scientist | Pharmacology | N | | N | |
| Braun, Peter | MD | Physician<br>Scientist | Internal Medicine/ Infectious<br>Disease | N | | N | |
| Brock, Jennifer | RN | Other Scientist | Nursing/ Oncology | N | | N | |
| Brown, Janice | RPh, MLS | Non-Scientist | Educator/ Librarian | N | | N | |
| Brzozowski, Jane | MS, BS | Non-Scientist | Patient Advocacy | N | | N | |
| Burkey, Madison | BSN, RN, OCN | Other Scientist | Nursing/ Oncology | Υ | | Υ | |
| Byers, Derek | MD, PhD, FCCP | Physician<br>Scientist | Internal Medicine/<br>Immunology | N | | N | |
| Carr, Raymond | RPh | Other Scientist | Pharmacist | N | | N | |
| Casabar, Ed | PharmD, BCPS,<br>AQ-ID | Other Scientist | Pharmacology | N | | N | |
| Cavagnaro, Joy | PhD, DABT, RAC | Other Scientist | Toxicology/ Regulatory Affairs Consultant | N | | N | |







| Name | Credentials | Role | Primary Expertise | Affiliated? | Chair? | Reviews<br>CAN<br>Research? | CAN:<br>Knowledgeable in<br>ethics and/or law? |
|---|---|---|---|---|---|---|---|
| Chukwu, Bernadette | PharmD | Other Scientist | Pharmacovigilance/ Drug<br>Safety | Υ | | N | |
| Cooper, Kindra | JD | Non-Scientist | Legal | N | | N | |
| Cooper, Phyllis | RN, BSN, OCN,<br>CCRP | Other Scientist | Nursing/ Oncology | N | | N | |
| Cosentino, Lidia | PhD | Other Scientist | Biology/ Protocol development | N | | Y | |
| Cram, Gary | AS | Non-Scientist | Ethics | N | | N | |
| Cullity, Connie | MD, MPH | Physician<br>Scientist | FDA Regulations | Υ | | N | |
| Cummings, Theresa | RN, MS | Other Scientist | Nursing/ Public Health | N | | N | |
| Davidson, Barbara | MS, RN, MSN,<br>CCRC | Other Scientist | Community Health Nursing | Υ | | Y | |
| Davidson, Susan | MD | Physician<br>Scientist | Infectious Disease/<br>Homeostasis | N | | N | |
| Davis, Hannah | BS, MS | Other Scientist | Biology / Biomedical | Υ | | N | |
| Desai, Pankaj | PhD | Other Scientist | Biopharmaceutics/<br>Pharmacokinetics | N | | N | |
| Dorsch, Kimberly | BS | Other Scientist | Stem Cell/ Tissue Research | N | | N | |
| Drada, Denisse | | Non-Scientist | Regulatory | Υ | | Υ | |
| Duhon, Bryson | PharmD, BCPS | Other Scientist | Pharmacology | N | | N | |
| Dyson, Maynard | MD, MA, CIP | Physician<br>Scientist | Pediatrician/ Pulmonology | N | | N | |
| Ebert, Susan | MS, CIP | Non-Scientist | Regulatory | Υ | Sr. Chair<br>Dir. | N | |
| Fernicola, Daniel | MD, FACC | Physician<br>Scientist | Cardiology | N | | N | |
| Ferrell, David | ThB, BA, MA | Non-Scientist | Religion / Ethics | N | | Y | Ethics |
| Fittizzi, Cheryl | RN, CIM, CIP | Other Scientist | Nursing/ Emergency Trauma/<br>Public Health | N | | N | |
| Fitzgerald, Michael | PhD | Other Scientist | Social Psychology | N | | N | |
| Fleck, David | PhD | Other Scientist | Psychiatry/ Behavioral<br>Neuroscience | N | | N | |





| Name | Credentials | Role | Primary Expertise | Affiliated? | Chair? | Reviews<br>CAN<br>Research? | CAN:<br>Knowledgeable in<br>ethics and/or law? |
|---|---|---|---|---|---|---|---|
| Flowers, Janelle | MEd | Non-Scientist | Guidance Counselor | N | | N | |
| Foster, Joyce | MS | Non-Scientist | Family Therapy | N | | N | |
| Garrick, Tania | RN, BScN, MA | Other Scientist | Nursing | N | | Υ | |
| Gelinas, Luke | PhD, MAR, AB | Non-Scientist | Ethics | Y | Sr. Chair<br>Dir. | Y | Ethics |
| Georgiadis, Nina | MD | Physician<br>Scientist | Neonatal Intensive Care | N | | Y | |
| Gill, Cyrus | RN, MS, CCRA | Other Scientist | Nursing/ Phase I | N | | N | |
| Ginnings, Susan | RPh | Other Scientist | Pharmacist | N | | N | |
| Gold, Herschel | BA, LLB | Non-scientist | Legal | N | | Υ | Ethics, Law |
| Goldman, Ran | MD, MHA, FRCPC | Physician<br>Scientist | Pediatrician | N | Chair | Y | Ethics |
| Gonzales, Yury | MD, FACP | Physician<br>Scientist | Internal Medicine | N | | Y | |
| Gordner, Linda | BA | Non-Scientist | Special Education | N | | Υ | |
| Gottke, Melissa | BA | Non-Scientist | Regulatory | Υ | | Υ | |
| Gray, Vernon | PhD | Non-Scientist | County Government<br>Administrator | N | | N | |
| Grimes, Brittany | MS | Non-Scientist | Regulatory | Υ | | Υ | |
| Groisman, Iris | PhD | Other Scientist | Biochemistry/ Radiobiology/<br>Pharmacogenetics | N | | Y | Ethics |
| Group, Melinda | BS, RPh | Other Scientist | Pharmacist/ Hospital<br>Research | N | | N | |
| Groza, Florina | MSc | Other Scientist | Biochemistry | Υ | | Υ | |
| Haffizulla, Farzanna | MD, FACP,<br>FAMWA | Physician<br>Scientist | Internal Medicine | N | | N | |
| Hartsmith, Lauren | JD, CIP | Non-Scientist | Legal | Υ | | N | |
| Hensler, Carolyn | BS | Non-Scientist | Regulatory | N | | N | |
| Henson, Tricia | BA, RN | Other Scientist | Nursing Sciences | Y | | Υ | |
| Hewes, Julia | MPH, BSN, RN,<br>OCN | Other Scientist | Nursing/ Oncology | N | | N | |
| Hierholzer, Robert | MD | Physician<br>Scientist | Psychiatrist | N | | N | |





| CHRC | Name | Credentials | Role | Primary Expertise | Affiliated? | Chair? | Reviews<br>CAN<br>Research? | CAN:<br>Knowledgeable in<br>ethics and/or law? |
|---|---|---|---|---|---|---|---|---|
| Hiller, David BSN, RN, AEMT, CIP Other Scientist Regulatory Critical Care Nursing Nurs | Higley, Amanda | PhD, CIP | Other Scientist | Psychology | Υ | Chair | N | |
| CIP | Hill, Margaret | RN, MS | Other Scientist | | N | | N | |
| Hoshower, Jason BS, CIP Non-Scientist Regulatory Y Y Houser, Patricia MD Physician Scientist Family Medicine N N Hsiao, Karin BS, MS, MBA Other Scientist Biomedical Engineering/ Device N N Jacobsen, Eric MD Physician Scientist Oncology/ Lymphoma N N Johnson, Dena BS, MEd, CCRP, CIP Non-Scientist Regulatory Y Chair N Jordan, William DO Physician Scientist Oncology/ Medical N N N Keely, Levering BSN, MPA Other Scientist Nursing/ Device specialist N N N Kim, James MD, MBA Physician Scientist General Practice/ Non-Scientist N N Y Kirk, Julia BA, CIP Non-Scientist Regulatory Y Y Y Kirk, Julia BA, CIP Non-Scientist Regulatory Y Y Y Kird, Ali BSCIP Non-Scientist | Hiller, David | | Other Scientist | | Y | Chair | N | |
| Houser, Patricia MD Physician Scientist Scientist Family Medicine N N N Hsiao, Karin BS, MS, MBA Other Scientist Device Biomedical Engineering/ Device N N N Jacobsen, Eric MD Physician Scientist Oncology/ Lymphoma N N N Johnson, Dena BS, MEd, CCRP, CIP Non-Scientist Regulatory Y Chair N Jordan, William DO Physician Scientist Oncology/ Medical N N N Keely, Levering BSN, MPA Other Scientist Nursing/ Device specialist N N N Kim, James MD, MBA Physician Scientist Cancer Pain Management N Y Y Kirk, Julia BA, CIP Non-Scientist Regulatory Y Y Y Klaff, Ali BSCIP Non-Scientist Regulatory Y Y Y Knopman, David MD Physician Alzheimer/ Neurology N N N Kronish, Daniel MD Non-Scientist Legal N Chair | Horton, Alicia | JD, MPH | Non-Scientist | Legal/ Public Health | N | | N | |
| Hsiao, Karin BS, MS, MBA Other Scientist Biomedical Engineering/ Device Jacobsen, Eric MD Physician Scientist Povice Johnson, Dena BS, MEd, CCRP, CIP Jordan, William DO Physician Scientist Nursing/ Device specialist N N N Keely, Levering BSN, MPA Other Scientist Nursing/ Device specialist N N Kim, James MD, MBA Physician Scientist Cancer Pain Management Kirk, Julia BA, CIP Non-Scientist Regulatory Y Y Y Klaff, Ali BSCIP Non-Scientist Regulatory Y Y Y Klaff, Ali BSCIP Non-Scientist Regulatory Y Y Knopman, David MD Physician Scientist Legal N Kopec, Frederick JD Non-Scientist Legal N Kronish, Daniel MD Physician Scientist Physician Scientist Physician Scientist Cancer Pain Menagement Kronish, Daniel MD Physician Scientist Regulatory Y Kuzmanovic, Dario BA, MHSc, CRA, Non-Scientist Bioethics N Non-Scientist Scientist Regulatory N Non-Scientist Legal N Non-Scientist Cancer Pain Menagement N Kuzmanovic, Dario BA, MHSc, CRA, Non-Scientist Bioethics N Non-Scientist Regulatory N N N N N N N N N N N N N | Hoshower, Jason | BS, CIP | Non-Scientist | Regulatory | Υ | | Υ | |
| Device D | Houser, Patricia | MD | | Family Medicine | N | | N | |
| Scientist Johnson, Dena BS, MEd, CCRP, CIP CIP Jordan, William DO Physician Scientist Keely, Levering BSN, MPA Other Scientist Nursing/ Device specialist N Kim, James MD, MBA Physician General Practice/ Non- N Scientist Cancer Pain Management Kirk, Julia BA, CIP Non-Scientist Regulatory Y Klaff, Ali BSCIP Non-Scientist Regulatory Y Knopman, David MD Physician Scientist Regulatory N Kopec, Frederick JD Non-Scientist Legal Non-Scientist N Kopec, Frederick Non-Scientist Regulatory N Non-Scientist Regulatory N N Chair N Kronish, Daniel MD Physician Oncology/ Pediatrician Scientist N Kuebler, Philip MD, PhD, BS Physician Internal Medicine/ Oncology/ Scientist Hematology Kuzmanovic, Dario BA, MHSc, CRA, CHRC NOn-Scientist Bioethics N Y Ethics, Lat | Hsiao, Karin | BS, MS, MBA | Other Scientist | | N | | N | |
| College | Jacobsen, Eric | MD | | Oncology/ Lymphoma | N | | N | |
| Scientist Scie | Johnson, Dena | | Non-Scientist | Regulatory | Y | Chair | N | |
| Kim, JamesMD, MBAPhysician ScientistGeneral Practice/ Non-ScientistNYKirk, JuliaBA, CIPNon-ScientistRegulatoryYYKlaff, AliBSCIPNon-ScientistRegulatoryYYKnopman, DavidMDPhysician ScientistAlzheimer/ Neurology<br>ScientistNChairNKopec, FrederickJDNon-ScientistLegalNChairNKronish, DanielMDPhysician ScientistOncology/ Pediatrician<br>ScientistYChairYKuebler, PhilipMD, PhD, BSPhysician ScientistInternal Medicine/ Oncology/ HematologyNNNKuzmanovic, DarioBA, MHSc, CRA, CHRCNon-ScientistBioethicsNYEthics, Later | Jordan, William | DO | | Oncology/ Medical | N | | N | |
| Kirk, Julia BA, CIP Non-Scientist Regulatory Y Y Y Klaff, Ali BSCIP Non-Scientist Regulatory Y Y Knopman, David MD Physician Scientist Legal N Chair N Kronish, Daniel MD Physician Scientist Kuebler, Philip MD, PhD, BS Physician Scientist Hematology Kuzmanovic, Dario BA, MHSc, CRA, CHRC Scientist Cancer Pain Management Regulatory Y Y Regulatory Y Y Y Y Y Y Y Y Y Y Y Y Y Y Y Y Y Y Y | Keely, Levering | BSN, MPA | Other Scientist | Nursing/ Device specialist | N | | N | |
| Klaff, AliBSCIPNon-ScientistRegulatoryYYKnopman, DavidMDPhysician ScientistAlzheimer/ NeurologyNNKopec, FrederickJDNon-ScientistLegalNChairNKronish, DanielMDPhysician ScientistOncology/ PediatricianYChairYKuebler, PhilipMD, PhD, BSPhysician ScientistInternal Medicine/ Oncology/ HematologyNNNKuzmanovic, DarioBA, MHSc, CRA, CHRCNon-ScientistBioethicsNYEthics, Lateral Medicine/ CHRC | Kim, James | MD, MBA | | | N | | Υ | |
| Knopman, DavidMDPhysician ScientistAlzheimer/ NeurologyNNKopec, FrederickJDNon-ScientistLegalNChairNKronish, DanielMDPhysician ScientistOncology/ PediatricianYChairYKuebler, PhilipMD, PhD, BSPhysician ScientistInternal Medicine/ Oncology/ HematologyNNKuzmanovic, DarioBA, MHSc, CRA, CHRCNon-ScientistBioethicsNYEthics, Larchics, Larchics | Kirk, Julia | BA, CIP | Non-Scientist | Regulatory | Υ | | Υ | |
| Kopec, Frederick JD Non-Scientist Legal N Chair N Kronish, Daniel MD Physician Scientist Kuebler, Philip MD, PhD, BS Physician Scientist Hematology Kuzmanovic, Dario BA, MHSc, CRA, CHRC Scientist Bioethics N Y Chair Y Scientist N N N Scientist Hematology Kuzmanovic, Dario Scientist Bioethics N Y Ethics, Large CHRC | Klaff, Ali | BSCIP | Non-Scientist | Regulatory | Υ | | Υ | |
| Kronish, DanielMDPhysician ScientistOncology/ PediatricianYChairYKuebler, PhilipMD, PhD, BSPhysician ScientistInternal Medicine/ Oncology/ HematologyNNKuzmanovic, DarioBA, MHSc, CRA, CHRCNon-ScientistBioethicsNYEthics, Large Chromatology | Knopman, David | MD | • | Alzheimer/ Neurology | N | | N | |
| Scientist Kuebler, Philip MD, PhD, BS Physician Scientist Internal Medicine/ Oncology/ Hematology N N Kuzmanovic, Dario BA, MHSc, CRA, CHRC Non-Scientist Bioethics N Y Ethics, Large CHRC | Kopec, Frederick | JD | Non-Scientist | Legal | N | Chair | N | |
| Scientist Hematology Kuzmanovic, Dario BA, MHSc, CRA, Non-Scientist Bioethics N Y Ethics, Later CHRC | Kronish, Daniel | MD | | Oncology/ Pediatrician | Y | Chair | Y | |
| Kuzmanovic, Dario BA, MHSc, CRA, Non-Scientist Bioethics N Y Ethics, Later CHRC | Kuebler, Philip | MD, PhD, BS | • | | N | | N | |
| Kysela Kathleen CIP Non-Scientist Regulatory Y Y | Kuzmanovic, Dario | | Non-Scientist | · • | N | | Υ | Ethics, Law |
| Typola, mainton on non-ordinate mogalatory | Kysela, Kathleen | CIP | Non-Scientist | Regulatory | Υ | | Υ | |
| LaCount, Peter MHS, MEd Non-Scientist Compliance Director N N | LaCount, Peter | MHS, MEd | Non-Scientist | Compliance Director | N | | N | |

IRB Roster/ Membership List © 2022 Advarra | All rights reserved | Updated: March 1, 2023 HQ: 6100 Merriweather Dr., Suite 600, Columbia, Maryland 21044

CAN Office: 372 Hollandview Trail, Suite 300, Aurora, Ontario, Canada L4G 0A5 5 of 10







| Name | Credentials | Role | Primary Expertise | Affiliated? | Chair? | Reviews<br>CAN<br>Research? | CAN:<br>Knowledgeable in<br>ethics and/or law? |
|---|---|---|---|---|---|---|---|
| Lawrence, Janice | PhD, MA, BA, BPE | Other Scientist | Physical Ed/ Life Coach | N | | Υ | |
| Leduc, Lucie | LLM | Non-Scientist | Legal/ Ethics | N | | Y | Ethics, Law |
| Leo, Jessica | AA, CIP | Non-Scientist | Regulatory | Υ | | Y | |
| Letko, Erik | MD | Physician<br>Scientist | Ophthalmology/ Surgery | N | | N | |
| Lettman, Robert | BA, MBA, JD, PA | Non-Scientist | Legal | N | | N | |
| Lind, Alecia | BS, CIP | Non-Scientist | Regulatory | Υ | | Υ | |
| Longstaff, Holly | PhD | Non-Scientist | Ethics | N | | Y | Ethics |
| Lopez, Bennie | MBA | Non-Scientist | Educator | N | | N | |
| Lossada, Mery | MD, PA | Physician<br>Scientist | Psychiatry/ Neurology | N | | N | |
| Maloof, Damiana | MSN, RN, OCN | Other Scientist | Nursing/ Oncology | N | | N | |
| Martin, Christopher | PharmD, MS | Other Scientist | Pharmacology | N | Chair | N | |
| McPhillips, Joseph | PhD | Other Scientist | Clinical Research Consultant | N | | N | |
| Mensah, Sharon | MS | Other Scientist | Biological Sciences/ Clinical<br>Research | N | | N | |
| Mihalov, Linda | MD, FACOG | Physician<br>Scientist | Oncology/ Gynecology | N | | N | |
| Mitchell, Cameron | BA | Non-Scientist | Regulatory | Υ | | Y | |
| Morse, Linda | RN, MSN, OCN | Other Scientist | Nursing/ Oncology | N | | N | |
| Mueller, Lava | MEd, MDiv | Non-scientist | Chaplain | N | | N | |
| Munk, Gary | PhD, MS, BS | Other Scientist | Virology/ Biosafety | N | | N | |
| Nattrass, Susan | OC, PhD, CBDT | Other Scientist | Osteoporosis and Women's<br>Health | N | | Y | |
| Neff, Robert | BS | Non-Scientist | Mobile Medical | N | | N | |
| Nolan, Joseph | PhD, MS, MA, BA,<br>BS | Other Scientist | Statistics | N | | N | |
| Noss, Michael | MD | Physician<br>Scientist | Family Medicine | N | | N | |
| O'Connell, Mary | | Non-Scientist | Regulatory | N | | N | |
| Odor, Erin | MA, CIP | Non-Scientist | Regulatory | Υ | Chair | N | |
| O'Leary, Maura | MD | Physician<br>Scientist | Oncology/ Pediatrician/<br>Hematology | N | | N | |





| Name | Credentials | Role | Primary Expertise | Affiliated? | Chair? | Reviews<br>CAN<br>Research? | CAN:<br>Knowledgeable in<br>ethics and/or law? |
|---|---|---|---|---|---|---|---|
| Oliver, Ayesha | BS | Non-Scientist | Regulatory | Υ | | Υ | |
| Ott, Carl | MD, MPH | Physician<br>Scientist | Internal Medicine | N | | N | |
| Parker, R. Lamar | MD, FACOG, CPI | Physician<br>Scientist | Obstetrics/ Gynecology | N | | N | |
| Patrick, Kyle | DO | Physician<br>Scientist | Medical Research | N | | N | |
| Pettey, Cheri | MA, BA | Non-Scientist | Bioethics/ Philosophy | Υ | Chair | N | |
| Pfeiffer, Matthew | PhD | Other Scientist | Pharmacology/ Toxicology | N | | N | |
| Popovici-Toma, Dan | MD | Physician<br>Scientist | Medical Advisor | N | | Y | Ethics |
| Povar, Gail | MD, MPH, FACP | Physician<br>Scientist | Internal Medicine | N | Chair | N | |
| Psenicka, Eva | BSc | Non-Scientist | Physiology/ Regulatory | N | | Υ | |
| Ramjiawan, Bram | PhD | Other Scientist | Pharmacology | N | | Υ | |
| Randolph, Robert | DMin | Non-Scientist | Chaplain | N | | N | |
| Razzetti, Albert | MD | Physician<br>Scientist | Internal Medicine/<br>Pulmonology | N | | N | |
| Reddish, Mitchell | PhD | Non-Scientist | Professor/ Religious Studies/<br>Ethicist | N | | N | |
| Renner, Laura | BA | Non-Scientist | Regulatory | Υ | | N | |
| Rewers, Mae, Edna | MS, JD, MBA | Non-Scientist | Legal/ Healthcare/ Research<br>Compliance | N | | N | |
| Reynolds, Deborah | RN, OCN | Other Scientist | Nursing/ Oncology | N | | N | |
| Robinson, Deana | MPH, BS, LPN,<br>CPhT | Other Scientist | Clinical Research LPN | Υ | | Y | |
| Robinson, Richard | MD | Physician<br>Scientist | Medical Oncology/ Internal<br>Medicine | N | | N | |
| Romain, Michael | MD | Physician<br>Scientist | Internal Medicine | N | | N | |
| Romanchuk, Robert | BS, HS, CIP,<br>CCRCP, CCRC | Other Scientist | Clinical Research<br>Administration/ Respiratory<br>Therapy | Υ | Chair | Υ | |







| Name | Credentials | Role | Primary Expertise | Affiliated? | Chair? | Reviews<br>CAN<br>Research? | CAN:<br>Knowledgeable in<br>ethics and/or law? |
|---|---|---|---|---|---|---|---|
| Rush, Jason | BS, CIP | Non-Scientist | Regulatory | Υ | | N | |
| Ruwart, Mary | PhD, BS | Other Scientist | Biophysics/ Biochemistry | N | Chair | N | |
| Ryan, Laurajo | PharmD, MSc,<br>BCPS | Other Scientist | Pharmacology | N | | N | |
| Sadorra, Carol | PhD | Non-Scientist | Regulatory | Υ | | Υ | |
| Salama, Suzette | BPharm, MSc, PhD | Other Scientist | Ethicist/ Pharmacology | N | | Υ | Ethics, Law |
| Saylor, Brenda | RN, BSN, ARM | Other Scientist | Community Health Nursing | Υ | | Υ | |
| Selsky, Clifford | PhD, MD | Physician<br>Scientist | Pediatrics, Hematology<br>Oncology | N | | N | |
| Sever, John | MD, PhD | Physician<br>Scientist | Pediatrician/ Infectious<br>Diseases | N | | N | |
| Shachar, Carmel | JD, MPH | Non-Scientist | Legal | N | | N | |
| Shafer, Michaela | PhD, RN | Other Scientist | Biomedical Research/<br>Nursing | N | | N | |
| Sheedy, Carmen | BA | Non-Scientist | Regulatory | Υ | | Υ | |
| Shulman, Mitchell | MDCM, FRCPC,<br>CSPQ | Physician<br>Scientist | Emergency Medicine | N | | Y | |
| Siegmann, Glenn | MS, RPh | Other Scientist | Pharmacist | N | | N | |
| Singh, Sukhbir | MD, MBA | Physician<br>Scientist | Psychiatry Research | Y | Chair | N | |
| Skroback, Judith | BM | Other Scientist | Devices | Υ | | Υ | |
| Somerstein, Shari | RPh | Other Scientist | Pharmacist | N | | N | |
| Sommer, Dane | DMin, MDiv, BCC | Non-Scientist | Ministry | N | | N | |
| Spaulding, Trevor | BA, CIP | Non-Scientist | Regulatory | Υ | | Υ | |
| Stoltz, Randall | MD, CPI | Physician<br>Scientist | Phase I Research/<br>Cardiovascular | N | | N | |
| Stone, Kurt | DD | Non-Scientist | Ministry | N | | N | |
| Strull, William | MD | Physician<br>Scientist | Internal Medicine | N | | N | |
| Taucher, Kate | PharmD, MHA,<br>BCOP | Other Scientist | Pharmacology | N | | N | |
| Teal, Marilyn | PharmD, BS | Other Scientist | Pharmacology | N | | Υ | Ethics |
| Tillman, Beverly | RN, MSN | Other Scientist | Public Health | N | | N | |

IRB Roster/ Membership List © 2022 Advarra | All rights reserved | Updated: March 1, 2023 HQ: 6100 Merriweather Dr., Suite 600, Columbia, Maryland 21044

CAN Office: 372 Hollandview Trail, Suite 300, Aurora, Ontario, Canada L4G 0A5







| Name | Credentials | Role | Primary Expertise | Affiliated? | Chair? | Reviews<br>CAN<br>Research? | CAN:<br>Knowledgeable in<br>ethics and/or law? |
|---|---|---|---|---|---|---|---|
| Tkaczuk, Katherine | MD | Physician<br>Scientist | Oncology/ Hematology | N | | N | |
| Vanderwel, Marianne | MEng, MSc | Other Scientist | Quality Assurance/ Research<br>Ethics | N | | Y | Ethics, Law |
| Vernon, Kim | JD | Non-Scientist | Legal/ Prisoner Advocate | N | | N | |
| Walker, Christina | MD | Physician<br>Scientist | Family Medicine | N | | N | |
| Way, Cynthia | CIP | Non-Scientist | Regulatory/ Phase I<br>Research | N | | N | |
| Wells, Christine | MD | Physician<br>Scientist | Neurology/ Patient Advocate | N | | Υ | Ethics |
| Westby, Christian | PhD | Other Scientist | Physiology | Υ | Chair | N | |
| Wood, Leslie | BA | Non-scientist | Communications | N | | Υ | Ethics |
| Wright-Moore,<br>Conschetta | RN, MPH | Other Scientist | Nursing/ Clinical Research | Y | | Υ | |







# **Changes from All Member Roster Dated 12/01/2022**

| Member Name | Change | Date Change Made |
|-----------------|---------|------------------|
| Hannah Davis | Added | 12/20/2022 |
| Beth Overmoyer | Removed | 07/01/2022 |
| Nicole Sieffert | Removed | 12/09/2022 |







# About Advarra's IRB Roster/ Membership List

Advarra maintains one roster and follows specific regulations and policies to determine how each individual panel that reviews research will be comprised. Each convened IRB meeting that reviews research will include:

- No fewer than 5 voting members and no more than 9 voting members
- At least 1 scientific member for meetings reviewing US based research, and 2 scientific members for meetings reviewing Canadian research
- At least 1 non-scientific member
- Both men and women
- At least 1 person who is not otherwise affiliated with Advarra
  - These individuals may be referred to as "unaffiliated" or "community" members
  - These members are identified in the list below with the letter "N" in the "Affiliated?" column



### Additional Information about IRB Review of Canadian Research

In addition to the requirements above, meetings where Canadian research is reviewed will include:

- At least 1 member knowledgeable in ethics
- At least 1 member knowledgeable in Canadian laws relevant to the biomedical research to be approved

All IRB members can review US based research. Members eligible to review Canada-based research are identified below with the letter "Y" in the "Reviews CAN Research?" column. Additionally, whether these members are deemed to be knowledgeable in ethics and/or knowledgeable in Canadian laws relevant to the biomedical research to be approved will be identified in the "CAN: Knowledgeable in ethics and/or law?" column.

#### About the IRB

Advarra is organized and operates in compliance with the US and Canadian regulations and policies governing research with human subjects, as applicable.

- Advarra's IRB is registered with <u>FDA and OHRP</u>.
- Advarra's voluntary Federal wide Assurance (FWA) has been approved by <u>OHRP</u>.
  - o IRB Organization (IORG) Number: 0000635
  - FWA Number: 00023875
  - IRB Registration Number: 00000971
- Advarra is fully accredited by the <u>Association for the Accreditation of Human Research Protection Programs (AAHRPP)</u>

| Name | Credentials | Role | Primary Expertise | Affiliated? | Chair? | Primary(P) or<br>Alternate(A)? | Reviews<br>CAN<br>Research? | CAN:<br>Knowledgeable<br>in ethics and/or<br>law? |
|---|---|---|---|---|---|---|---|---|
| Altier, Sarah | EdD | Non-Scientist | Educator | N | | Α | N | |
| Ambrosini, Daniel | BA, LLB, MSc,<br>PhD | Other Scientist | Psychiatry/ Legal | N | | Α | Υ | Ethics, Law |







| Name | Credentials | Role | Primary Expertise | Affiliated? | Chair? | Primary(P) or<br>Alternate(A)? | Reviews<br>CAN<br>Research? | CAN:<br>Knowledgeabl<br>in ethics and/o<br>law? |
|---|---|---|---|---|---|---|---|---|
| Aramburu Alegria,<br>Christine | PhD, RN | Other Scientist | Nursing/ Social<br>Psychology/<br>Transgender Issues | N | | Α | N | |
| Astein, Diego | MD | Physician<br>Scientist | Radiology | Υ | Chair | Α | Y | Ethics |
| Baird, Kristin | MD | Physician<br>Scientist | Oncology/ Pediatrician/<br>Hematology | N | | Α | N | |
| Barr, Hallie | PharmD, MBA,<br>BCOP | Other Scientist | Pharmacy / Oncology | Y | | Α | N | |
| Benedict, Wendy | BA | Non-Scientist | Social Worker | N | | Α | N | |
| Bergstrom, Steven | MD | Physician<br>Scientist | Oncology/ Pediatrician/<br>Hematology | N | | Α | N | |
| Berlin, Suzanne | DO | Physician<br>Scientist | Oncology/ Women's<br>Cancers | N | | Α | N | |
| Bernstein, Erica | PharmD, BCPS | Other Scientist | Pharmacology | N | | Α | N | |
| Berry, Donna | PhD, RN, AOCN,<br>FAAN | Other Scientist | Nursing/ Oncology | N | | Α | N | |
| Block, Michelle | MS, BS, RAC,<br>CIP | Non-Scientist | Regulatory/DoD<br>Regulated Research | Y | | Α | Y | |
| Blum, Robert | PharmD | Other Scientist | Pharmacology | N | Chair | Α | N | |
| Bode, Kate | BS | Non-Scientist | Regulatory | Y | | Α | N | |
| Booker, Burthia | PhD | Other Scientist | Biomedical Sciences | N | | Α | N | |
| Borgatta, Lynn | MD, MPH | Physician<br>Scientist | Obstetrics/ Gynecology | N | | Α | Y | |
| Bottorff, Michael | PharmD | Other Scientist | Pharmacology | N | | Α | N | |
| Braun, Peter | MD | Physician<br>Scientist | Internal Medicine/<br>Infectious Disease | N | | Α | N | |
| Brown, Janice | RPh, MLS | Non-Scientist | Educator/ Librarian | N | | Α | N | |
| Brzozowski, Jane | MS, BS | Non-Scientist | Patient Advocacy | N | | Α | N | |
| Burkey, Madison | BSN, RN, OCN | Other Scientist | Nursing/ Oncology | Υ | | Α | Υ | |
| Byers, Derek | MD, PhD, FCCP | Physician<br>Scientist | Internal Medicine/<br>Immunology | N | | Α | N | |





| Name | Credentials | Role | Primary Expertise | Affiliated? | Chair? | Primary(P) or<br>Alternate(A)? | Reviews<br>CAN<br>Research? | CAN:<br>Knowledgeable<br>in ethics and/or<br>law? |
|---|---|---|---|---|---|---|---|---|
| Campbell, Laura | MD | Physician<br>Scientist | Oncology/ Hematology/<br>Pediatrics/ Bioethics | N | | Α | N | |
| Carr, Raymond | RPh | Other Scientist | Pharmacist | N | | Α | N | |
| Cavagnaro, Joy | PhD, DABT, RAC | Other Scientist | Toxicology/ Regulatory<br>Affairs Consultant | N | | Р | N | |
| Cesary, Kelly | MSN, APN, ANP-<br>BC, AOCNP | Other Scientist | Oncology / Hematology / Nursing | N | | Α | N | |
| Chukwu, Bernadette | PharmD | Other Scientist | Pharmacovigilance/<br>Drug Safety | Y | | Α | N | |
| Cooper, Kindra | JD | Non-Scientist | Legal | N | | Α | N | |
| Cooper, Phyllis | RN, BSN, OCN,<br>CCRP | Other Scientist | Nursing/ Oncology | N | | Α | N | |
| Cosentino, Lidia | PhD | Other Scientist | Biology/ Protocol development | N | | Α | Y | |
| Cram, Gary | AS | Non-Scientist | Ethics | N | | Α | N | |
| Cullity, Connie | MD, MPH | Physician<br>Scientist | FDA Regulations | Y | | Α | N | |
| <b>Cummings, Theresa</b> | RN, MS | Other Scientist | Nursing/ Public Health | N | | Α | N | |
| Davidson, Barbara | MS, RN, MSN,<br>CCRC | Other Scientist | Community Health<br>Nursing | Y | | Α | Y | |
| Davidson, Susan | MD | Physician<br>Scientist | Infectious Disease/<br>Homeostasis | N | | Α | N | |
| Davis, Hannah | BS, MS | Other Scientist | Biology / Biomedical | Υ | | Α | N | |
| Desai, Pankaj | PhD | Other Scientist | Biopharmaceutics/<br>Pharmacokinetics | N | | Α | N | |
| Dorsch, Kimberly | BS | Other Scientist | Stem Cell/ Tissue<br>Research | N | | Α | N | |
| Drada, Denisse | | Non-Scientist | Regulatory | Υ | | Α | Υ | |
| Duhon, Bryson | PharmD, BCPS | Other Scientist | Pharmacology | N | | Α | N | |
| Dyson, Maynard | MD, MA, CIP | Physician<br>Scientist | Pediatrician/<br>Pulmonology | N | | Α | N | |







| Name | Credentials | Role | Primary Expertise | Affiliated? | Chair? | Primary(P) or<br>Alternate(A)? | Reviews<br>CAN<br>Research? | CAN:<br>Knowledgeable<br>in ethics and/or<br>law? |
|---|---|---|---|---|---|---|---|---|
| Ebert, Susan | MS, CIP | Non-Scientist | Regulatory | Υ | Sr.<br>Chair<br>Dir. | Р | N | |
| Fernicola, Daniel | MD, FACC | Physician<br>Scientist | Cardiology | N | | Α | N | |
| Ferrell, David | ThB, BA, MA | Non-Scientist | Religion / Ethics | N | | Α | Y | Ethics |
| Fittizzi, Cheryl | RN, CIM, CIP | Other Scientist | Nursing/ Emergency<br>Trauma/ Public Health | N | | Α | N | |
| Fitzgerald, Michael | PhD | Other Scientist | Social Psychology | N | | Α | N | |
| Fleck, David | PhD | Other Scientist | Psychiatry/ Behavioral<br>Neuroscience | N | | Α | N | |
| Flowers, Janelle | MEd | Non-Scientist | Guidance Counselor | N | | Α | N | |
| Foster, Joyce | MS | Non-Scientist | Family Therapy | N | | Α | N | |
| Garrick, Tania | RN, BScN, MA | Other Scientist | Nursing | N | | Α | Υ | |
| Gelinas, Luke | PhD, MAR, AB | Non-Scientist | Ethics | Υ | Sr.<br>Chair<br>Dir. | Р | Y | Ethics |
| Georgiadis, Nina | MD | Physician<br>Scientist | Neonatal Intensive<br>Care | N | | Α | Υ | |
| Ginnings, Susan | RPh | Other Scientist | Pharmacist | N | | Α | N | |
| Gold, Herschel | BA, LLB | Non-scientist | Legal | N | | Α | Υ | Ethics, Law |
| Goldman, Ran | MD, MHA,<br>FRCPC | Physician<br>Scientist | Pediatrician | N | Chair | Α | Υ | Ethics |
| Gonzales, Yury | MD, FACP | Physician<br>Scientist | Internal Medicine | N | | Р | Y | |
| Gordner, Linda | BA | Non-Scientist | Special Education | N | | Α | Υ | |
| Gorman, Richard | MD | Physician<br>Scientist | Pediatrics / Infectious<br>Diseases | N | | Α | N | |
| Gottke, Melissa | BA | Non-Scientist | Regulatory | Υ | | Α | Υ | |
| Gray, Vernon | PhD | Non-Scientist | County Government<br>Administrator | N | | Α | N | |
| Grimes, Brittany | MS | Non-Scientist | Regulatory | Υ | | Α | Υ | |

1, 2023 d 21044 4G 0A5 4 of 11





| Name | Credentials | Role | Primary Expertise | Affiliated? | Chair? | Primary(P) or<br>Alternate(A)? | Reviews<br>CAN<br>Research? | CAN:<br>Knowledgeable<br>in ethics and/or<br>law? |
|---|---|---|---|---|---|---|---|---|
| Groisman, Iris | PhD | Other Scientist | Biochemistry/<br>Radiobiology/<br>Pharmacogenetics | N | | А | Y | Ethics |
| Group, Melinda | BS, RPh | Other Scientist | Pharmacist/ Hospital<br>Research | N | | Р | N | |
| Groza, Florina | MSc | Other Scientist | Biochemistry | Y | | Α | Y | |
| Haffizulla, Farzanna | MD, FACP,<br>FAMWA | Physician<br>Scientist | Internal Medicine | N | | Р | N | |
| Hensler, Carolyn | BS | Non-Scientist | Regulatory | N | | Α | N | |
| Henson, Tricia | BA, RN | Other Scientist | Nursing Sciences | Υ | | Α | Υ | |
| Hewes, Julia | MPH, BSN, RN,<br>OCN | Other Scientist | Nursing/ Oncology | N | | Α | N | |
| Hierholzer, Robert | MD | Physician<br>Scientist | Psychiatrist | N | | Α | N | |
| Higley, Amanda | PhD, CIP | Other Scientist | Psychology | Υ | Chair | Α | N | |
| Hill, Margaret | RN, MS | Other Scientist | Nursing/ Oncology/<br>Clinical Trials Research | N | | Α | N | |
| Hiller, David | BSN, RN, AEMT,<br>CIP | Other Scientist | Regulatory Critical Care<br>Nursing | Υ | Chair | Α | N | |
| Horton, Alicia | JD, MPH | Non-Scientist | Legal/ Public Health | N | | Α | N | |
| Hoshower, Jason | BS, CIP | Non-Scientist | Regulatory | Υ | | Α | Υ | |
| Houser, Patricia | MD | Physician<br>Scientist | Family Medicine | N | | Α | N | |
| Hsiao, Karin | BS, MS, MBA | Other Scientist | Biomedical<br>Engineering/ Device | N | | Α | N | |
| Hubbard, Tyler | MA, CIP | Non-Scientist | Social and Behavioral<br>Research / Regulatory | Υ | | Α | N | |
| Jacobsen, Eric | MD | Physician<br>Scientist | Oncology/ Lymphoma | N | | Α | N | |
| Johnson, Dena | BS, MEd, CCRP,<br>CIP | Non-Scientist | Regulatory | Υ | Chair | Α | N | |







| Name | Credentials | Role | Primary Expertise | Affiliated? | Chair? | Primary(P) or<br>Alternate(A)? | Reviews<br>CAN<br>Research? | CAN:<br>Knowledgeable<br>in ethics and/or<br>law? |
|---|---|---|---|---|---|---|---|---|
| Jordan, William | DO | Physician<br>Scientist | Oncology/ Medical | N | | Α | N | |
| Kaul, Neha | MA, MS, BSc | Other Scientist | Social and Behavioral<br>Research; Regulatory;<br>Bioethics/Ethics;<br>Molecular Biology | Y | Chair | А | N | |
| Keely, Levering | BSN, MPA | Other Scientist | Nursing/ Device specialist | N | | Α | N | |
| Kim, James | MD, MBA | Physician<br>Scientist | General Practice/ Non-<br>Cancer Pain<br>Management | N | | Α | Y | |
| Kirk, Julia | BA, CIP | Non-Scientist | Regulatory | Y | | Α | Y | |
| Klaff, Ali | BSCIP | Non-Scientist | Regulatory | Υ | | Α | Υ | |
| Knopman, David | MD | Physician<br>Scientist | Alzheimer/ Neurology | N | | Α | N | |
| Kopec, Frederick | JD | Non-Scientist | Legal | N | Chair | Α | N | |
| Kronish, Daniel | MD | Physician<br>Scientist | Oncology/ Pediatrician | Y | Chair | Α | Y | |
| Kuebler, Philip | MD, PhD, BS | Physician<br>Scientist | Internal Medicine/<br>Oncology/ Hematology | N | | Α | N | |
| Kuzmanovic, Dario | BA, MHSc, CRA,<br>CHRC | Non-Scientist | Bioethics | N | | Α | Υ | Ethics, Law |
| Kysela, Kathleen | CIP | Non-Scientist | Regulatory | Υ | | Α | Υ | |
| LaCount, Peter | MHS, MEd | Non-Scientist | Compliance Director | N | | Р | N | |
| Lawrence, Janice | PhD, MA, BA,<br>BPE | Other Scientist | Physical Ed/ Life Coach | N | | Α | Y | |
| Leduc, Lucie | LLM | Non-Scientist | Legal/ Ethics | N | | Α | Υ | Ethics, Law |
| Leo, Jessica | AA, CIP | Non-Scientist | Regulatory | Υ | | Α | Υ | |
| Letko, Erik | MD | Physician<br>Scientist | Ophthalmology/<br>Surgery | N | | Α | N | |
| Lettman, Robert | BA, MBA, JD, PA | Non-Scientist | Legal | N | | Α | N | |
| Lind, Alecia | BS, CIP | Non-Scientist | Regulatory | Υ | | Α | Y | |

A





| Name | Credentials | Role | Primary Expertise | Affiliated? | Chair? | Primary(P) or<br>Alternate(A)? | Reviews<br>CAN<br>Research? | CAN:<br>Knowledgeable<br>in ethics and/or<br>law? |
|---|---|---|---|---|---|---|---|---|
| Longstaff, Holly | PhD | Non-Scientist | Ethics | N | | Α | Υ | Ethics |
| Lopez, Bennie | MBA | Non-Scientist | Educator | N | | Α | N | |
| Lossada, Mery | MD, PA | Physician<br>Scientist | Psychiatry/ Neurology | N | | Α | N | |
| Maloof, Damiana | MSN, RN, OCN | Other Scientist | Nursing/ Oncology | N | | Α | N | |
| Martin, Christopher | PharmD, MS | Other Scientist | Pharmacology | N | Chair | Α | N | |
| McPhillips, Joseph | PhD | Other Scientist | Clinical Research<br>Consultant | N | | Α | N | |
| Mensah, Sharon | MS | Other Scientist | Biological Sciences/<br>Clinical Research | N | | Α | N | |
| Mihalov, Linda | MD, FACOG | Physician<br>Scientist | Oncology/ Gynecology | N | | Α | N | |
| Mitchell, Cameron | BA | Non-Scientist | Regulatory | Υ | Chair | Α | Υ | |
| Morse, Linda | RN, MSN, OCN | Other Scientist | Nursing/ Oncology | N | | Α | N | |
| Mueller, Lava | MEd, MDiv | Non-scientist | Chaplain | N | | Α | N | |
| Munk, Gary | PhD, MS, BS | Other Scientist | Virology/ Biosafety | N | | Α | N | |
| Nattrass, Susan | OC, PhD, CBDT | Other Scientist | Osteoporosis and<br>Women's Health | N | | Α | Y | |
| Neff, Robert | BS | Non-Scientist | Mobile Medical | N | | Α | N | |
| Nolan, Joseph | PhD, MS, MA,<br>BA, BS | Other Scientist | Statistics | N | | Α | N | |
| Noss, Michael | MD | Physician<br>Scientist | Family Medicine | N | | Α | N | |
| O'Connell, Mary | | Non-Scientist | Regulatory | N | | Α | N | |
| Odor, Erin | MA, CIP | Non-Scientist | Regulatory | Υ | Chair | Α | N | |
| O'Leary, Maura | MD | Physician<br>Scientist | Oncology/ Pediatrician/<br>Hematology | N | | Α | N | |
| Oliver, Ayesha | BS | Non-Scientist | Regulatory | Υ | | Α | Υ | |
| Ott, Carl | MD, MPH | Physician<br>Scientist | Internal Medicine | N | | Α | N | |
| Parker, R. Lamar | MD, FACOG, CPI | Physician<br>Scientist | Obstetrics/ Gynecology | N | | Α | N | |





| Name | Credentials | Role | Primary Expertise | Affiliated? | Chair? | Primary(P) or<br>Alternate(A)? | Reviews<br>CAN<br>Research? | CAN:<br>Knowledgeable<br>in ethics and/or<br>law? |
|---|---|---|---|---|---|---|---|---|
| Patrick, Kyle | DO | Physician<br>Scientist | Medical Research | N | | Α | N | |
| Pfeiffer, Matthew | PhD | Other Scientist | Pharmacology/<br>Toxicology | N | | Α | N | |
| Popovici-Toma, Dan | MD | Physician<br>Scientist | Medical Advisor | N | | Α | Y | Ethics |
| Povar, Gail | MD, MPH, FACP | Physician<br>Scientist | Internal Medicine | N | Chair | Α | N | |
| Psenicka, Eva | BSc | Non-Scientist | Physiology/ Regulatory | N | | Α | Υ | |
| Ramjiawan, Bram | PhD | Other Scientist | Pharmacology | N | | Α | Υ | |
| Randolph, Robert | DMin | Non-Scientist | Chaplain | N | | Α | N | |
| Razzetti, Albert | MD | Physician<br>Scientist | Internal Medicine/<br>Pulmonology | N | | Α | N | |
| Reddish, Mitchell | PhD | Non-Scientist | Professor/ Religious<br>Studies/ Ethicist | N | | Α | N | |
| Renner, Laura | BA | Non-Scientist | Regulatory | Y | | Α | N | |
| Rewers, Mae, Edna | MS, JD, MBA | Non-Scientist | Legal/ Healthcare/<br>Research Compliance | N | | Α | N | |
| Reynolds, Deborah | RN, OCN | Other Scientist | Nursing/ Oncology | N | | Α | N | |
| Robinson, Deana | MPH, BS, LPN,<br>CPhT | Other Scientist | Clinical Research LPN | Υ | | Α | Y | |
| Robinson, Richard | MD | Physician<br>Scientist | Medical Oncology/<br>Internal Medicine | N | | Α | N | |
| Romain, Michael | MD | Physician<br>Scientist | Internal Medicine | N | | Α | N | |
| Romanchuk, Robert | BSHS, CIP,<br>CCRCP | Other Scientist | Clinical Research<br>Administration/<br>Respiratory Therapy | N | | Α | Υ | |
| Rush, Jason | BS, CIP | Non-Scientist | Regulatory | Υ | | Α | N | |
| Ruwart, Mary | PhD, BS | Other Scientist | Biophysics/<br>Biochemistry | N | | Α | N | |







| Name | Credentials | Role | Primary Expertise | Affiliated? | Chair? | Primary(P) or<br>Alternate(A)? | Reviews<br>CAN<br>Research? | CAN:<br>Knowledgeable<br>in ethics and/or<br>law? |
|---|---|---|---|---|---|---|---|---|
| Ryan, Laurajo | PharmD, MSc,<br>BCPS | Other Scientist | Pharmacology | N | | Α | N | |
| Sadorra, Carol | PhD | Non-Scientist | Regulatory | Y | | Α | Y | |
| Salama, Suzette | BPharm, MSc,<br>PhD | Other Scientist | Ethicist/ Pharmacology | N | | Α | Y | Ethics, Law |
| Saylor, Brenda | RN, BSN, ARM | Other Scientist | Community Health<br>Nursing | Y | | Α | Y | |
| Selsky, Clifford | PhD, MD | Physician<br>Scientist | Pediatrics, Hematology<br>Oncology | N | | Α | N | |
| Shafer, Michaela | PhD, RN | Other Scientist | Biomedical Research/<br>Nursing | N | | Α | N | |
| Sheedy, Carmen | BA | Non-Scientist | Regulatory | Υ | | Α | Υ | |
| Shulman, Mitchell | MDCM, FRCPC,<br>CSPQ | Physician<br>Scientist | Emergency Medicine | N | | Α | Y | |
| Siegmann, Glenn | MS, RPh | Other Scientist | Pharmacist | N | | Α | N | |
| Singh, Sukhbir | MD, MBA | Physician<br>Scientist | Psychiatry Research | Υ | Chair | Α | N | |
| Skroback, Judith | BM | Other Scientist | Devices | Υ | | Α | Υ | |
| Somerstein, Shari | RPh | Other Scientist | Pharmacist | N | | Α | N | |
| Sommer, Dane | DMin, MDiv, BCC | Non-Scientist | Ministry | N | | Α | N | |
| Spaulding, Trevor | BA, CIP | Non-Scientist | Regulatory | Υ | | Α | Υ | |
| Stoltz, Randall | MD, CPI | Physician<br>Scientist | Phase I Research/<br>Cardiovascular | N | | Α | N | |
| Stone, Kurt | DD | Non-Scientist | Ministry | N | | Α | N | |
| Strull, William | MD | Physician<br>Scientist | Internal Medicine | N | | Α | N | |
| Taucher, Kate | PharmD, MHA,<br>BCOP | Other Scientist | Pharmacology | N | | Α | N | |
| Teal, Marilyn | PharmD, BS | Other Scientist | Pharmacology | N | | Р | Υ | Ethics |
| Tillman, Beverly | RN, MSN | Other Scientist | Public Health | N | | Α | N | |
| Tkaczuk, Katherine | MD | Physician<br>Scientist | Oncology/ Hematology | N | | Α | N | |

A





| Name | Credentials | Role | Primary Expertise | Affiliated? | Chair? | Primary(P) or<br>Alternate(A)? | Reviews<br>CAN<br>Research? | Knowledgeable<br>in ethics and/or<br>law? |
|---|---|---|---|---|---|---|---|---|
| Vanderwel, Marianne | MEng, MSc | Other Scientist | Quality Assurance/<br>Research Ethics | N | | Α | Y | Ethics, Law |
| Vernon, Kim | JD | Non-Scientist | Legal/ Prisoner<br>Advocate | N | | Α | N | |
| Walker, Christina | MD | Physician<br>Scientist | Family Medicine | N | | Α | N | |
| Way, Cynthia | CIP | Non-Scientist | Regulatory/ Phase I<br>Research | N | | Α | N | |
| Wells, Christine | MD | Physician<br>Scientist | Neurology/ Patient<br>Advocate | N | | Α | Y | Ethics |
| Westby, Christian | PhD | Other Scientist | Physiology | Y | Chair | Р | N | |
| Witkowski, Amy | CIP | Non-Scientist | IRB Professional | N | | Α | N | |
| Wood, Leslie | BA | Non-scientist | Communications | N | | Α | Υ | Ethics |
| Wright-Moore,<br>Conschetta | RN, MPH | Other Scientist | Nursing/ Clinical<br>Research | Y | | Α | Y | |







# **Roster Changes:**

| Member Name | Change | Date Change Made |
|------------------|-------------------------|------------------|
| Cheri Pettey | Removed | 11/01/2023 |
| Cyrus Gill | Removed | 11/02/2023 |
| Jennifer Brock | Removed | 11/15/2023 |
| Kelly Cesary | Added | 11/16/2023 |
| Kate Bode | Added | 11/22/2023 |
| Cameron Mitchell | Added Chair designation | 11/27/2023 |
| Hallie Barr | Added | 11/28/2023 |

# INFORMED CONSENT FORM AND

#### AUTHORIZATION TO USE AND DISCLOSE PROTECTED HEALTH INFORMATION

Sponsor / Study Title: Mindset Medical, LLC / "A Multi-Center Prospective Open

Label Study of a Web-based Application for Pulse Rate in Adult

Patients"

Protocol Number: IVC-400-006

**Principal Investigator:** 

(Study Doctor)

«PiFullName»

Telephone: «IcfPhoneNumber»

Address: «PiLocations»

#### **KEY INFORMATION**

You are invited to take part in a research study. This research study is designed to evaluate the accuracy of Informed Vital Core (IVC App, IVC), a web-based application designed for measurements of vital signs including pulse rate (PR). Your Investigator will explain the clinical study to you. Clinical studies include only people who choose to take part voluntarily, after considering all the information in this document. Please take your time to make your decisions about taking part.

Clinical studies help us improve and grow our knowledge on the safety and effectiveness of investigational devices. For this reason, the law requires that investigational devices must be clinically tested. As required by law, this clinical study has been reviewed by an Institution Review Board, (IRB) and the United States Food and Drug Administration (FDA). This clinical study will be conducted in the United Sates. The clinical study is being investigated, organized, and financed by Mindset Medical, LLC.

Your participation in this clinical study is voluntary. Therefore, you will only be included in the clinical study if you give your written consent. You may choose to not participate, or you may withdraw from the study for any reason without penalty or loss of benefits to which you are otherwise entitled and without any effect on your future medical care. The Investigator or the sponsor can stop your participation at any time without your consent for the following reasons:

- If you fail to follow directions for participating in the study;
- If it is discovered that you do not meet the study requirements;
- If the study is canceled; or
- For administrative reasons.

Please do not hesitate to discuss questions with your Investigator. Afterward, you will be given plenty of time to think about whether you wish to take part in this study before you will be asked to decide.

#### WHY IS THE CLINCIAL STUDY BEING CONDUCTED?

The clinical study involves research. The objective of this study is to evaluate the investigational software (IVC APP, IVC) as a simple and non-invasive way to measure vital signs. This is a research study to test a new software application detecting Pulse Rate (PR). This study will compare the PR measurement using the IVC App to the heart rate (HR) measured by an electrocardiogram (ECG) device (reference device).

It is hypothesized that the accuracy of the IVC App is non-inferior to the accuracy of an FDA-cleared/approved vital sign monitoring device (reference device). This research is to evaluate the accuracy of measurement for each Pulse Rate vital sign with the IVC App, compared to appropriate reference devices.

You are being asked to participate in this research study because you are between the ages of 22-85.

#### WHAT INFORMATION WILL BE COLLECTED AND USED FOR THIS STUDY?

The study staff working on the study will collect information about you. This includes your health information.

Data collected will be entered into the electronic data capture (EDC) system and used for analysis.

The following data will be collected:

- Date of Birth/Age
- Gender
- Ethnicity
- Skin Tone as rated by the Fitzpatrick Scale
- Facial variables (glasses, facial hair, facial tattoos, and/or makeup)
- Cardiac Medical History
- Chronic Medical Conditions
- Pulse Rate taken by IVC App (conducted twice)
- Heart Rate taken by ECG (conducted twice)

In the future, we may publish results of this study in scientific journals and may present it at scientific meetings. If we do, we will not identify you. Only summarized data from the entire study will be presented.

If the researchers learn about potential serious harm to you or someone else or other public health concerns, it will be shared with the appropriate authorities.
#### HOW MANY PEOPE WILL TAKE PART IN THE STUDY?

About 85 people will take part in the study.

The study will recruit volunteers from clinics, hospitals, and the general public.

#### WHAT WILL HAPPEN IF I TAKE PART IN THIS RESEARCH STUDY?

If you decide to take part in the clinical study, you will complete the entire study today.

The duration of the study is one day.

Table 1 – Overview of study activities/visit schedules

| | Screening /Baseline Day 1 |
|---|---|
| Study Visit/Day | Visit 1 |
| Informed Consent | X |
| Eligibility | X |
| Demographics | X |
| Fitzpatrick Scale Assignment** | X |
| Medical History | X |
| Concomitant Medication (medications you are taking) | X |
| Adverse Event Form (If applicable) | X |
| Pulse Rate (IVC)* | X |
| ECG (reference device)* | X |

<sup>\*</sup>The collection of pulse rate from the IVC App and HR from ECG reference device should be taken twice for all subjects.

During this one visit you will be asked to read and sign this informed consent form prior to participating in any study-related activities. After you have provided your consent for study participation, you will be asked a series of questions related to your eligibility into this study, demographic, relevant medical history, and relevant medications. You will also be visually evaluated by the Investigator for your skin type, using the Fitzpatrick Classification Scale for Skin Types. One image of your face will be captured to be used by the Sponsor to evaluate lighting, environmental conditions, and your Fitzpatrick Classification Scale Skin Type. All the information will be collected and used for evaluation purposes at the end of the study and will not contain any Protected Health Information (PHI).

You will not be able to wear a mask or bandage that obstructs your forehead, cheeks, or chin. You will need to agree to remove makeup, sunscreen, lotion, clothing, or items obstructing the face for the duration of the measurement. You will also need to be able to remain still for 60 seconds at a time.

You will be attached to an ECG device using 3 disposable tab electrodes attached to the inside of your left forearm, the inside of your right forearm, and just above the inside of the left ankle

<sup>\*\*</sup>Investigator to perform

to read the ECG results. At the same time you will be asked to sit still for one minute looking at the phone in the stand while the IVC App takes measurements of your face.

You will then be asked if there were any adverse events (side effects) that you experienced while in the study.

#### **HOW LONG WILL I BE IN THIS STUDY?**

Your participation in this study is less than one hour unless there is a technical issue encountered, in which case you will be asked to come back and complete the visit if the study is still enrolling subjects.

#### WHAT SIDE EFFECTS OR RISKS CAN I EXPECT FROM BEING IN THE STUDY?

There are no foreseeable risks or known side effects to this study.

There may be slight discomfort from remaining still for 1 minute.

Skin irritation is rare but could occur during an ECG from the electrodes or gel that is used.

You will have photographs of your face taken for this study. It is possible that your face may be recognizable and your identity may be known.

#### **UNFORESEEN RISKS**

Since the study is using investigational software, there may be other risks that are unknown but it is highly unlikely.

#### ARE THERE BENEFITES TO TAKING PART IN THE STUDY?

This study is for research purposes only. There is no direct benefit to you from your participation in the study. Information learned from the study may help other people in the future.

Since the IVC App is a web-based application, it can easily be utilized at hospitals (replacing vital signs carts), physician offices, clinics, and at patient's homes without the need for a trained nurse to capture the vitals. The IVC App can easily be utilized at a patient's home without the need to purchase specialized equipment.

Traditional pulse rate devices rely on physical contact of a patient, either placed on a wrist, arm, fingertip, or some other part of the body. This IVC App does not require any physical contact of a patient, rather they will simply look directly into the camera embedded on the phone device.

#### **ALTERNATIVES**

This research study is for research purposes only. The only alternative is to not participate in this study.

#### COMPENSATION FOR PARTICIPATION

#### «Compensation»

You will be paid up to a total of \$75.00 if you complete this study. If you have any questions regarding your compensation for participation, please contact the study staff.

#### CONFIDENTIALITY

Records of your participation in this study will be held confidential except when sharing the information is required by law or as described in this informed consent. The Investigator, the sponsor or persons working on behalf of the sponsor, and under certain circumstances, the United States Food and Drug Administration (FDA) and the Institutional Review Board (IRB) will be able to inspect and copy confidential study-related records which identify you by name. This means that absolute confidentiality cannot be guaranteed. If the results of this study are published or presented at meetings, you will not be identified.

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

To make sure that the health information collected in this study is accurate, it will need to be checked from time to time against your medical records. Some persons may need to see these records in order to monitor the research and verify the accuracy of the study data, including:

- A limited number of representatives from the study sponsoring company (namely its monitors and auditors),
- The institutional review board Advarra IRB (an independent committee that reviewed the aspects of this study to help protect the rights and welfare of study subjects),
- Government regulatory authorities including, the US Food and Drug Administration (FDA) and other foreign regulatory agencies.

Your study records including confidential information about you collected during the study will be kept at a secure location.

While every effort will be made to protect the privacy of your information, absolute confidentiality cannot be guaranteed. This does not limit the duty of the researchers and others to protect your privacy.

By signing this information and consent form, you consent to the collection, access, use and disclosure of your information as described above.

#### **COMPENSATION FOR INJURY**

If you become ill or are injured while you are in the study, get the medical care that you need right away. You should inform the healthcare professional treating you that you are

participating in this study. If you tell the study staff that you think you have been injured, then they will help you get the care you need.

If you are injured as a result from procedures done for the purpose of this study, the sponsor will pay for those medical expenses necessary to treat your injury that are not covered by your medical insurance or any other third-party coverage. By signing this document, you will not lose any of your legal rights or release anyone involved in the research from responsibility for mistakes.

To pay medical expenses, the sponsor will need to know some information about you like your name, date of birth, and Medicare Beneficiary Identifier (MBI). This is because the sponsor has to check to see if you receive Medicare and if you do, report the payment it makes to Medicare.

#### **COSTS**

There will be no charge to you for your participation in this study. The study device, study-related procedures, and study visit will be provided at no charge to you or your insurance company.

#### WHOM TO CONTACT ABOUT THIS STUDY

During the study, if you experience any medical problems, suffer a research-related injury, or have questions, concerns, or complaints about the study such as:

- Whom to contact in the case of a research-related injury or illness;
- Payment or compensation for being in the study, if any;
- Your responsibilities as a research subject;
- Eligibility to participate in the study;
- The Investigator's or study site's decision to withdraw you from participation;
- Results of tests and/or procedures;

# <u>Please contact the Investigator at the telephone number listed on the first page of this consent document.</u>

If you seek emergency care, or hospitalization is required, alert the treating physician that you are participating in this research study.

An institutional review board (IRB) is an independent committee established to help protect the rights of research subjects. If you have any questions about your rights as a research subject, contact:

#### By <u>mail</u>:

Study Subject Adviser Advarra IRB 6100 Merriweather Dr., Suite 600 Columbia, MD 21044

• or call **toll free**: 877-992-4724

• or by <u>email</u>: <u>adviser@advarra.com</u>

Please reference the following number when contacting the Study Subject Adviser: Pro00070500.

#### PRIMARY HEALTH CARE PROVIDER NOTIFICATION OPTION

**TYES** (If yes, please complete the information below)

I consent to having my family doctor or primary health care provider notified by the study site of my participation in this study and/or any significant findings related to my health (please check yes or no).

| Name and address of family | Name: |
|-------------------------------|----------|
| doctor or primary health care | Address: |
| provider: | |
| Talanhana and Fay Number | Tel: |
| Telephone and Fax Number: | Fax: |

□NO

#### **CONSENT**

I have read and understand the information in this informed consent document. I have had an opportunity to ask questions and all of my questions have been answered to my satisfaction. I voluntarily agree to participate in this study until I decide otherwise. I do not give up any of my legal rights by signing this consent document. I will receive a copy of this signed consent document.

| Subject's Printed Name | |
|--------------------------------------------------------------|----------|
| Subject's Signature | <br>Date |
| Printed Name of the Person Conducting the Consent Discussion | |
| Signature of the Person Conducting the Consent Discussion | Date |

#### CONSENT FOR OPTIONAL SUBSTUDY

You are also being asked to participate in an optional substudy.

"Informed Vital Core, Data Collection Protocol (Respiratory Rate, Pulse Oxygen Saturation, and Blood Pressure)" is the substudy.

If you leave the substudy for any reason, the Investigator may ask you to have some end-of-study tests for your safety (for example, if you have experienced any adverse or serious adverse events while participating in the substudy.

## WHY IS THE CLINICAL SUBSTUDY BEING CONDUCTED?

The scope of this substudy is to gather data from an FDA approved device called the Masimo MightySat Rx Fingertip Pulse Oximeter and/or Caretaker Vital Stream continuous blood pressure device) while gathering real-time environmental images to improve the measurement of pulse rate (PR), respiratory rate (RR), blood oxygen saturation (SpO2), and blood pressure (BP) for the purpose of training the algorithms of the IVC App.

You will be asked to provide four measurements of either SpO2 or blood pressure. You may be asked to do four measurements of one or the other, or a combination of two sessions of each, etc.

You will be asked to sit for 120 seconds while the IVC App takes continuous photos of your face and/or fingertip while you wear the reference device.

#### WHAT INFORMATION WILL BE COLLECTED AND USED FOR THIS SUBSTUDY?

- Sex
- Race
- Ethnicity
- Skin Tone as rated by the Fitzpatrick Scale
- Age
- Height/Weight
- Facial variables (glasses, facial hear, facial tattoos, and/ or makeup)
- Permission to collect photos. You will be asked to sit for 120 seconds while the IVC APP takes continuous photos of your face and/ or fingertip.
- Pulse Rate, Respiratory rate, SpO2, and Blood Pressure

#### **RISKS**

You will have photographs of your face taken for this substudy. It is possible that your face may be recognizable and your identity may be known.

There may be other risks that are unknown.

#### **BENEFITS**

This substudy is for research purposes only. There is no direct benefit to you from your participation in the substudy. Information learned from the substudy may help other people in the future.

#### **ALTERNATIVES**

This research substudy is for research purposes only. The only alternative is to not participate in this substudy.

#### CONFIDENTIALITY

Records of your participation in this study will be held confidential except when sharing the information is required by law or as described in this informed consent. The Investigator, the sponsor or persons working on behalf of the sponsor, and under certain circumstances, the United States Food and Drug Administration (FDA) and the Institutional Review Board (IRB) will be able to inspect and copy confidential study-related records which identify you by name. This means that absolute confidentiality cannot be guaranteed. If the results of this study are published or presented at meetings, you will not be identified.

#### **COMPENSATION FOR INJURY**

If you become ill or are injured while you are in the substudy, get the medical care that you need right away. You should inform the healthcare professional treating you that you are participating in this substudy. If you tell the study staff that you think you have been injured then they will help you get the care you need.

If you are injured as a result of procedures done for the purpose of this substudy, the sponsor will pay for those medical expenses necessary to treat your injury that are not covered by your medical insurance or any other third-party coverage. By signing this document, you will not lose any of your legal rights or release anyone involved in the research from responsibility for mistakes.

To pay medical expenses, the sponsor will need to know some information about you like your name, date of birth, and Medicare Beneficiary Identifier (MBI). This is because the sponsor has to check to see if you receive Medicare and if you do, report the payment it makes to Medicare.

### **COMPENSATION FOR PARTICIPATION**

«Compensation»

You will be paid up to a total of \$75.00 for 4 data collection sessions if you complete this substudy.

If you have any questions regarding your compensation for participation, please contact the study staff.

There will be no charge to you for your participation in this substudy.

You may decide not to participate in the optional substudy or you may choose to withdraw from the substudy for any reason. If you decide not to participate in the substudy, your decision will have no impact on your ability to participate in the initial study and will have no impact on any other benefits to which you would otherwise be entitled.

The Investigator or the sponsor can stop your participation at any time without your consent for the following reasons:

- If you fail to follow directions for participating in the study;
- If it is discovered that you do not meet the study requirements;
- If the study is canceled; or
- For administrative reasons.

Please indicate your preference below:

| ☐YES (initials) I agree to participate in the substudy described above. | |
|---|---|
| □NO (initials) I do not agree to participa | ate in the substudy described above |
| Subject's Printed Name | |
| Subject's Signature | <br>Date |
| Printed Name of the Person Conducting the Consent Discussion | |
| Signature of the Person Conducting the Consent Discussion | <br>Date |

### **AUTHORIZATION TO USE AND DISCLOSE PROTECTED HEALTH INFORMATION**

If you decide to be in this study, the Investigator and study staff will use and share health data about you to conduct the study. Health data may include:

- Your name
- Address
- Phone number
- Date of birth
- Medical history
- Information from your study visits, including all test results

Health data may come from your study records or from existing records kept by your doctor or other health care workers.

For this study, the study staff may share health data about you with authorized users. Authorized users may include:

- Representatives of Mindset Medical, LLC
- Representatives of Total Clinical Trial Management (TOTAL CRO)
- Representatives of Advarra IRB (an Institutional Review Board that reviews this study)
- The Food and Drug Administration (FDA) and other US federal and state agencies
- Government agencies to whom certain diseases (like HIV, hepatitis, and STDs) must be reported
- Governmental agencies of other countries
- Outside individuals and companies, such as laboratories and data storage companies, that work with the researchers and sponsor and need to access your information to conduct this study
- Other research doctors and medical centers participating in this study, if applicable

Your health data will be used to conduct and oversee the research, including for instance:

- To see if the study device/Software works and is safe
- To compare the study device/Software to other devices/Software
- For other research activities related to the study device/Software

Once your health data has been shared with authorized users, it may no longer be protected by federal privacy law and could possibly be used or disclosed in ways other than those listed here.

Your permission to use and share health data about you will end in 50 years unless you revoke it (take it back) sooner.

You may revoke (take back) your permission to use and share health data about you at any time by writing to the Investigator at the address listed on the first page of this form. If you do this, you will not be able to stay in this study. No new health data that identifies you will be gathered after your written request is received. However, health data about you that has already been gathered may still be used and given to others as described in this form.

Your right to access your health data in the study records will be suspended during the study to keep from changing the study results. When the study is over, you can access your study health data from your doctor.

If you decide not to sign this form, you will not be able to take part in the study.

#### STATEMENT OF AUTHORIZATION

I have read this form and its contents were explained. My questions have been answered. I voluntarily agree to allow study staff to collect, use and share my health data as specified in this form. I will receive a signed and dated copy of this form for my records. I am not giving up any of my legal rights by signing this form.

| Printed Name of Subject | |
|-------------------------|------|
| Signature of Subject | Date |

| No. | Site Name | PI Name | Staff | Credentials | Phone # | Role | Address | City | State | Zip Code |
|---|---|---|---|---|---|---|---|---|---|---|
| 301 | Velocity Clinical Research | Gregg Lucksinger | Victor Haas | BS, GCP, IATA | 512-506-8287 | Coordinator | 1900 Cypress Creek, Suite 200 | Cedar Park | Texas | 78613 |
| 301 | Velocity Clinical Research | Gregg Lucksinger | Valencia Smith | MA, GCP, IATA | 512-506-8287 | Coordinator | 1900 Cypress Creek, Suite 200 | Cedar Park | Texas | 78613 |
| 301 | Velocity Clinical Research | Gregg Lucksinger | Amy Vester | BS, GCP, IATA, BLS | 512-506-8287 | Coordinator | 1900 Cypress Creek, Suite 200 | Cedar Park | Texas | 78613 |
| 301 | Velocity Clinical Research | Gregg Lucksinger | Angel Cervantes | GCP, IATA | 512-506-8287 | Coordinator | 1900 Cypress Creek, Suite 200 | Cedar Park | Texas | 78613 |
| 301 | Velocity Clinical Research | Gregg Lucksinger | Tambra Dora | Certified Medical Assistant, Phlebotomy, CPR, GCP, | 512-506-8287 | Coordinator | 1900 Cypress Creek, Suite 200 | Cedar Park | Texas | 78613 |
| 301 | Velocity Clinical Research | Gregg Lucksinger | Therese Spalding | RN, IATA, BLS, GCP, CPR | 512-506-8287 | Coordinator | 1900 Cypress Creek, Suite 200 | Cedar Park | Texas | 78613 |
| 301 | Velocity Clinical Research | Gregg Lucksinger | Yasmin Mota | NRCMA, CPR, BCLS, IATA, GCP | 512-506-8287 | Coordinator | 1900 Cypress Creek, Suite 200 | Cedar Park | Texas | 78613 |
| 302 | Velocity Clinical Research | Marian Shaw | Kate Lyon | CPR, GCP | 208-377-8653 | Coordinator | 2950 E. Magic View Dr., Suite 182 | Meridian | Idaho | 83642 |
| 302 | Velocity Clinical Research | Marian Shaw | Paula Dockstader | CPhT, CPR, GCP | 208-377-8653 | Coordinator | 2950 E. Magic View Dr., Suite 182 | Meridian | Idaho | 83642 |
| 302 | Velocity Clinical Research | Marian Shaw | Audra Weslowski | GCP, IATA | 208-377-8653 | Coordinator | 2950 E. Magic View Dr., Suite 182 | Meridian | Idaho | 83642 |
| 302 | Velocity Clinical Research | Marian Shaw | Erika Calhoun | AS, GCP | 208-377-8653 | Coordinator | 2950 E. Magic View Dr., Suite 182 | Meridian | Idaho | 83642 |
| 302 | Velocity Clinical Research | Marian Shaw | Westin Payne | BA, GCP | 208-377-8653 | Coordinator | 2950 E. Magic View Dr., Suite 182 | Meridian | Idaho | 83642 |
| 302 | Velocity Clinical Research | Marian Shaw | Cecelia Pena | BS, IATA, GCP | 208-377-8653 | Coordinator | 2950 E. Magic View Dr., Suite 182 | Meridian | Idaho | 83642 |
| 302 | Velocity Clinical Research | Marian Shaw | Ronnie Moore | AS, GCP | 208-377-8653 | Research Assistant | 2950 E. Magic View Dr., Suite 182 | Meridian | Idaho | 83642 |
| 302 | Velocity Clinical Research | Marian Shaw | Tyler Scoggins | BA, GCP | 208-377-8653 | Research Assistant | 2950 E. Magic View Dr., Suite 182 | Meridian | Idaho | 83642 |
| 304 | Velocity Clinical Research | Margaret Rhee | Alanna Billups | BA, CITI Protection of Human Services, CITI GCP for | 216-682-0320 | Coordinator | 3619 Park East Dr., Suite 300 | Cleveland | Ohio | 44122 |
| 304 | Velocity Clinical Research | Margaret Rhee | Maggie Jedlinsky | MSW, BSW (Bach. of Social Work), ACRP GCP cert. | 216-682-0320 | Coordinator | 3619 Park East Dr., Suite 300 | Cleveland | Ohio | 44122 |
| 304 | Velocity Clinical Research | Margaret Rhee | Cameron Robinson | BS, ACRP GCP | 216-682-0320 | Coordinator | 3619 Park East Dr., Suite 300 | Cleveland | Ohio | 44122 |
| 304 | Velocity Clinical Research | Margaret Rhee | Casssie Uminski | Community College, Health Carreers Program | 216-682-0320 | Data Entry Coordinator | 3619 Park East Dr., Suite 300 | Cleveland | Ohio | 44122 |
| 304 | Velocity Clinical Research | Margaret Rhee | Jane Boggan | CITI GCP (health info privacy/security for clinical), | 216-682-0320 | Data Entry Coordinator | 3619 Park East Dr., Suite 300 | Cleveland | Ohio | 44122 |
| 304 | Velocity Clinical Research | Margaret Rhee | Lisle Merriman | BA, CITI human subjects research GCP & HIPS, GCP for | 216-682-0320 | Data Entry Coordinator | 3619 Park East Dr., Suite 300 | Cleveland | Ohio | 44122 |
| 305 | Velocity Clinical Research | Greg Feldman, MD, CPI | Keith Cullum | Associate degree (x2), BLS, IATA, ACRP intro to GCP | 803-766-2680 | Site Operations Manager | 1655 Bernardin Ave. Suite 300 | Columbia | South Carolina | 29204 |
| 305 | Velocity Clinical Research | Greg Feldman, MD, CPI | Laura Weier | BS | 803-766-2680 | Coordinator | 1655 Bernardin Ave. Suite 300 | Columbia | South Carolina | 29204 |
| 305 | Velocity Clinical Research | Greg Feldman, MD, CPI | Brandon Harp | MHA, BS (x2) | 803-766-2680 | Coordinator | 1655 Bernardin Ave. Suite 300 | Columbia | South Carolina | 29204 |
| 305 | Velocity Clinical Research | Greg Feldman, MD, CPI | Sharon Williams | Phlebotomy certification | 803-766-2680 | Research Assistant | 1655 Bernardin Ave. Suite 300 | Columbia | South Carolina | 29204 |
| 305 | Velocity Clinical Research | Greg Feldman, MD, CPI | Catherine Mann | Technical college (3 areas), CPR, ACRP GCP Simulation, | 803-766-2680 | Research Assistant | 1655 Bernardin Ave. Suite 300 | Columbia | South Carolina | 29204 |
| 305 | Velocity Clinical Research | Greg Feldman, MD, CPI | DeAnn Tucker | BBA, Associate of Arts, foster care courses | 803-766-2680 | Regualtory Coordinator | 1655 Bernardin Ave. Suite 300 | Columbia | South Carolina | 29204 |
| 306 | Velocity Clinical Research | Lawrence J. Sindel, MD | Jessica Miller, RN | RN | 251-263-5669 | Coordinator | 3715 Dauphin St, Bldg 2, Ste 503B | Mobile | Alabama | 36608 |
| 306 | Velocity Clinical Research | Lawrence J. Sindel, MD | Myia McMillian, B.S., Assistant CRC | BS, Assistant CRC, | 251-263-5669 | Coordinator | 3715 Dauphin St, Bldg 2, Ste 503B | Mobile | Alabama | 36608 |
| 306 | Velocity Clinical Research | Lawrence J. Sindel, MD | Laura Hill | BS, CCRC | 251-263-5669 | Coordinator | 3715 Dauphin St, Bldg 2, Ste 503B | Mobile | Alabama | 36608 |
| 306 | Velocity Clinical Research | Lawrence J. Sindel, MD | Mike Weichman | N/A | 251-263-5669 | Research Assistant | 3715 Dauphin St, Bldg 2, Ste 503B | Mobile | Alabama | 36608 |
| 306 | Velocity Clinical Research | Lawrence J. Sindel, MD | Robyn Robertson | Administrative Clinical Assistant, CITI GCP, IATA, OSHA | 251-263-5669 | Regulatory Coordinator | 3715 Dauphin St, Bldg 2, Ste 503B | Mobile | Alabama | 36608 |
| 306 | Velocity Clinical Research | Lawrence J. Sindel, MD | Danny Kakish | GCP | 251-263-5669 | Coordinator | 3715 Dauphin St, Bldg 2, Ste 503B | Mobile | Alabama | 36608 |
| 307 | Velocity Clinical Research | J. Scott Overcash, MD | Lakeyla Bates | BA, AA, ACPR Intro to GCP, CITI IRB Chair, ACRP | 619-567-1550 | Senior Regulatory Specialist | 5565 Grossmont Center Dr, Bldg 2, Suite 1 | La Mesa | California | 91942 |
| 307 | Velocity Clinical Research | J. Scott Overcash, MD | Angela Anorve | BS, ACRP GCP, OSHA Bloodborne Pathogen | (619) 567-1550 | Coordinator | 5565 Grossmont Center Dr, Bldg 2, Suite 1 | La Mesa | California | 91942 |
| 307 | Velocity Clinical Research | J. Scott Overcash, MD | Ashliegh Lindsay | CPT I, Phlebotomy program, college (current), CA | (619) 567-1550 | Coordinator | 5565 Grossmont Center Dr, Bldg 2, Suite 1 | La Mesa | California | 91942 |
| 307 | Velocity Clinical Research | J. Scott Overcash, MD | Audrey Sanchez | Clinical Research Coordinator, BA, | (619) 567-1550 | Coordinator | 5565 Grossmont Center Dr, Bldg 2, Suite 1 | La Mesa | California | 91942 |
| 307 | Velocity Clinical Research | J. Scott Overcash, MD | Hunter Asmann | BBA (bachelor's of business administration), GCP for | (619) 567-1550 | Coordinator | 5565 Grossmont Center Dr, Bldg 2, Suite 1 | La Mesa | California | 91942 |
| 307 | Velocity Clinical Research | J. Scott Overcash, MD | Keji Kubari | BS | (619) 567-1550 | Coordinator | 5565 Grossmont Center Dr, Bldg 2, Suite 1 | La Mesa | California | 91942 |
| 307 | Velocity Clinical Research | J. Scott Overcash, MD | Kevin Fong | BA, Teaching english as a foregin language, GCP (intro | (619) 567-1550 | Data Entry Coordinator | 5565 Grossmont Center Dr, Bldg 2, Suite 1 | La Mesa | California | 91942 |
| 307 | Velocity Clinical Research | J. Scott Overcash, MD | Stephanie Esquer-Soto | Phlebotomy, Certified Phlebotomy Tech | (619) 567-1550 | Data Entry Coordinator | 5565 Grossmont Center Dr, Bldg 2, Suite 1 | La Mesa | California | 91942 |
| 307 | Velocity Clinical Research | J. Scott Overcash, MD | Sylvia Lindholm | CPR, CITI HIPS, NIH Protecting Human Research Particip | (619) 567-1550 | Coordinator | 5565 Grossmont Center Dr, Bldg 2, Suite 1 | La Mesa | California | 91942 |
| 307 | Velocity Clinical Research | J. Scott Overcash, MD | Pat Kappen, CCRP | CCRP, Edu. in Clinical Trials Design/Management, Certif | (619) 567-1550 | Regulatory Coordinator | 5565 Grossmont Center Dr, Bldg 2, Suite 1 | La Mesa | California | 91942 |

Listing 16.2.1.1 Subject Disposition All-Enrolled Population

| | D 1 6 | | | | | | Reason ITC<br>subject is |
|---|---|---|---|---|---|---|---|
| Subject | Date of<br>Informed | Completion or Discontinuation | | Reason for | ITC | PP | excluded from PP |
| ID | Consent | Date | Status | Discontinuation | | Population | population |
| 301-001 | 02JUN2023 | 02JUN2023 | COMPLETED | | Yes | No | Rhythm strip not uploaded |
| 301-002 | 02JUN2023 | 02JUN2023 | COMPLETED | | Yes | Yes | |
| 301-003 | 09JUN2023 | 09JUN2023 | COMPLETED | | Yes | No | Rhythm strip not uploaded |
| 301-004 | 12JUN2023 | 12JUN2023 | COMPLETED | | Yes | Yes | |
| 301-005 | 13JUN2023 | 13JUN2023 | COMPLETED | | Yes | Yes | |
| 301-006 | 13JUN2023 | 13JUN2023 | COMPLETED | | Yes | Yes | |
| 301-007 | 14JUN2023 | 14JUN2023 | DISCONTINUED | SCREEN FAILURE | No | No | |
| 301-008 | 14JUN2023 | 14JUN2023 | COMPLETED | | Yes | Yes | |
| 301-009 | 15JUN2023 | 15JUN2023 | COMPLETED | | Yes | Yes | |
| 301-010 | 16JUN2023 | 16JUN2023 | COMPLETED | | Yes | Yes | |
| 301-011 | 16JUN2023 | 16JUN2023 | COMPLETED | | Yes | Yes | |
| 301-012 | 16JUN2023 | 16JUN2023 | COMPLETED | | Yes | Yes | |
| 301-013 | 20JUN2023 | 20JUN2023 | COMPLETED | | Yes | Yes | |
| 301-014 | 20JUN2023 | 20JUN2023 | COMPLETED | | Yes | Yes | |
| 301-015 | 21JUN2023 | 21JUN2023 | COMPLETED | | Yes | Yes | |
| 301-016 | 21JUN2023 | 21JUN2023 | COMPLETED | | Yes | Yes | |
| 301-017 | 22JUN2023 | 22JUN2023 | COMPLETED | | Yes | Yes | |
| 301-018 | 22JUN2023 | 22JUN2023 | COMPLETED | | Yes | Yes | |
| 301-019 | 22JUN2023 | 22JUN2023 | COMPLETED | | Yes | Yes | |

Listing 16.2.1.1 Subject Disposition All-Enrolled Population

| Subject<br>ID | Date of<br>Informed<br>Consent | Completion or<br>Discontinuation<br>Date | Status | Reason for<br>Discontinuation | ITC<br>Population | PP<br>Population | Reason ITC subject is excluded from PP population |
|---|---|---|---|---|---|---|---|
| 301-020 | 23JUN2023 | 23JUN2023 | COMPLETED | | Yes | No | Rhythm strip not uploaded |
| 301-021 | 26JUN2023 | 26JUN2023 | COMPLETED | | Yes | Yes | |
| 301-022 | 27JUN2023 | 27JUN2023 | COMPLETED | | Yes | Yes | |
| 302-001 | 02JUN2023 | 02JUN2023 | COMPLETED | | Yes | Yes | |
| 302-002 | 05JUN2023 | 05JUN2023 | COMPLETED | | Yes | Yes | |
| 302-003 | 06JUN2023 | 06JUN2023 | COMPLETED | | Yes | Yes | |
| 302-004 | 07JUN2023 | 07JUN2023 | COMPLETED | | Yes | Yes | |
| 302-005 | 07JUN2023 | 07JUN2023 | COMPLETED | | Yes | Yes | |
| 302-006 | 13JUN2023 | 13JUN2023 | COMPLETED | | Yes | Yes | |
| 302-007 | 14JUN2023 | 14JUN2023 | COMPLETED | | Yes | Yes | |
| 302-008 | 14JUN2023 | 14JUN2023 | COMPLETED | | Yes | Yes | |
| 302-009 | 15JUN2023 | 15JUN2023 | COMPLETED | | Yes | Yes | |
| 302-010 | 15JUN2023 | 15JUN2023 | COMPLETED | | Yes | Yes | |
| 302-011 | 16JUN2023 | 16JUN2023 | COMPLETED | | Yes | Yes | |
| 302-012 | 16JUN2023 | 16JUN2023 | COMPLETED | | Yes | Yes | |
| 302-013 | 20JUN2023 | 20JUN2023 | COMPLETED | | Yes | Yes | |
| 302-014 | 21JUN2023 | 21JUN2023 | COMPLETED | | Yes | Yes | |
| 302-015 | 21JUN2023 | 21JUN2023 | COMPLETED | | Yes | No | Rhythm strip not uploaded |
| 302-016 | 22JUN2023 | 22JUN2023 | COMPLETED | | Yes | Yes | |
| 302-017 | 22JUN2023 | 22JUN2023 | COMPLETED | | Yes | Yes | |

Listing 16.2.1.1 Subject Disposition All-Enrolled Population

| Subject<br>ID | Date of<br>Informed<br>Consent | Completion or<br>Discontinuation<br>Date | Status | Reason for Discontinuation | ITC<br>Population | PP<br>Population | Reason ITC subject is excluded from PP population |
|---|---|---|---|---|---|---|---|
| 302-018 | 22JUN2023 | 22JUN2023 | COMPLETED | | Yes | Yes | |
| 302-019 | 23JUN2023 | 23JUN2023 | COMPLETED | | Yes | Yes | |
| 302-020 | 27JUN2023 | 27JUN2023 | COMPLETED | | Yes | Yes | |
| 302-021 | 28JUN2023 | 28JUN2023 | COMPLETED | | Yes | Yes | |
| 304-001 | 20JUN2023 | 20JUN2023 | COMPLETED | | Yes | Yes | |
| 304-002 | 20JUN2023 | 20JUN2023 | DISCONTINUED | PROTOCOL<br>DEVIATION | No | No | Rhythm strip not uploaded |
| 304-003 | 21JUN2023 | 21JUN2023 | COMPLETED | | Yes | Yes | |
| 304-004 | 21JUN2023 | 21JUN2023 | COMPLETED | | Yes | Yes | |
| 304-005 | 22JUN2023 | 22JUN2023 | COMPLETED | | Yes | Yes | |
| 304-006 | 22JUN2023 | 22JUN2023 | COMPLETED | | Yes | Yes | |
| 304-007 | 27JUN2023 | 27JUN2023 | COMPLETED | | Yes | Yes | |
| 304-008 | 27JUN2023 | 27JUN2023 | COMPLETED | | Yes | Yes | |
| 304-009 | 27JUN2023 | 27JUN2023 | COMPLETED | | Yes | Yes | |
| 304-010 | 28JUN2023 | 28JUN2023 | COMPLETED | | Yes | Yes | |
| 304-011 | 28JUN2023 | 28JUN2023 | COMPLETED | | Yes | Yes | |
| 304-012 | 28JUN2023 | 28JUN2023 | COMPLETED | | Yes | Yes | |
| 304-013 | 29JUN2023 | 29JUN2023 | COMPLETED | | Yes | Yes | |
| 305-001 | 06JUN2023 | 06JUN2023 | COMPLETED | | Yes | No | Rhythm strip not uploaded |
| 305-002 | 06JUN2023 | 06JUN2023 | COMPLETED | | Yes | No | Rhythm strip not uploaded |
| 305-003 | 08JUN2023 | 08JUN2023 | COMPLETED | | Yes | No | Rhythm strip not uploaded |

Listing 16.2.1.1 Subject Disposition All-Enrolled Population

| Subject<br>ID | Date of<br>Informed<br>Consent | Completion or<br>Discontinuation<br>Date | Status | Reason for Discontinuation | ITC<br>Population | PP<br>Population | Reason ITC subject is excluded from PP population |
|---|---|---|---|---|---|---|---|
| 305-004 | 09JUN2023 | 09JUN2023 | COMPLETED | | Yes | Yes | |
| 305-005 | 23JUN2023 | 23JUN2023 | COMPLETED | | Yes | Yes | |
| 305-006 | 23JUN2023 | 23JUN2023 | COMPLETED | | Yes | No | Rhythm strip not uploaded |
| 305-007 | 26JUN2023 | 26JUN2023 | COMPLETED | | Yes | No | Rhythm strip not uploaded |
| 305-008 | 26JUN2023 | 26JUN2023 | COMPLETED | | Yes | No | Rhythm strip not uploaded |
| 305-009 | 28JUN2023 | 28JUN2023 | COMPLETED | | Yes | Yes | |
| 305-010 | 29JUN2023 | 29JUN2023 | COMPLETED | | Yes | Yes | |
| 305-011 | 29JUN2023 | 29JUN2023 | DISCONTINUED | OTHER | No | No | Study closed prior to assessment. |
| 305-012 | 29JUN2023 | 29JUN2023 | COMPLETED | | Yes | Yes | |
| 306-001 | 22JUN2023 | 22JUN2023 | COMPLETED | | Yes | No | Rhythm strip not uploaded |
| 306-002 | 22JUN2023 | 22JUN2023 | COMPLETED | | Yes | No | Rhythm strip not uploaded |
| 306-003 | 26JUN2023 | 26JUN2023 | COMPLETED | | Yes | Yes | |
| 306-004 | 26JUN2023 | 26JUN2023 | COMPLETED | | Yes | No | The reference device does not collect data |
| 306-005 | 28JUN2023 | 28JUN2023 | COMPLETED | | Yes | Yes | |
| 306-006 | 28JUN2023 | 28JUN2023 | COMPLETED | | Yes | Yes | |
| 306-007 | 29JUN2023 | 29JUN2023 | COMPLETED | | Yes | Yes | |
| 307-001 | 14JUN2023 | 14JUN2023 | COMPLETED | | Yes | Yes | |
| 307-002 | 14JUN2023 | 14JUN2023 | COMPLETED | | Yes | Yes | |
| 307-003 | 22JUN2023 | 22JUN2023 | COMPLETED | | Yes | Yes | |
| 307-004 | 22JUN2023 | 22JUN2023 | COMPLETED | | Yes | Yes | |

Mindset Medical, LLC IVC-400-006


Listing 16.2.1.1 Subject Disposition All-Enrolled Population

| Subject<br>ID | Date of<br>Informed<br>Consent | Completion or<br>Discontinuation<br>Date | Status | Reason for Discontinuation | ITC<br>Population | PP<br>Population | Reason ITC subject is excluded from PP population |
|---|---|---|---|---|---|---|---|
| 307-005 | 22JUN2023 | 22JUN2023 | COMPLETED | | Yes | No | The reference device does not collect data |
| 307-006 | 23JUN2023 | 23JUN2023 | COMPLETED | | Yes | Yes | |
| 307-007 | 23JUN2023 | 23JUN2023 | DISCONTINUED | SCREEN FAILURE | No | No | |
| 307-008 | 23JUN2023 | 23JUN2023 | COMPLETED | | Yes | Yes | |
| 307-009 | 26JUN2023 | 26JUN2023 | COMPLETED | | Yes | Yes | |
| 307-010 | 26JUN2023 | 26JUN2023 | COMPLETED | | Yes | No | Thumb drive not recognized by pixel phone. USB was sent back to sponsor for review on 7/20/23 |
| 307-011 | 28JUN2023 | 28JUN2023 | COMPLETED | | Yes | Yes | |

Program name: 1\_16\_2\_1\_1.sas Run Date: 21NOV2023

| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 3 | THIS DOCUMENT SUPERSEDES VERSION: 2 | <b>PAGE:</b><br>1 OF 15 |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 1 0 1 2 5 |
| Active | Informed Vital Core - Statistical Analysis Plan | IVC-400-006d | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| June 22, 2023 | Chris Joslin | Mark Whitehouse | |

Protocol Number: IVC-400-006
Informed Vital Core Application (IVC App)
Statistical Analysis Plan

# A Multi-Center Prospective Open Label Study of a Web-based Application for Pulse Rate in Adult Patients

Mindset Medical, LLC Version 3 Date: June 22, 2023

| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 3 | THIS DOCUMENT SUPERSEDES VERSION: 2 | PAGE:<br>2 OF 15 |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | |
| Active | Informed Vital Core - Statistical Analysis Plan | IVC-400-006d | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| June 22, 2023 | Chris Joslin | Mark Whitehouse | |

Signature Table

| Name | Signature | Date |
|------------------------|-----------|------|
| Elaine Thompson | | |
| Study Biostatistician/ | | |
| Biostatistician Review | | |
| Dan Lubelski, M.D. | | |
| Medical Reviewer | | |
| Kereshmeh Shahriari | | |
| Regulatory Reviewer | | |

| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 3 | THIS DOCUMENT SUPERSEDES VERSION: 2 | PAGE:<br>3 OF 15 |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | |
| Active | Informed Vital Core - Statistical Analysis Plan | IVC-400-006d | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| June 22, 2023 | Chris Joslin | Mark Whitehouse | |

# **Summary of Changes**

| Original | Amendment Change | Reason for Change |
|---|---|---|
| Original release | N/A | |
| Version 2 | Throughout – updated protocol version and date, updated study design, Fitzpatrick numbers, UADE language, and total sessions collected to two. | Update to Clinical Protocol. |
| | Throughout - updated reference device from Kardia to Edan. Updated language from PR to HR throughout the document in sections that reference the Edan ECG. Removed reference to Bluetooth. | Change in reference device. |
| | Product description updated to current language. | Specified language |
| | Throughout – confidentiality notice added to footer, added summary of changes table, minor edits to improve clarify and consistency. | Document Versioning |
| | Removed duplicative information that is in the Clinical Protocol. | Organization |
| | Updated ITC group description for<br>new 12 RR-interval analysis and to<br>add clarification of the disposition of<br>subjects who withdraw during<br>collection. | Clarity |
| | Removed all non-applicable sections. | |
| | Clarified descriptive statistics. | |
| | Moved power analysis to the end, added reference. | |
| | Added health condition and conmeds coding. | |

| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 3 | THIS DOCUMENT SUPERSEDES VERSION: 2 | PAGE:<br>4 OF 15 |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | |
| Active | Informed Vital Core - Statistical Analysis Plan | IVC-400-006d | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| June 22, 2023 | Chris Joslin | Mark Whitehouse | |

| Original | Amendment Change | Reason for Change |
|---|---|---|
| Version 3 | Section 6.2 updated the Fitzpatrick 5 or 6 group to 15% of the Per Protocol group and included language for targeted enrollment if needed. | Specified language |

| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 3 | THIS DOCUMENT SUPERSEDES VERSION: 2 | <b>PAGE</b> : 5 OF 15 |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | |
| Active | Informed Vital Core - Statistical Analysis Plan | IVC-400-006d | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| June 22, 2023 | Chris Joslin | Mark Whitehouse | |

# Contents

| LIST OF A | BBREVIATIONS | 6 |
|---|---|---|
| 1.0 IN | NTRODUCTION | 7 |
| 2.0 S | TUDY OBJECTIVES AND ENDPOINTS | 7 |
| <u>2.1</u> | STUDY OBJECTIVE | |
| <u>2.1.2</u> | | |
| 3.0 S | TUDY HYPOTHESIS | 7 |
| 4.0 S | TATISTICAL AND ANALYTICAL PROCEDURES | 7 |
| <u>4.1</u> | ANALYSIS POPULATIONS AND COLLECTION GROUPS | |
| 4.1.2 | | |
| 4.1.2 | | |
| 4.1.3 | <u> </u> | |
| 4.1.4 | <del>-</del> | |
| 4.1.5 | | |
| <u>4.2</u> | ANALYSIS VARIABLES | |
| 4.2.2 | | |
| 4.2.2 | | |
| 4.2.3 | <u> </u> | |
| 4.2.4 | <del>-</del> | |
| 4.2.5 | <del>-</del> | |
| <u>4.2.6</u> | 6 Adverse Events (AE) | 10 |
| <u>5.0</u> <u>S</u> | TATISTICAL METHODS | 11 |
| 5.1 | SOFTWARE | 11 |
| 5.2 | GENERAL CONSIDERATIONS | 11 |
| 5.2.2 | | 11 |
| 5.2.2 | 2 <u>Descriptive Statistics and Summary Tables</u> | 11 |
| 5.3 | ENDPOINT DATA ANALYSIS METHODS | |
| 5.3.2 | | 11 |
| 5.3.2 | 2 <u>IVC App PR Reporting Rate</u> | |
| 6.0 B | ACKGROUND, SAMPLE SIZE | 12 |
| <u>6.1</u> | Power Analysis Methodology | |
| <u>6.2</u> | POWER ANALYSIS FOR SAMPLE SIZE | |
| <u>6.3</u> | SAFETY ANALYSIS | |
| <u>6.4</u> | EXPLORATORY ANALYSES | 15 |
| 7.0 R | EFERENCES | 15 |

| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 3 | THIS DOCUMENT SUPERSEDES VERSION: 2 | PAGE:<br>6 OF 15 |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | |
| Active | Informed Vital Core - Statistical Analysis Plan | IVC-400-006d | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| June 22, 2023 | Chris Joslin | Mark Whitehouse | |

# List Of Abbreviations

The following abbreviations and special terms are used in this Statistical Analysis Plan.

| Explanation |
|--------------------------------------------------------------------------|
| Adverse Event |
| Average Root Mean Square |
| Body Mass Index |
| Blood Pressure |
| Beats per Minute |
| Confidence Interval |
| Clinical Study Report |
| Electrocardiogram |
| electronic Case Report Form |
| Electronic Data Capture |
| Food and Drug Administration |
| Heart Rate |
| Informed Consent Form |
| International Conference on Harmonization |
| Institutional Review Board |
| Intent-to-Capture |
| Informed Vital Core Application |
| Medical Dictionary for Regulatory Activities |
| Per Protocol |
| Pulse Rate |
| Preferred Term |
| Photoplethysmography |
| Red, Green, and Blue |
| Root Mean Square |
| Remote Photoplethysmography |
| The time elapsed between two successive R waves of the QRS signal on the |
| electrocardiogram (and its reciprocal, the HR). |
| Serious Adverse Event |
| Statistical Analysis Plan |
| System Organ Class |
| Treatment Emergent Adverse Event |
| Unanticipated Adverse Device Effect |

| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 3 | THIS DOCUMENT SUPERSEDES VERSION: 2 | <b>PAGE</b> : 7 OF 15 |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | |
| Active | Informed Vital Core - Statistical Analysis Plan | IVC-400-006d | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| June 22, 2023 | Chris Joslin | Mark Whitehouse | |

#### 1.0 Introduction

This documentation describes the planned data analyses for clinical study IVC-400-006 sponsored by Mindset Medical, LLC.

This SAP supersedes the statistical considerations identified in the protocol; where considerations are substantially different, and these differences will be identified. If additional analyses are required to supplement objectives described in the SAP, they may be performed and will be identified in the Clinical Study Report (CSR) or through an SAP addendum (as warranted).

Analyses described in the current SAP version is based on the protocol version 1 IVC-400-006 dated March 31, 2023.

# 2.0 Study Objectives and Endpoints

## 2.1 Study Objective

The primary objective of the study is to establish that pulse rate (PR) measured with the IVC App are accurate to within +/- 3 BPM ARMS (average root mean square) of Heart Rate (HR) measured with the reference ECG device.

## 2.1.1 Primary Endpoint

The primary endpoint is a non-inferiority comparison to an FDA approved reference device to establish that PR measured with the IVC App are accurate to an ARMS of +/- 3 BPM. In accordance with ISO 80601-2-61:2017(E) accuracy will be calculated as the RMS difference between the IVC App and the heart rate measured by the ECG reference device.

# 3.0 Study Hypothesis

The IVC App can measure pulse rate between 50 and 130 BPM to an accuracy of  $\pm$ 0 BPM average RMS. The hypothesis will be tested in a non-inferiority design. PR will be collected simultaneously with the IVC App and HR with an ECG reference device, and the ARMS and its 95% confidence interval calculated. If the upper limit of the 95% confidence interval of the ARMS is < 3.0, the IVC App will be determined to be non-inferior and the hypothesis that it is accurate to an ARMS of  $\pm$ 0.0 accepted.

# 4.0 Statistical and Analytical Procedures

## 4.1 Analysis Populations and Collection Groups

The following populations will be considered for the study:

#### 4.1.1 All-Enrolled Population

The All-Enrolled population will be defined as all subjects who signed the ICF. The number of screen failures and the reasons for failure will be tabulated and reported. Subjects who consent but withdraw before data collection will be tabulated and reported.

| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 3 | THIS DOCUMENT SUPERSEDES VERSION: 2 | <b>PAGE:</b> 8 OF 15 |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | |
| Active | Informed Vital Core - Statistical Analysis Plan | IVC-400-006d | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| June 22, 2023 | Chris Joslin | Mark Whitehouse | |

## 4.1.2 Intent-to-Capture Population (ITC)

The Intent-to-Capture (ITC) population will be defined as all consented subjects who passed screening and completed at least one data collection session without withdrawing.

#### 4.1.3 Per-Protocol Population (PP)

In order to compare devices, subjects must have a simultaneous PR measurement from the IVC App and an HR measurement from the reference ECG device. Therefore, the Per Protocol analysis group for the primary endpoint will consist of subjects from whom PR measurement from the IVC App and a successful HR data collection from the ECG reference device were collected during the same window.

In preliminary testing of the ECG reference device, not all collections produced a rhythm strip suitable for analysis. The ECG data are processed after the subject's participation in the study ends, so there is no way to detect an unusable ECG collection during the study. In order to increase the likelihood of collecting usable ECG data, two sessions will be collected from each subject.

Subjects will be asked to collect up to 3 additional sessions as technical fallbacks if a collection failure occurs from the reference device or if conditions at the study site interfere with the functionality of the IVC App. Examples of technical difficulties include, but are not limited to, frozen or stuttering video during data capture, failure of the reference device to produce a rhythm strip, connection issues with the reference device, interruptions during data collection that require the subject to leave the camera frame, or upload failures.

### 4.1.4 Successful Data Collection

ECG rhythm analysis will be performed and calculated using a synchronized moving average across 12-RR intervals as described in IVC-400-006i — Informed Vital Core Heart Rate Rhythm Analysis Procedure. A successful data collection is defined as a session that produces a measurement from the IVC App and the ECG reference device where the moving average of the HR measurement from the reference device does not vary by more than 15 BPM during the 1 minute of measurement. A 15 BPM threshold is applied to the ECG data because variability in contact with the electrodes, subject movement, or atypical ECG waveforms can result in processing artifacts that appear as unrealistically large jumps or fluctuations in HR during the session. In instances where the reference HR is found to vary by more than 15 BPM, the second data collection session will be used for analysis.

The second session will not be treated as a fallback for the IVC App. The study is designed to represent a patient encounter with the IVC App. Under the intended use, if the IVC App cannot collect video from which a PR can be determined after prompts to stop moving or improve lighting, patients are instructed to retry up to twice. If the HR collection with the ECG reference device is successful but the IVC App does not produce a PR, the subject will be excluded from the PP analysis group and considered to be an IVC App collection failure.

All subjects in the ITC group who were not included in the PP group will be listed with the reason they were excluded from the analysis. Subjects will be excluded if the reference device does not collect data, the ECG

| INFORMED | DOCUMENT VERSION: 3 | THIS DOCUMENT SUPERSEDES VERSION: 2 | PAGE: |
|---|---|---|---|
| MINDSET MEDICAL | | | 9 OF 15 |
| STATUS: | TITLE: | IDENTIFICATION: | |
| Active | Informed Vital Core - Statistical Analysis Plan | IVC-400-006d | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| June 22, 2023 | Chris Joslin | Mark Whitehouse | |

from both reference device collections is not suitable for rhythm analysis as defined above, or the IVC App does not report a PR during the first session where the ECG collection is successful.

A subject could withdraw before all data collection attempts and technical fallbacks are completed. If the subject has a successful collection, they will still be included in the PP group. Otherwise, they will be excluded from the PP group. If they completed an IVC App collection without a reference HR, that collection will be included when calculating the IVC App success rate as described in section 5.3.2.

### 4.1.5 Data Collection Groups

Simultaneous data collection from the ECG reference device and IVC App device will be performed on all subjects so there is only one data collection group.

## 4.2 Analysis Variables

### 4.2.1 Subject's Disposition and Analysis Sets

Disposition will be summarized descriptively with counts and percentages using the All-Enrolled population for both devices (IVC App and reference device) data collection and all Intent to Collect and all Per Protocol subjects. The number and percentage of subjects who prematurely discontinued from the study along with reasons for study discontinuation will be summarized as well.

A subject's eligibility with inclusion/exclusion criteria failed/met will be listed, along with the list of protocol deviations.

#### 4.2.2 Demographics and Baseline Characteristics

Demographic data and baseline characteristics will include:

- Sex
- Ethnicity
- Race
- Fitzpatrick scale- Fitzpatrick scale skin tones will be grouped into light (Fitzpatrick 1 and 2), medium (Fitzpatrick 3 and 4) and dark (Fitzpatrick 5 and 6).
- Age (years)
- Height (cm)
- Weight (kg)
- BMI (kg/m²)

Demographics and baseline characteristics will be tabulated and summarized as described in section 5.2.2.

The summary results will be based on the ITC population.

#### 4.2.3 Health Conditions and Concomitant Medications

Self-reported health conditions will be coded using MedDRA, tabulated and reported.

Concomitant medications will be coded with WHODrug, tabulated, and reported.

| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 3 | THIS DOCUMENT SUPERSEDES VERSION: 2 | <b>PAGE</b> : 10 OF 15 |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | |
| Active | Informed Vital Core - Statistical Analysis Plan | IVC-400-006d | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| June 22, 2023 | Chris Joslin | Mark Whitehouse | |

The summary results will be based on the ITC population.

#### 4.2.4 Endpoint Variables

The endpoint variables are the IVC App PR and ECG reference device HR.

Summary statistics of the HR and PR measured for each device within the PP group will be tabulated and reported as described in section 5.2.2.

Subjects in the PP group will be tabulated by IVC App PR in groups of 10 bpm and the number of subjects and percentages in each pulse rate group reported.

### 4.2.5 Subgroup Analysis

No subgroup analyses will be performed, since the study is not powered or sized for subgroup analysis.

## 4.2.6 Adverse Events (AE)

While adverse events are not anticipated in this clinical study, if the reason for removal of a subject from the study is an adverse event, the event will be recorded on the appropriate eCRF(s) and will be reported to Mindset Medical per the AE reporting guidelines (Required Reporting Timelines per Regulatory Guidance). All efforts will be made to follow the subject until the condition resolves, or the Investigator determines that the subject's health has returned to an acceptable state.

All verbatim AE terms will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) of the latest version and summarized by system organ class (SOC) and preferred term (PT).

An Unanticipated Adverse Device Effect (UADE) is "any serious" adverse effect on health or safety or any lifethreatening problem or death caused by, or associated with, a device, if that effect, problem, or death was not previously identified in any nature, severity, or degree of incidence in the investigational plan or any other unanticipated serious problem associated with a device that relates to the rights, safety, and welfare of subjects.

All Life-Threatening AEs will be considered as Severe.

All AEs will be classified in one of two types of relation to device:

- Not Related
- Related (Definitely Related and Possibly Related)

AEs in the ITC population will be tabulated and summarized by type, severity, and MedDRA codes as described in section 5.2.2.

| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 3 | THIS DOCUMENT SUPERSEDES VERSION: 2 | <b>PAGE:</b><br>11 OF 15 |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | |
| Active | Informed Vital Core - Statistical Analysis Plan | IVC-400-006d | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| June 22, 2023 | Chris Joslin | Mark Whitehouse | |

## 5.0 Statistical Methods

#### 5.1 Software

The primary endpoint analyses will be performed using CRAN R Version 4.3.0 or higher using the boot package version 1.3-28.1 or above. Tables and listings will be produced using R and SAS version 9.4 (SAS Institute Inc.)

#### 5.2 General Considerations

## 5.2.1 Listings

All study data will be included in the study data listings. Both the captured data and the MedDRA and WHODrug codes will be provided. Listings will be displayed by subject in chronological order, if not stated otherwise.

Study data will be provided in electronic format, either as SAS XPT V5 files or CSV files.

## 5.2.2 Descriptive Statistics and Summary Tables

The total number of subjects in the study group (N) under the stated population will be displayed in the header of summary tables.

For age, height, weight, and BMI, the mean, standard deviation, minimum and maximum will be presented along with the n size from which the statistics were calculated.

PR and HR data will be presented as median, lower, and upper quartiles, min, max, and n size because they were not normally distributed in product development data (5.1.4).

For categorical variables, count, and percentage of subjects/counts in each device group and/or category will be presented. Percentages will be based on number of subjects with non-missing values, if not specified otherwise.

## 5.3 Endpoint Data Analysis Methods

## 5.3.1 Primary Endpoint

For the primary endpoint analysis, the ARMS will be calculated as the square root of the mean difference between the devices, as described in ISO 80601-2-61:2017(E). All PP subjects will be included in the primary endpoint analysis. The 95% CI for the primary endpoint analysis will be determined by jackknifing 100,000 samples with replacement and calculating a 95% CI from the distribution of ARMS among the jackknifed samples. If the ARMS and its upper 95% confidence interval are below the target of 3.0, the device will be determined to be non-inferior.

| INFORMED | DOCUMENT VERSION: 3 | THIS DOCUMENT SUPERSEDES VERSION: 2 | PAGE: |
|---|---|---|---|
| MINDSET MEDICAL | | | 12 OF 15 |
| STATUS: | TITLE: | IDENTIFICATION: | |
| Active | Informed Vital Core - Statistical Analysis Plan | IVC-400-006d | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| June 22, 2023 | Chris Joslin | Mark Whitehouse | |

A Bland-Altman plot will be constructed from the differences vs. the average measured PRs and HRs for all PP subjects to assist in visualizing the differences between devices and the full range of PR and HR measurements. Since the differences were not normally distributed due to the "white coat" effect on PR in the product development data, upper and lower  $95^{th}$  percentiles will be drawn on the graph to aid in visualization rather than two standard deviations. Visible outliers with greater than +/- 6.0 BPM difference from the reference device will be tabulated. A threshold of +/- 6.0 BPM will be considered outlying because under a labelled ARMS of +/- 3.0, 95% of the differences should fall in the range of +/- 6.0 BPM against the reference.

#### 5.3.2 IVC App PR Reporting Rate

The overall PR reporting rate of the IVC App will be calculated from the ITC population. All subjects with an IVC App PR from the first non-fallback session will be counted as IVC App collections. The total count of subjects with IVC App collections will be divided by the count of subjects in the ITC group to calculate the overall PR reporting rate for the IVC App.

A second rate will be calculated as above, only excluding subjects who had no IVC App sessions collected due to repeated technical failures. The second rate reflects the proportion of subjects who were able to use the IVC App and is more reflective of proportion of sessions where a reliable PR can be determined from the analyzed video frames. The number of subjects excluded due to technical failures will also be reported.

## 6.0 BACKGROUND, SAMPLE SIZE

## 6.1 Power Analysis Methodology

Power analysis and enrollment percentages for the PR measures were based on data collected from 571 consented subjects who attempted one or more simultaneous data collections from a Masimo MightySat fingertip PPG device (reference device) and the IVC App. The data collection rate across the 571 subjects was used to determine how many subjects to enroll in order to meet the target n size for the non-inferiority analysis. Collection success defined as a successful data collection from the IVC App was 80.5% (95% CI of 79% - 82%).

The measured PRs from both the reference device and the IVC App had a high kurtosis, as did the differences between devices. Data were also not Box-Cox normal, so they were treated as nonparametric. Deviation from a normal distribution has previously been observed in measured PR during studies and is attributed to a "white coat" phenomenon, with people who have higher 24-hour resting heart rates showing a more pronounced increase (1).

Under the assumption that the IVC App is non-inferior to the reference device, at 90% power the upper bound of the bootstrapped 95% CI should fall below 3.0, 90% of the time. Subsampling the differences between the devices at systematically varied n sizes and calculating an ARMS and its 95% CI on each subsample gives a distribution of 95% confidence intervals for each n size. The distribution of confidence

| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 3 | THIS DOCUMENT SUPERSEDES VERSION: 2 | PAGE:<br>13 OF 15 |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | |
| Active | Informed Vital Core - Statistical Analysis Plan | IVC-400-006d | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| June 22, 2023 | Chris Joslin | Mark Whitehouse | |

intervals is used to determine power at that n size. Since the distribution of differences was nonparametric, 95% CI distributions were bagged (bootstrap aggregated). The bagging procedure was performed as follows:

- 1. A cohort of 475 or 484 subjects with one paired PR measurement each was established as described later.
- 2. Random subsamples with replacement were selected from the cohort at n sizes from 20 to 100 in intervals of 5. For each n size, 4,000 subsamples were generated.
- 3. The 95% confidence interval on the Arms was bootstrapped on each subsample by jackknifing with replacement 2,000 times.
- 4. The 95% confidence interval upper bounds were aggregated for each n size to produce a distribution of upper 95% confidence intervals.
- 5. 90th and 95th percentiles were calculated to find the power at each n size.

## 6.2 Power Analysis for Sample Size

A total of 85 subjects (n = 85) will be enrolled.



**Figure 1**. Power analysis workflow. The first sessions were selected as representative of the study design for the initial power analysis (left). A second set of sessions with the largest difference from the reference device were used in a conservative scenario (right).

A total of 475 subjects out of the 571 in the product development cohort had data collected the IVC App in from the first PR collection and were included in the initial power analysis. Only the first PR sessions were used in order to accurately model the clinical study design, where subjects will have only one IVC App collection. The overall ARMS was 0.9 BPM. The bagging procedure was performed on n sizes ranging from 20 to 100 subjects (Figure 2). At all n sizes in the analysis, the 95<sup>th</sup> percentile of the confidence intervals was below the target ARMS of 3.0. Thus, n sizes of 20 or greater are powered at 95%.

| INFORMED | DOCUMENT VERSION: 3 | THIS DOCUMENT SUPERSEDES VERSION: 2 | PAGE: |
|---|---|---|---|
| MINDSET MEDICAL | | | 14 OF 15 |
| STATUS: | TITLE: | IDENTIFICATION: | |
| Active | Informed Vital Core - Statistical Analysis Plan | IVC-400-006d | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| June 22, 2023 | Chris Joslin | Mark Whitehouse | |



**Figure 2**. Bagging results for sample sizes ranging from 20 to 100. The filled-in squares show the 95th percentile and the open circles show the 90th percentile of the upper bound of the confidence intervals. The x-axis shows the sample size of the subsamples and the y-axis is the RMS. All 95th percentiles are below the target ARMS of 3.0.

As well as the first IVC App collection attempt used in the power analysis above, some of the subjects provided additional data collection sessions under varied conditions for product development. To perform a more conservative power analysis, the session with the largest absolute difference from the reference device was selected for each subject. The same bagging analysis over 484 "worst case" collections with an ARMS of 1.5 BPM showed 90% power with 40 subjects and 95% power with 45 subjects. The conservative power analysis was used to establish a PP group goal of 55 subjects to ensure that power is at or above 95%. Additionally, a sample size greater than 50 subjects ensures that the sample is likely to be representative of the IVC App performance under the Central Limit Theorem. Since the IVC App is designed to report only reliable results and inform the user that a PR could not be collected otherwise, not all sessions result in a successful PR measurement. As mentioned above, the PR collection rate for the IVC app was 80%, so the study will be overenrolled to reach the target PP group size. A total of 85 subjects will be enrolled, allowing for screening failures, withdrawals, technical failures, and sessions where the IVC App does not report a PR.

In order to ensure a diverse PP group, the enrollment target for the PP group is 15% in the dark (Fitzpatrick 5-6) skin tone group. Initially enrollment will be random, but targeted enrollment may be used to meet skin tone goals if the dark skin tone PP group is projected to fall below the 15% goal.

| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 3 | THIS DOCUMENT SUPERSEDES VERSION: 2 | <b>PAGE</b> : 15 OF 15 |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | |
| Active | Informed Vital Core - Statistical Analysis Plan | IVC-400-006d | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| June 22, 2023 | Chris Joslin | Mark Whitehouse | |

## 6.3 Safety Analysis

No safety analysis is planned. The IVC App is a remote device so no device related AEs are anticipated.

# 6.4 Exploratory Analyses

All exploratory analyses will be based on ITC and PP populations.

## 7.0 References

**1)** Paolo Palatini, Edoardo Casiglia, Paolo Pauletto, Jan Staessen, Niko Kaciroti and Stevo Julius. Relationship of Tachycardia With High Blood Pressure and Metabolic Abnormalities. A Study With Mixture Analysis in Three Populations. Hypertension 30:1267–1273 (1997). https://doi.org/10.1161/01.HYP.30.5.1267

| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE: |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 1 OF 18 |
| | | | ļ |
| Active | Rhythm Strip Analysis Procedure for | IVC-400-006i | |
| | IVC-400-006 | | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| May 30, 2023 | Chris Joslin | Mark Whitehouse | |

# Informed Vital Core Rhythm Strip Analysis Procedure for IVC-400-006

IVC-400-006i Rev. 1

Mindset Medical, LLC

| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | <b>PAGE</b> : 2 OF 18 |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 20110 |
| Active | Rhythm Strip Analysis Procedure for IVC-400-006 | IVC-400-006i | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| May 30, 2023 | Chris Joslin | Mark Whitehouse | |

# **Table of Contents**

# Contents

| 2. SCOPE | 1. | INTRODUCTION | | |
|---|---|---|---|---|
| 3. REFERENCES 4. PROCEDURE 4.1. GENERAL PROCEDURE FOR COLLECTING ECG RHYTHM STRIP XML FILE 4.2. RHYTHM STRIP ANALYSIS OF ELECTROCARDIOGRAM SIGNAL FOR REFERENCE HEART RATE 5. REFERENCES APPENDIX A – README | | | | |
| 4. PROCEDURE | 2. | SCOPE | | |
| 4. PROCEDURE | 3. | REFER | ENCES | 3 |
| 4.1. GENERAL PROCEDURE FOR COLLECTING ECG RHYTHM STRIP XML FILE | | | | |
| 4.2. RHYTHM STRIP ANALYSIS OF ELECTROCARDIOGRAM SIGNAL FOR REFERENCE HEART RATE | | | | |
| 5. REFERENCES | | | | |
| APPENDIX A – README | | 4.2. | RHYTHM STRIP ANALYSIS OF ELECTROCARDIOGRAM SIGNAL FOR REFERENCE HEART RATE | ∠ |
| | 5. | REFER | ENCES | |
| | ADDENDIV A — DE ADME | | | |
| APPENDIX B – RHYTHM STRIP ANALYSIS VALIDATION | AFFENDIA A TRADIVIE | | | |
| | ΑP | PENDIX | B – RHYTHM STRIP ANALYSIS VALIDATION | |

| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE:<br>3 OF 18 |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | |
| Active | Rhythm Strip Analysis Procedure for IVC-400-006 | IVC-400-006i | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| May 30, 2023 | Chris Joslin | Mark Whitehouse | |

## 1. Introduction

Mindset Medical is the developer of the new, prescription use, Informed Vital Core Application (IVC App). The IVC App is intended to measure the vital signs including the pulse rate (PR). The IVC App will be available by prescription use, intended for use in hospitals, clinics, long-term care, and home and is designed to be used as a web-based application.

This procedure uses the rhythm strip from the Edan SE-301 ECG device to determine the heart rate measured by the ECG device during the Informed Vital Core Pulse Rate Clinical Study. The terms heart rate analysis and rhythm strip analysis may be used interchangeably in this document, as they are both defined as the procedure by which the Edan SE-301 ECG-produced rhythm strip is analyzed to determine a heart rate.

## 2. Scope

The scope of this document is limited to determining the heart rate obtained by the Edan SE-301 ECG device used in IVC-400-006 Pulse Rate Clinical Study. This document does not include the procedure for heart rate determination or analysis produced by the IVC App.

## 3. References

| Document Number | Description |
|---|---|
| IVC-400-006 | Informed Vital Core – Clinical Study Protocol |
| IVC-400-006g | Informed Vital Core – Clinical Study Site Instruction Guide: Pulse Rate |

## 4. Procedure

Heart rate (HR) is calculated using lead-I from a 6-lead ECG taken with the Edan SE-301 (ECG). The ECG unit is configured to conduct a 60 second ECG recording conducted simultaneously with an IVC App PR measurement session. The results of the ECG recording are stored in a standardized XML format and are referred to as the ECG XML Rhythm Strip file(s) (or rhythm strip(s)). Simple averaging over the course of the session is not precise due to natural heart rate variability. In order to achieve high enough precision to validate the accuracy of the IVC App, the inter-session heart rate must match the measurement times reported by the ECG device.

A Python script (or script) reads the ECG XML Rhythm Strip files, aligns the data collection windows, and performs the heart rate analysis; calculating a heart rate that is accurately synchronized to the IVC App data collection window. The heart rates produced from the rhythm strip by the Python script will be used as the reference for the primary endpoint analysis.

| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | <b>PAGE:</b> 4 OF 18 |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 7 . 5. 25 |
| Active | Rhythm Strip Analysis Procedure for IVC-400-006 | IVC-400-006i | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| May 30, 2023 | Chris Joslin | Mark Whitehouse | |

The Python script has been validated on stable releases of standard publicly available libraries and runs in a virtual environment configured from a requirements text file that lists the specific packages and versions (Xie, et. al., 2023). Heart rate analysis is performed using the WFDB package described in Waveform Database Software Package (WFDB) for Python (version 4.1.0). The SHA # will be documented on the Rhythm Strip Analysis Report (RSAR). Validation of the procedure in Section 4.1 and 4.2 will be outlined in Appendix B.

## 4.1. General Procedure for Collecting ECG Rhythm Strip XML File

- 1. After the ECG measurement has been collected from the subject per the clinical study protocol, the clinical site staff will upload the ECG Rhythm Strip XML File to a shared drive per the IVC-400-006g Pulse Rate Clinical Study Site Instruction Guide.
- 2. The subject ID will be on the ECG Rhythm Strip XML file and the file will be copied by Mindset Medical staff to a file folder on SharePoint.
- 3. The Rhythm Strip Analysis Report will be stored on SharePoint.
- 4. The ECG Rhythm Strip XML files and Heart Rate Analysis Reports will be stored per 21 CFR 812.140 (b), (d), and (e) when the trial is complete.

## 4.2. Rhythm Strip Analysis of Electrocardiogram Signal for Reference Heart Rate

Steps involved for the Mindset Medical staff in generating the reference heart rate are listed below:

- 1. Access the ECG Rhythm Strip XML file from the SharePoint folder.
- 2. Download the metadata file produced by the IVC App.
- 3. Run the Python Script on the XML file and the IVC App metadata file. The script can be run from the command line in a Python virtual environment that enforces the version control with arguments that point to the ECG XML Rhythm Strip file and the IVC App metadata file. The Python script performs the following steps:
  - a. Read the ECG Rhythms Strip XML file and return the lead-I signal in millivolts at a 1 kHz sample rate.
  - b. Adjust for the 2.3 second buffer delay added by the Edan SE-301 to synchronize timing with the reference device clock.
  - c. Apply the WFDB XQRS peak detection algorithm.
  - d. Plot and save the ECG signal with peak markers for visual validation.
  - e. Compute the moving average heart rate (HR-MA) by using a sliding window of 12 RR-intervals. Boundary values are imputed using expanding windows.
  - f. Sample the HR-MA at the solution times reported by IVC App metadata and average.
| INFORMED | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE: |
|---|---|---|---|
| MINDSET MEDICAL | | | 5 OF 18 |
| STATUS: | TITLE: | IDENTIFICATION: | |
| Active | Rhythm Strip Analysis Procedure for | IVC-400-006i | |
| | IVC-400-006 | | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| May 30, 2023 | Chris Joslin | Mark Whitehouse | |

- 4. Visual validation of the Rhythm Strip Analysis Report is performed by two Mindset Medical reviewers. The first review is the primary reviewer and the second reviewer will perform a quality control review.
  - a. Discrepancies identified will be documented and reviewed by management for inclusion or exclusion in the final analysis.
- 5. The result is a single integer value for reference heart rate that is entered into the study electronic data capture system.

Note: The script will warn if there is a timing discrepancy or if the reference range violates the study protocol which can be included in the notes field.

| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | <b>PAGE</b> :<br>6 OF 18 |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 0 OF 18 |
| Active | Rhythm Strip Analysis Procedure for IVC-400-006 | IVC-400-006i | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| May 30, 2023 | Chris Joslin | Mark Whitehouse | |

## 5. References

Xie, C., McCullum, L., Johnson, A., Pollard, T., Gow, B., & Moody, B. (2023). Waveform Database Software Package (WFDB) for Python (version 4.1.0). *PhysioNet*. <a href="https://doi.org/10.13026/9njx-6322">https://doi.org/10.13026/9njx-6322</a>

| [ INFORMED | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | PAGE: |
|---|---|---|---|
| MINDSET MEDICAL | | | 7 OF 18 |
| STATUS: | TITLE: | IDENTIFICATION: | |
| Active | Rhythm Strip Analysis Procedure for | IVC-400-006i | |
| 1.00.70 | IVC-400-006 | | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| May 30, 2023 | Chris Joslin | Mark Whitehouse | |

# Appendix A – Readme

- Create venv with Python 3.9.16
- pip install -r requirements.txt
- Run using command below

python edan\_se301\_ra.py file\_name\_ecg file\_name\_ivc timezone\_name

where timezone\_name is US/Pacific or US/Mountain etc. Output prints hr reference value and saves ecg with annotations as pdf

| INFORMED<br>MINDSET MEDICAL | DOCUMENT VERSION: 1 | THIS DOCUMENT SUPERSEDES VERSION: X | <b>PAGE</b> :<br>8 OF 18 |
|---|---|---|---|
| STATUS: | TITLE: | IDENTIFICATION: | 0 01 10 |
| Active | Rhythm Strip Analysis Procedure for IVC-400-006 | IVC-400-006i | |
| EFFECTIVE DATE: | AUTHOR: | APPROVED BY: | |
| May 30, 2023 | Chris Joslin | Mark Whitehouse | |

## Appendix B – Rhythm Strip Analysis Validation

To validate the heart rate Rhythm Analysis Procedure for IVC-400-600 using the ECG XML Rhythm Strip, ten (10) trial sessions simulating the conditions of the clinical protocol were conducted. Validation included following the procedure in Sections 4.1 and 4.2 with 100% accuracy in automated peak detection.

Demonstrated accuracy is evaluated by visual inspection of two reviewers using the annotated report generated by the standard script. Though the official implementation allows for documented human correction, the validation standard is zero false positive or false negative automated classifications.

Each of these criteria has been successfully met as can be verified in the annotated figures included in the appendix. The black signal line reproducing the cardiograph confirms the first requirement. Red crosses indicate automated peak detections. If there are corrected false positives they would be overlaid with large gray x's; false negatives corrected by a reviewer would be indicated with large blue crosses. The absence of such annotations indicates automated accuracy of 100% for this sample. The bottom plot shows the instantaneous heart rate and its 10 second moving average; blue dots on that MA line show the IVC sample timestamps synchronized with ECG demonstrate completion of criteria two.

## 20230418-113534-001.xml



## 20230418-113913-001.xml



#### 20230418-114056-001.xml



## 20230418-114244-001.xml



## 20230418-115738-001.xml



Confidential – Mindset Medical, LLC Do not distribute without permission.

HR [bpm]

## 20230418-115928-001.xml



## 20230418-120134-001.xml



## 20230418-120313-001.xml



## 20230418-120509-001.xml



## 20230419-110011-001.xml



Listing 16.2.1.1 Subject Disposition All-Enrolled Population

| | D 1 6 | | | | | | Reason ITC<br>subject is |
|---|---|---|---|---|---|---|---|
| Subject | Date of<br>Informed | Completion or Discontinuation | | Reason for | ITC | PP | excluded from PP |
| ID | Consent | Date | Status | Discontinuation | | Population | population |
| 301-001 | 02JUN2023 | 02JUN2023 | COMPLETED | | Yes | No | Rhythm strip not uploaded |
| 301-002 | 02JUN2023 | 02JUN2023 | COMPLETED | | Yes | Yes | |
| 301-003 | 09JUN2023 | 09JUN2023 | COMPLETED | | Yes | No | Rhythm strip not uploaded |
| 301-004 | 12JUN2023 | 12JUN2023 | COMPLETED | | Yes | Yes | |
| 301-005 | 13JUN2023 | 13JUN2023 | COMPLETED | | Yes | Yes | |
| 301-006 | 13JUN2023 | 13JUN2023 | COMPLETED | | Yes | Yes | |
| 301-007 | 14JUN2023 | 14JUN2023 | DISCONTINUED | SCREEN FAILURE | No | No | |
| 301-008 | 14JUN2023 | 14JUN2023 | COMPLETED | | Yes | Yes | |
| 301-009 | 15JUN2023 | 15JUN2023 | COMPLETED | | Yes | Yes | |
| 301-010 | 16JUN2023 | 16JUN2023 | COMPLETED | | Yes | Yes | |
| 301-011 | 16JUN2023 | 16JUN2023 | COMPLETED | | Yes | Yes | |
| 301-012 | 16JUN2023 | 16JUN2023 | COMPLETED | | Yes | Yes | |
| 301-013 | 20JUN2023 | 20JUN2023 | COMPLETED | | Yes | Yes | |
| 301-014 | 20JUN2023 | 20JUN2023 | COMPLETED | | Yes | Yes | |
| 301-015 | 21JUN2023 | 21JUN2023 | COMPLETED | | Yes | Yes | |
| 301-016 | 21JUN2023 | 21JUN2023 | COMPLETED | | Yes | Yes | |
| 301-017 | 22JUN2023 | 22JUN2023 | COMPLETED | | Yes | Yes | |
| 301-018 | 22JUN2023 | 22JUN2023 | COMPLETED | | Yes | Yes | |
| 301-019 | 22JUN2023 | 22JUN2023 | COMPLETED | | Yes | Yes | |

Listing 16.2.1.1 Subject Disposition All-Enrolled Population

| Subject<br>ID | Date of<br>Informed<br>Consent | Completion or<br>Discontinuation<br>Date | Status | Reason for<br>Discontinuation | ITC<br>Population | PP<br>Population | Reason ITC subject is excluded from PP population |
|---|---|---|---|---|---|---|---|
| 301-020 | 23JUN2023 | 23JUN2023 | COMPLETED | | Yes | No | Rhythm strip not uploaded |
| 301-021 | 26JUN2023 | 26JUN2023 | COMPLETED | | Yes | Yes | |
| 301-022 | 27JUN2023 | 27JUN2023 | COMPLETED | | Yes | Yes | |
| 302-001 | 02JUN2023 | 02JUN2023 | COMPLETED | | Yes | Yes | |
| 302-002 | 05JUN2023 | 05JUN2023 | COMPLETED | | Yes | Yes | |
| 302-003 | 06JUN2023 | 06JUN2023 | COMPLETED | | Yes | Yes | |
| 302-004 | 07JUN2023 | 07JUN2023 | COMPLETED | | Yes | Yes | |
| 302-005 | 07JUN2023 | 07JUN2023 | COMPLETED | | Yes | Yes | |
| 302-006 | 13JUN2023 | 13JUN2023 | COMPLETED | | Yes | Yes | |
| 302-007 | 14JUN2023 | 14JUN2023 | COMPLETED | | Yes | Yes | |
| 302-008 | 14JUN2023 | 14JUN2023 | COMPLETED | | Yes | Yes | |
| 302-009 | 15JUN2023 | 15JUN2023 | COMPLETED | | Yes | Yes | |
| 302-010 | 15JUN2023 | 15JUN2023 | COMPLETED | | Yes | Yes | |
| 302-011 | 16JUN2023 | 16JUN2023 | COMPLETED | | Yes | Yes | |
| 302-012 | 16JUN2023 | 16JUN2023 | COMPLETED | | Yes | Yes | |
| 302-013 | 20JUN2023 | 20JUN2023 | COMPLETED | | Yes | Yes | |
| 302-014 | 21JUN2023 | 21JUN2023 | COMPLETED | | Yes | Yes | |
| 302-015 | 21JUN2023 | 21JUN2023 | COMPLETED | | Yes | No | Rhythm strip not uploaded |
| 302-016 | 22JUN2023 | 22JUN2023 | COMPLETED | | Yes | Yes | |
| 302-017 | 22JUN2023 | 22JUN2023 | COMPLETED | | Yes | Yes | |

Listing 16.2.1.1 Subject Disposition All-Enrolled Population

| Subject<br>ID | Date of<br>Informed<br>Consent | Completion or<br>Discontinuation<br>Date | Status | Reason for Discontinuation | ITC<br>Population | PP<br>Population | Reason ITC subject is excluded from PP population |
|---|---|---|---|---|---|---|---|
| 302-018 | 22JUN2023 | 22JUN2023 | COMPLETED | | Yes | Yes | |
| 302-019 | 23JUN2023 | 23JUN2023 | COMPLETED | | Yes | Yes | |
| 302-020 | 27JUN2023 | 27JUN2023 | COMPLETED | | Yes | Yes | |
| 302-021 | 28JUN2023 | 28JUN2023 | COMPLETED | | Yes | Yes | |
| 304-001 | 20JUN2023 | 20JUN2023 | COMPLETED | | Yes | Yes | |
| 304-002 | 20JUN2023 | 20JUN2023 | DISCONTINUED | PROTOCOL<br>DEVIATION | No | No | Rhythm strip not uploaded |
| 304-003 | 21JUN2023 | 21JUN2023 | COMPLETED | | Yes | Yes | |
| 304-004 | 21JUN2023 | 21JUN2023 | COMPLETED | | Yes | Yes | |
| 304-005 | 22JUN2023 | 22JUN2023 | COMPLETED | | Yes | Yes | |
| 304-006 | 22JUN2023 | 22JUN2023 | COMPLETED | | Yes | Yes | |
| 304-007 | 27JUN2023 | 27JUN2023 | COMPLETED | | Yes | Yes | |
| 304-008 | 27JUN2023 | 27JUN2023 | COMPLETED | | Yes | Yes | |
| 304-009 | 27JUN2023 | 27JUN2023 | COMPLETED | | Yes | Yes | |
| 304-010 | 28JUN2023 | 28JUN2023 | COMPLETED | | Yes | Yes | |
| 304-011 | 28JUN2023 | 28JUN2023 | COMPLETED | | Yes | Yes | |
| 304-012 | 28JUN2023 | 28JUN2023 | COMPLETED | | Yes | Yes | |
| 304-013 | 29JUN2023 | 29JUN2023 | COMPLETED | | Yes | Yes | |
| 305-001 | 06JUN2023 | 06JUN2023 | COMPLETED | | Yes | No | Rhythm strip not uploaded |
| 305-002 | 06JUN2023 | 06JUN2023 | COMPLETED | | Yes | No | Rhythm strip not uploaded |
| 305-003 | 08JUN2023 | 08JUN2023 | COMPLETED | | Yes | No | Rhythm strip not uploaded |

Listing 16.2.1.1 Subject Disposition All-Enrolled Population

| Subject<br>ID | Date of<br>Informed<br>Consent | Completion or<br>Discontinuation<br>Date | Status | Reason for Discontinuation | ITC<br>Population | PP<br>Population | Reason ITC subject is excluded from PP population |
|---|---|---|---|---|---|---|---|
| 305-004 | 09JUN2023 | 09JUN2023 | COMPLETED | | Yes | Yes | |
| 305-005 | 23JUN2023 | 23JUN2023 | COMPLETED | | Yes | Yes | |
| 305-006 | 23JUN2023 | 23JUN2023 | COMPLETED | | Yes | No | Rhythm strip not uploaded |
| 305-007 | 26JUN2023 | 26JUN2023 | COMPLETED | | Yes | No | Rhythm strip not uploaded |
| 305-008 | 26JUN2023 | 26JUN2023 | COMPLETED | | Yes | No | Rhythm strip not uploaded |
| 305-009 | 28JUN2023 | 28JUN2023 | COMPLETED | | Yes | Yes | |
| 305-010 | 29JUN2023 | 29JUN2023 | COMPLETED | | Yes | Yes | |
| 305-011 | 29JUN2023 | 29JUN2023 | DISCONTINUED | OTHER | No | No | Study closed prior to assessment. |
| 305-012 | 29JUN2023 | 29JUN2023 | COMPLETED | | Yes | Yes | |
| 306-001 | 22JUN2023 | 22JUN2023 | COMPLETED | | Yes | No | Rhythm strip not uploaded |
| 306-002 | 22JUN2023 | 22JUN2023 | COMPLETED | | Yes | No | Rhythm strip not uploaded |
| 306-003 | 26JUN2023 | 26JUN2023 | COMPLETED | | Yes | Yes | |
| 306-004 | 26JUN2023 | 26JUN2023 | COMPLETED | | Yes | No | The reference device does not collect data |
| 306-005 | 28JUN2023 | 28JUN2023 | COMPLETED | | Yes | Yes | |
| 306-006 | 28JUN2023 | 28JUN2023 | COMPLETED | | Yes | Yes | |
| 306-007 | 29JUN2023 | 29JUN2023 | COMPLETED | | Yes | Yes | |
| 307-001 | 14JUN2023 | 14JUN2023 | COMPLETED | | Yes | Yes | |
| 307-002 | 14JUN2023 | 14JUN2023 | COMPLETED | | Yes | Yes | |
| 307-003 | 22JUN2023 | 22JUN2023 | COMPLETED | | Yes | Yes | |
| 307-004 | 22JUN2023 | 22JUN2023 | COMPLETED | | Yes | Yes | |

Mindset Medical, LLC IVC-400-006


Listing 16.2.1.1 Subject Disposition All-Enrolled Population

| Subject<br>ID | Date of<br>Informed<br>Consent | Completion or<br>Discontinuation<br>Date | Status | Reason for Discontinuation | ITC<br>Population | PP<br>Population | Reason ITC subject is excluded from PP population |
|---|---|---|---|---|---|---|---|
| 307-005 | 22JUN2023 | 22JUN2023 | COMPLETED | | Yes | No | The reference device does not collect data |
| 307-006 | 23JUN2023 | 23JUN2023 | COMPLETED | | Yes | Yes | |
| 307-007 | 23JUN2023 | 23JUN2023 | DISCONTINUED | SCREEN FAILURE | No | No | |
| 307-008 | 23JUN2023 | 23JUN2023 | COMPLETED | | Yes | Yes | |
| 307-009 | 26JUN2023 | 26JUN2023 | COMPLETED | | Yes | Yes | |
| 307-010 | 26JUN2023 | 26JUN2023 | COMPLETED | | Yes | No | Thumb drive not recognized by pixel phone. USB was sent back to sponsor for review on 7/20/23 |
| 307-011 | 28JUN2023 | 28JUN2023 | COMPLETED | | Yes | Yes | |

# Listing 16.2.1.3 Protocol Deviation All-Enrolled Subjects

| Subject<br>ID | Date of Deviation | Type of Deviation | Specification for Other | Brief Description of Deviation |
|---|---|---|---|---|
| 301-015 | 21JUN2023 | Other | The ECG was conducted but not uploaded to the drive | t The first ECG that I performed on the subject was not saved due to the disk drive was not in the ecg |
| 302-019 | 23JUN2023 | Deviation From<br>Protocol Defined<br>Procedure | | ECG limb leads were inadvertently reversed. |
| 304-002 | 20JUN2023 | Deviation From<br>Protocol Defined<br>Procedure | | PR PRO's were not completed per protocol. |
| 305-001 | 06JUN2023 | Deviation From<br>Protocol Defined<br>Procedure | | PRO HR data not captured despite multiple attempts and 2nd visit attempts per PM instructions. |
| 305-002 | 06JUN2023 | Deviation From<br>Protocol Defined<br>Procedure | | The second PRO assessment was not completed per protocol per PM instruction. |
| 306-001 | 22JUN2023 | Deviation From<br>Protocol Defined<br>Procedure | | Leads on ECG were reversed |
| | | | | Less than 2 PROs collected in the mainstudy. |

| Subject | Did the subject meet all the inclusion and none of the | | |
|---|---|---|---|
| ID | exclusion criteria? | Criterion Type | Description |
| 301-001 | Yes | | |
| 301-002 | Yes | | |
| 301-003 | Yes | | |
| 301-004 | Yes | | |
| 301-005 | Yes | | |
| 301-006 | Yes | | |
| 301-007 | No | EXCLUSION | SUBJECTS WITH CARDIAC ARRHYTHMIA |
| 301-008 | Yes | | |
| 301-009 | Yes | | |
| 301-010 | Yes | | |
| 301-011 | Yes | | |
| 301-012 | Yes | | |
| 301-013 | Yes | | |
| 301-014 | Yes | | |
| 301-015 | Yes | | |
| 301-016 | Yes | | |
| 301-017 | Yes | | |
| 301-018 | Yes | | |
| 301-019 | Yes | | |

| 0.1.1.1 | Did the subject meet all the | | |
|---|---|---|---|
| Subject<br>ID | inclusion and none of the exclusion criteria? | Criterion Type | Description |
| 301-020 | Yes | | |
| 301-021 | Yes | | |
| 301-022 | Yes | | |
| 302-001 | Yes | | |
| 302-002 | Yes | | |
| 302-003 | Yes | | |
| 302-004 | Yes | | |
| 302-005 | Yes | | |
| 302-006 | Yes | | |
| 302-007 | Yes | | |
| 302-008 | Yes | | |
| 302-009 | Yes | | |
| 302-010 | Yes | | |
| 302-011 | Yes | | |
| 302-012 | Yes | | |
| 302-013 | Yes | | |
| 302-014 | Yes | | |
| 302-015 | Yes | | |
| 302-016 | Yes | | |
| 302-017 | Yes | | |

| 0.1.1.1 | Did the subject meet all the | | |
|---|---|---|---|
| Subject<br>ID | inclusion and none of the exclusion criteria? | Criterion Type | Description |
| 302-018 | Yes | | |
| 302-019 | Yes | | |
| 302-020 | Yes | | |
| 302-021 | Yes | | |
| 304-001 | Yes | | |
| 304-002 | Yes | | |
| 304-003 | Yes | | |
| 304-004 | Yes | | |
| 304-005 | Yes | | |
| 304-006 | Yes | | |
| 304-007 | Yes | | |
| 304-008 | Yes | | |
| 304-009 | Yes | | |
| 304-010 | Yes | | |
| 304-011 | Yes | | |
| 304-012 | Yes | | |
| 304-013 | Yes | | |
| 305-001 | Yes | | |
| 305-002 | Yes | | |
| 305-003 | Yes | | |

| Subject | Did the subject meet all the inclusion and none of the | | |
|---|---|---|---|
| ID | exclusion criteria? | Criterion Type | Description |
| 305-004 | Yes | | |
| 305-005 | Yes | | |
| 305-006 | Yes | | |
| 305-007 | Yes | | |
| 305-008 | Yes | | |
| 305-009 | Yes | | |
| 305-010 | Yes | | |
| 305-011 | Yes | | |
| 305-012 | Yes | | |
| 306-001 | Yes | | |
| 306-002 | Yes | | |
| 306-003 | Yes | | |
| 306-004 | Yes | | |
| 306-005 | Yes | | |
| 306-006 | Yes | | |
| 306-007 | Yes | | |
| 307-001 | Yes | | |
| 307-002 | Yes | | |
| 307-003 | Yes | | |
| 307-004 | Yes | | |

Mindset Medical, LLC IVC-400-006


#### Listing 16.2.1.2 Eligibility Criteria All-Enrolled Population

| Subject<br>ID | Did the subject meet all the inclusion and none of the exclusion criteria? | Criterion Type | Description |
|---|---|---|---|
| 307-005 | Yes | | |
| 307-006 | Yes | | |
| 307-007 | No | EXCLUSION | SUBJECTS WITH CARDIAC ARRHYTHMIA |
| 307-008 | Yes | | |
| 307-009 | Yes | | |
| 307-010 | Yes | | |
| 307-011 | Yes | | |

Mindset Medical, LLC IVC-400-006


Listing 16.2.6.1

IVC App Pulse Rate and ECG Reference Device Heart Rate

ITC Population

| Subject ID | Session | Was the pulse rate taken by IVC? | Reason Pulse<br>was Not Taken | | Reason ECG<br>was Not<br>performed | Was ECG<br>Strip<br>Uploaded? | Reason ECG<br>Strip Was<br>Not Uploaded | Reason not<br>able to<br>Analyze | Pulse<br>Rate (BPM)<br>by IVC app | ECG<br>Reference<br>Device<br>Heart<br>Rate (BPM) |
|---|---|---|---|---|---|---|---|---|---|---|
| 301-001 | 1 | No | App not able to measure vitals | Yes | | Yes | | Null IVC<br>solution | | |
| | 2 | No | App not able to measure vitals | Yes | | Yes | | Null IVC solution | | |
| 301-002 | 1 | Yes | | Yes | | Yes | | | 60 | 60 |
| | 2 | Yes | | Yes | | Yes | | | 66 | 62 |
| 301-003 | 1 | No | App was not able to measure vitals | No | | Yes | | | | |
| | 2 | No | App was not able to measure vitals | No | | Yes | | | | |
| 301-004 | 1 | Yes | | Yes | | Yes | | | 69 | 69 |
| | 2 | Yes | | Yes | | Yes | | | 67 | 68 |
| 301-005 | 1 | Yes | | Yes | | Yes | | | 57 | 58 |
| | 2 | Yes | | Yes | | Yes | | | 57 | 57 |
| 301-006 | 1 | Yes | | Yes | | Yes | | | 69 | 69 |
| | 2 | Yes | | Yes | | Yes | | | 66 | 66 |

ITC = Intent-to-Capture.

Mindset Medical, LLC IVC-400-006


Listing 16.2.6.1

IVC App Pulse Rate and ECG Reference Device Heart Rate

ITC Population

| Subject<br>ID | Session | Was the pulse rate take by IVC? | n Reason Pulse Was ECG<br>was Not Taken performed? | Reason ECG<br>was Not<br>performed | Was ECG<br>Strip<br>Uploaded? | Reason ECG<br>Strip Was<br>Not Uploaded | Reason not able to Analyze | Pulse<br>Rate (BPM) | |
|---|---|---|---|---|---|---|---|---|---|
| 301-008 | 1 | | <del>-</del> | perrormed | - | Not opioaded | Allalyze | | Rate (BPM) |
| 301-008 | 1 | Yes | Yes | | Yes | | | 67 | 67 |
| | 2 | Yes | Yes | | Yes | | | 68 | 69 |
| 301-009 | 1 | Yes | Yes | | Yes | | | 71 | 70 |
| | 2 | Yes | Yes | | Yes | | | 71 | 71 |
| 301-010 | 1 | Yes | Yes | | Yes | | | 81 | 81 |
| | 2 | Yes | Yes | | Yes | | | 79 | 78 |
| 301-011 | 1 | Yes | Yes | | Yes | | | 64 | 65 |
| | 2 | Yes | Yes | | Yes | | | 60 | 61 |
| 301-012 | 1 | Yes | Yes | | Yes | | | 76 | 77 |
| | 2 | Yes | Yes | | Yes | | | 78 | 78 |
| 301-013 | 1 | Yes | Yes | | Yes | | | 72 | 72 |
| | 2 | Yes | Yes | | Yes | | | 73 | 74 |
| 301-014 | 1 | Yes | Yes | | Yes | | | 67 | 67 |

ITC = Intent-to-Capture.

Mindset Medical, LLC IVC-400-006


Listing 16.2.6.1

IVC App Pulse Rate and ECG Reference Device Heart Rate

ITC Population

| Subject | | Was the pulse | n Reason Pulse | Mag. ECC | Reason ECG<br>was Not | Was ECG<br>Strip | Reason ECG<br>Strip Was | Reason not able to | Pulse<br>Rate (BPM) | ECG<br>Reference<br>Device |
|---|---|---|---|---|---|---|---|---|---|---|
| ID | Session | by IVC? | was Not Taken | | performed | Uploaded? | Not Uploaded | | | Rate (BPM) |
| 301-014 | 2 | Yes | | Yes | • | Yes | * | | 68 | 69 |
| 301-015 | 1 | Yes | | No | | Yes | | | 70 | |
| | 2 | Yes | | Yes | | Yes | | | 67 | 66 |
| 301-016 | 1 | Yes | | Yes | | Yes | | | 73 | 73 |
| | 2 | Yes | | Yes | | Yes | | | 73 | 73 |
| 301-017 | 1 | Yes | | Yes | | Yes | | | 84 | 83 |
| | 2 | Yes | | Yes | | Yes | | | 83 | 83 |
| 301-018 | 1 | Yes | | Yes | | Yes | | | 67 | 67 |
| | 2 | Yes | | Yes | | Yes | | | 67 | 67 |
| 301-019 | 1 | Yes | | Yes | | Yes | | | 60 | 60 |
| | 2 | Yes | | Yes | | Yes | | | 60 | 60 |
| 301-020 | 1 | No | App not able | Yes | | Yes | | Null IVC | | |
| | | | to measure<br>vitals | | | | | solution | | |
| | 2 | No | App not able | Yes | | Yes | | Null IVC | | |
| | | | to measure<br>vitals | | | | | solution | | |
| 301-021 | 1 | Yes | | Yes | | Yes | | | 54 | 53 |

ITC = Intent-to-Capture.

Mindset Medical, LLC

IVC-400-006


Listing 16.2.6.1

IVC App Pulse Rate and ECG Reference Device Heart Rate

ITC Population

| Subject<br>ID | Session | Was the pulse rate take by IVC? | n Reason Pulse Was ECG<br>was Not Taken performed? | Reason ECG<br>was Not<br>performed | Was ECG<br>Strip<br>Uploaded? | Reason ECG<br>Strip Was<br>Not Uploaded | Reason not<br>able to<br>Analyze | Pulse<br>Rate (BPM)<br>by IVC app | ECG<br>Reference<br>Device<br>Heart<br>Rate (BPM) |
|---|---|---|---|---|---|---|---|---|---|
| 301-021 | 2 | Yes | Yes | | Yes | | | 53 | 53 |
| 301-022 | 1 | Yes | Yes | | Yes | | | 61 | 61 |
| | 2 | Yes | Yes | | Yes | | | 64 | 63 |
| 302-001 | 1 | Yes | Yes | | Yes | | | 80 | 80 |
| | 2 | Yes | Yes | | Yes | | | 79 | 79 |
| 302-002 | 1 | Yes | Yes | | Yes | | | 81 | 80 |
| | 2 | Yes | Yes | | Yes | | | 80 | 79 |
| 302-003 | 1 | Yes | Yes | | Yes | | | 65 | 67 |
| | 2 | Yes | Yes | | Yes | | | 68 | 68 |
| 302-004 | 1 | Yes | Yes | | Yes | | | 60 | 61 |
| | 2 | Yes | Yes | | Yes | | | 61 | 62 |
| 302-005 | 1 | Yes | Yes | | Yes | | | 69 | 69 |
| | 2 | Yes | Yes | | Yes | | | 69 | 69 |
| 302-006 | 1 | Yes | Yes | | Yes | | | 78 | 79 |

ITC = Intent-to-Capture.

Mindset Medical, LLC IVC-400-006


Listing 16.2.6.1

IVC App Pulse Rate and ECG Reference Device Heart Rate

ITC Population

| Subject<br>ID | Session | Was the pulse rate taker by IVC? | n Reason Pulse Was ECG<br>was Not Taken performed? | Reason ECG<br>was Not<br>performed | Was ECG<br>Strip<br>Uploaded? | Reason ECG<br>Strip Was<br>Not Uploaded | Reason not<br>able to<br>Analyze | Pulse<br>Rate (BPM)<br>by IVC app | ECG<br>Reference<br>Device<br>Heart<br>Rate (BPM) |
|---|---|---|---|---|---|---|---|---|---|
| 302-006 | 2 | Yes | Yes | | Yes | | | 78 | 78 |
| 302-007 | 1 | Yes | Yes | | Yes | | | 64 | 64 |
| | 2 | Yes | Yes | | Yes | | | 64 | 64 |
| 302-008 | 1 | Yes | Yes | | Yes | | | 53 | 54 |
| | 2 | Yes | Yes | | Yes | | | 55 | 55 |
| 302-009 | 1 | Yes | Yes | | Yes | | | 53 | 53 |
| | 2 | Yes | Yes | | Yes | | | 53 | 53 |
| 302-010 | 1 | Yes | Yes | | Yes | | | 57 | 57 |
| | 2 | Yes | Yes | | Yes | | | 54 | 55 |
| 302-011 | 1 | Yes | Yes | | Yes | | | 67 | 68 |
| | 2 | Yes | Yes | | Yes | | | 71 | 70 |
| 302-012 | 1 | Yes | Yes | | Yes | | | 64 | 64 |
| | 2 | Yes | Yes | | Yes | | | 64 | 64 |
| 302-013 | 1 | Yes | Yes | | Yes | | | 75 | 75 |

ITC = Intent-to-Capture.

Mindset Medical, LLC IVC-400-006


Listing 16.2.6.1

IVC App Pulse Rate and ECG Reference Device Heart Rate

ITC Population

| Subject<br>ID | Session | Was the pulse rate taken by IVC? | Reason Pulse<br>was Not Taken | | Reason ECG<br>was Not<br>performed | Was ECG<br>Strip<br>Uploaded? | Reason ECG<br>Strip Was<br>Not Uploaded | Reason not<br>able to<br>Analyze | Pulse<br>Rate (BPM)<br>by IVC app | ECG<br>Reference<br>Device<br>Heart<br>Rate (BPM) |
|---|---|---|---|---|---|---|---|---|---|---|
| 302-013 | 2 | Yes | | Yes | | Yes | | | 75 | 75 |
| 302-014 | 1 | Yes | | Yes | | Yes | | | 76 | 76 |
| | 2 | Yes | | Yes | | Yes | | | 78 | 78 |
| 302-015 | 1 | No | App not able<br>to measure<br>vitals | Yes | | Yes | | null IVC<br>solution | | |
| | 2 | No | App not able to measure vitals | Yes | | Yes | | null IVC<br>solution | | |
| 302-016 | 1 | Yes | | Yes | | Yes | | | 60 | 60 |
| | 2 | Yes | | Yes | | Yes | | | 61 | 61 |
| 302-017 | 1 | Yes | | Yes | | Yes | | | 86 | 87 |
| | 2 | Yes | | Yes | | Yes | | | 87 | 87 |
| 302-018 | 1 | Yes | | Yes | | Yes | | | 103 | 103 |
| | 2 | Yes | | No | | Yes | | | 105 | |
| 302-019 | 1 | Yes | | Yes | | Yes | | | 50 | 50 |
| | 2 | Yes | | Yes | | Yes | | | 50 | 50 |
| 302-020 | 1 | Yes | | Yes | | Yes | | | 85 | 84 |

ITC = Intent-to-Capture.

Mindset Medical, LLC IVC-400-006


Listing 16.2.6.1

IVC App Pulse Rate and ECG Reference Device Heart Rate

ITC Population

| | | Was the | | | C Was ECC | | | | ECG<br>Reference |
|---|---|---|---|---|---|---|---|---|---|
| Subject | | pulse<br>rate take | n Reason Pulse Was ECG | Reason ECG<br>was Not | Was ECG<br>Strip | Reason ECG<br>Strip Was | Reason not able to | Pulse<br>Rate (BPM) | Device<br>Heart |
| ID | Session | by IVC? | was Not Taken performed? | performed | Uploaded? | Not Uploaded | Analyze | by IVC app | Rate (BPM) |
| 302-020 | 2 | Yes | Yes | | Yes | | | 82 | 83 |
| 302-021 | 1 | Yes | Yes | | Yes | | | 74 | 75 |
| | 2 | Yes | Yes | | Yes | | | 78 | 79 |
| 304-001 | 1 | Yes | Yes | | Yes | | | 67 | 68 |
| | 2 | Yes | Yes | | Yes | | | 71 | 70 |
| 304-003 | 1 | Yes | Yes | | Yes | | | 53 | 53 |
| | 2 | Yes | Yes | | Yes | | | 53 | 52 |
| 304-004 | 1 | Yes | Yes | | Yes | | | 96 | 95 |
| | 2 | Yes | Yes | | Yes | | | 96 | 96 |
| 304-005 | 1 | Yes | Yes | | Yes | | | 71 | 70 |
| | 2 | Yes | Yes | | Yes | | | 71 | 70 |
| 304-006 | 1 | Yes | Yes | | Yes | | | 78 | 79 |

ITC = Intent-to-Capture.

Mindset Medical, LLC IVC-400-006


Listing 16.2.6.1

IVC App Pulse Rate and ECG Reference Device Heart Rate

ITC Population

| Subject<br>ID | Session | Was the pulse rate taker by IVC? | n Reason Pulse Was ECG<br>was Not Taken performed? | Reason ECG<br>was Not<br>performed | Was ECG<br>Strip<br>Uploaded? | Reason ECG<br>Strip Was<br>Not Uploaded | Reason not<br>able to<br>Analyze | Pulse<br>Rate (BPM)<br>by IVC app | ECG<br>Reference<br>Device<br>Heart<br>Rate (BPM) |
|---|---|---|---|---|---|---|---|---|---|
| 304-006 | 2 | Yes | Yes | | Yes | <del>-</del> | <del>_</del> | 78 | 78 |
| 304-007 | 1 | Yes | Yes | | Yes | | | 68 | 69 |
| | 2 | Yes | Yes | | Yes | | | 74 | 73 |
| 304-008 | 1 | Yes | Yes | | Yes | | | 74 | 73 |
| | 2 | Yes | Yes | | Yes | | | 75 | 75 |
| 304-009 | 1 | Yes | Yes | | Yes | | | 78 | 79 |
| | 2 | Yes | Yes | | Yes | | | 78 | 77 |
| 304-010 | 1 | Yes | Yes | | Yes | | | 67 | 67 |
| | 2 | Yes | Yes | | Yes | | | 67 | 67 |
| 304-011 | 1 | Yes | Yes | | Yes | | | 75 | 74 |
| | 2 | Yes | Yes | | Yes | | | 74 | 74 |
| 304-012 | 1 | Yes | Yes | | Yes | | | 71 | 70 |
| | 2 | Yes | Yes | | Yes | | | 68 | 69 |
| 304-013 | 1 | Yes | Yes | | Yes | | | 71 | 70 |

ITC = Intent-to-Capture.

Mindset Medical, LLC IVC-400-006


Listing 16.2.6.1

IVC App Pulse Rate and ECG Reference Device Heart Rate

ITC Population

| Subject<br>ID | Session | Was the pulse rate taken by IVC? | Reason Pulse Was ECG<br>was Not Taken performed? | Reason ECG<br>was Not<br>performed | Was ECG<br>Strip<br>Uploaded? | Reason ECG<br>Strip Was<br>Not Uploaded | Reason not<br>able to<br>Analyze | Pulse<br>Rate (BPM)<br>by IVC app | | e |
|---|---|---|---|---|---|---|---|---|---|---|
| 304-013 | 2 | Yes | Yes | | Yes | | | 73 | 72 | |
| 305-001 | 1 | No | app unable to Yes measure | | Yes | | Null IVC solution | | | |
| | 2 | No | app unable to No measure | | Yes | | | | | |
| 305-002 | 1 | No | app not able Yes<br>to measure | | Yes | | Null IVC solution | | | |
| | 2 | No | The second PRONo assessment was not completed per protocol per PM instruction. | | Yes | | | | | |
| 305-003 | 1 | No | App not able No to measure vitals. | | Yes | | | | | |
| | 2 | No | App not able No to measure vitals. | | Yes | | | | | |

ITC = Intent-to-Capture.

Mindset Medical, LLC

IVC-400-006


Listing 16.2.6.1

IVC App Pulse Rate and ECG Reference Device Heart Rate

ITC Population

| Subject<br>ID | Session | Was the pulse rate take by IVC? | n Reason Pulse Was ECG<br>was Not Taken performed: | Reason ECG<br>was Not<br>performed | Was ECG<br>Strip<br>Uploaded? | Reason ECG<br>Strip Was<br>Not Uploaded | Reason not<br>able to<br>Analyze | Pulse<br>Rate (BPM)<br>by IVC app | ECG<br>Reference<br>Device<br>Heart<br>Rate (BPM) |
|---|---|---|---|---|---|---|---|---|---|
| 305-004 | 1 | Yes | Yes | <del>_</del> | Yes | - | <del>-</del> | 64 | 65 |
| | 2 | Yes | Yes | | Yes | | | 64 | 64 |
| 305-005 | 1 | Yes | Yes | | Yes | | | 50 | 49 |
| | 2 | Yes | Yes | | Yes | | | 50 | 49 |
| 305-006 | 1 | No | App unable to Yes measure | | Yes | | Null IVC solution | | |
| | 2 | No | App unable to Yes measure | | Yes | | Null IVC solution | | |
| 305-007 | 1 | No | App unable to Yes measure | | Yes | | Null IVC solution | | |
| | 2 | No | App unable to Yes measure | | Yes | | Null IVC solution | | |
| 305-008 | 1 | No | App unable to Yes measure | | Yes | | Null IVC solution | | |
| | 2 | No | App unable to Yes measure | | Yes | | Null IVC solution | | |
| 305-009 | 1 | Yes | Yes | | Yes | | | 71 | 71 |
| | 2 | Yes | Yes | | Yes | | | 73 | 73 |
| 305-010 | 1 | Yes | Yes | | Yes | | | 53 | 53 |
| | 2 | Yes | Yes | | Yes | | | 52 | 53 |
| 305-012 | 1 | Yes | Yes | | Yes | | | 68 | 68 |
| | 2 | Yes | Yes | | Yes | | | 73 | 72 |
| 306-001 | 1 | No | App not able Yes<br>to measure<br>vitals | | Yes | | Null IVC<br>solution | | |
| | 2 | No | App not able No<br>to measure<br>vitals | | Yes | | | | |
| 306-002 | 1 | No | App not able No<br>to measure<br>vitals | | Yes | | | | |

ITC = Intent-to-Capture.

Mindset Medical, LLC IVC-400-006 

Listing 16.2.6.1

IVC App Pulse Rate and ECG Reference Device Heart Rate

ITC Population

| Subject ID | Session | Was the pulse rate taken by IVC? | Reason Pulse<br>was Not Taken | | Reason ECG<br>was Not<br>performed | Was ECG<br>Strip<br>Uploaded? | Reason ECG<br>Strip Was<br>Not Uploaded | Reason not<br>able to<br>Analyze | Pulse<br>Rate (BPM)<br>by IVC app | ECG<br>Reference<br>Device<br>Heart<br>Rate (BPM) |
|---|---|---|---|---|---|---|---|---|---|---|
| 306-002 | 2 | No | App not able to measure vitals | No | | Yes | | | | |
| 306-003 | 1 | Yes | | No | | Yes | | | 95 | |
| | 2 | Yes | | Yes | | Yes | | | 93 | 94 |
| 306-004 | 1 | No | <pre>app not able to measure vitals</pre> | Yes | | Yes | | Null IVC<br>solution | | |
| | 2 | Yes | | No | | Yes | | | 60 | |
| 306-005 | 1 | Yes | | Yes | | Yes | | | 63 | 62 |
| | 2 | Yes | | Yes | | Yes | | | 60 | 61 |
| 306-006 | 1 | Yes | | Yes | | Yes | | | 87 | 88 |
| | 2 | Yes | | Yes | | Yes | | | 87 | 87 |
| 306-007 | 1 | Yes | | Yes | | Yes | | | 77 | 77 |
| | 2 | Yes | | Yes | | Yes | | | 75 | 75 |
| 307-001 | 1 | Yes | | Yes | | Yes | | | 73 | 73 |
| | 2 | Yes | | Yes | | Yes | | | 75 | 74 |
| 307-002 | 1 | Yes | | Yes | | Yes | | | 84 | 83 |

ITC = Intent-to-Capture.
Mindset Medical, LLC IVC-400-006 

Listing 16.2.6.1

IVC App Pulse Rate and ECG Reference Device Heart Rate

ITC Population

| Subject<br>ID | Session | Was the pulse rate taken by IVC? | Reason Pulso | e Was ECG<br>en performed? | Reason ECG<br>was Not<br>performed | Was ECG<br>Strip<br>Uploaded? | Reason ECG<br>Strip Was<br>Not Uploaded | Reason not<br>able to<br>Analyze | Pulse<br>Rate (BPM)<br>by IVC app | ECG<br>Reference<br>Device<br>Heart<br>Rate (BPM) |
|---|---|---|---|---|---|---|---|---|---|---|
| 307-002 | 2 | Yes | | Yes | | Yes | | | 82 | 83 |
| 307-003 | 1 | Yes | | Yes | | Yes | | | 62 | 63 |
| | 2 | Yes | | Yes | | Yes | | | 62 | 62 |
| 307-004 | 1 | Yes | | Yes | | Yes | | | 64 | 65 |
| | 2 | Yes | | Yes | | Yes | | | 61 | 61 |
| 307-005 | 1 | Yes | | No | | Yes | | | 92 | |
| | 2 | Yes | | No | | Yes | | | 92 | |
| 307-006 | 1 | Yes | | Yes | | Yes | | | 77 | 76 |
| | 2 | Yes | | Yes | | Yes | | | 80 | 80 |
| 307-008 | 1 | No | app unable | to Yes | | Yes | | Null IVC | | |
| | | | measure | | | | | solution | | |
| | 2 | Yes | | Yes | | Yes | | | 79 | 79 |
| 307-009 | 1 | No | unable to | Yes | | Yes | | Null IVC | | |
| | | | measure<br>vitals | | | | | solution | | |

ITC = Intent-to-Capture.

Mindset Medical, LLC IVC-400-006 

Listing 16.2.6.1

IVC App Pulse Rate and ECG Reference Device Heart Rate

ITC Population

| Subject ID | Session | Was the pulse rate taker by IVC? | n Reason Pulse Was ECG<br>was Not Taken performed? | Reason ECG<br>was Not<br>performed | Was ECG<br>Strip<br>Uploaded? | Reason ECG<br>Strip Was<br>Not Uploaded | Reason not<br>able to<br>Analyze | Pulse<br>Rate (BPM)<br>by IVC app | |
|---|---|---|---|---|---|---|---|---|---|
| 307-009 | 2 | Yes | Yes | | Yes | | | 75 | 74 |
| 307-010 | 1 | No | no Pulse Rate No<br>obtained- App<br>not able to<br>measure<br>vitals | | No | Thumb drive not recognized by pixel phone. USB was sent back to sponsor for review on 7/20/23 | | | |
| | 2 | No | no Pulse Rate No<br>obtained- App<br>not able to<br>measure<br>vitals | | No | Thumb drive not recognized by pixel phone. USB was sent back to sponsor for review on 7/20/23 | | | |
| 307-011 | 1 | Yes | Yes | | Yes | | | 60 | 59 |
| | 2 | Yes | Yes | | Yes | | | 57 | 58 |

ITC = Intent-to-Capture.

Mindset Medical, LLC IVC-400-006


Listing 16.2.4.1

Demographic and Other Baseline Characteristics

ITC Population

| Subject ID | Age<br>(years) | Sex | Race | Ethnicity | Fitzpatrick Scale<br>Assignment | Is the subject wearing Glasses ? | |
|---|---|---|---|---|---|---|---|
| 301-001 | 29 | Female | BLACK OR AFRICAN AMERICAN | NOT HISPANIC OR LATINO | 6 - Deeply Pigmented Dark Brown to<br>Black Skin | Yes | No |
| 301-002 | 36 | Female | BLACK OR AFRICAN AMERICAN | NOT HISPANIC OR LATINO | 5 - Dark Brown Skin | No | No |
| 301-003 | 43 | Male | BLACK OR AFRICAN AMERICAN | NOT HISPANIC OR LATINO | 5 - Dark Brown Skin | No | Yes |
| 301-004 | 51 | Male | WHITE | NOT HISPANIC OR LATINO | 2 - White Skin | Yes | Yes |
| 301-005 | 56 | Male | WHITE | HISPANIC OR LATINO | 3 - Light Brown Skin | Yes | No |
| 301-006 | 27 | Female | WHITE | NOT HISPANIC OR LATINO | 2 - White Skin | No | No |
| 301-008 | 70 | Female | WHITE | NOT HISPANIC OR LATINO | 1 - Pale White Skin | No | No |
| 301-009 | 69 | Female | WHITE | NOT HISPANIC OR LATINO | 2 - White Skin | Yes | No |
| 301-010 | 62 | Female | ASIAN | NOT HISPANIC OR LATINO | 4 - Moderate Brown Skin | No | No |
| 301-011 | 53 | Female | BLACK OR AFRICAN AMERICAN | NOT HISPANIC OR LATINO | 5 - Dark Brown Skin | Yes | No |
| 301-012 | 40 | Female | BLACK OR AFRICAN AMERICAN | NOT HISPANIC OR LATINO | 3 - Light Brown Skin | No | No |
| 301-013 | 60 | Female | WHITE | NOT HISPANIC OR LATINO | 1 - Pale White Skin | Yes | No |
| 301-014 | 35 | Male | WHITE | NOT HISPANIC OR LATINO | 3 - Light Brown Skin | No | No |
| 301-015 | 45 | Female | WHITE | NOT HISPANIC OR LATINO | 2 - White Skin | Yes | No |
| 301-016 | 37 | Female | WHITE | NOT HISPANIC OR LATINO | 1 - Pale White Skin | No | No |
| 301-017 | 67 | Female | WHITE | NOT HISPANIC OR LATINO | 2 - White Skin | Yes | No |
| 301-018 | 62 | Male | BLACK OR AFRICAN AMERICAN | NOT HISPANIC OR LATINO | 6 - Deeply Pigmented Dark Brown to<br>Black Skin | No | Yes |

ITC = Intent-to-Capture.

Mindset Medical, LLC IVC-400-006


Listing 16.2.4.1

Demographic and Other Baseline Characteristics

ITC Population

| Subject ID | Age<br>(years) | Sex | Race | Ethnicity | Fitzpatrick Scale<br>Assignment | Is the subject wearing Glasses ? | |
|---|---|---|---|---|---|---|---|
| 301-019 | 66 | Female | WHITE | NOT HISPANIC OR LATINO | 2 - White Skin | Yes | No |
| 301-020 | 33 | Female | BLACK OR AFRICAN AMERICAN | NOT HISPANIC OR LATINO | 6 - Deeply Pigmented Dark Brown to<br>Black Skin | No | No |
| 301-021 | 30 | Male | BLACK OR AFRICAN AMERICAN | NOT HISPANIC OR LATINO | 5 - Dark Brown Skin | No | Yes |
| 301-022 | 62 | Male | WHITE | NOT HISPANIC OR LATINO | 3 - Light Brown Skin | Yes | No |
| 302-001 | 48 | Male | WHITE | HISPANIC OR LATINO | 5 - Dark Brown Skin | No | Yes |
| 302-002 | 76 | Female | WHITE | NOT HISPANIC OR LATINO | 2 - White Skin | Yes | No |
| 302-003 | 32 | Male | BLACK OR AFRICAN AMERICAN | NOT HISPANIC OR LATINO | 6 - Deeply Pigmented Dark Brown to<br>Black Skin | No | Yes |
| 302-004 | 55 | Female | WHITE | NOT HISPANIC OR LATINO | 3 - Light Brown Skin | No | No |
| 302-005 | 53 | Female | WHITE | NOT HISPANIC OR LATINO | 1 - Pale White Skin | Yes | No |
| 302-006 | 61 | Male | ASIAN | NOT HISPANIC OR LATINO | 3 - Light Brown Skin | Yes | Yes |
| 302-007 | 65 | Female | WHITE | NOT HISPANIC OR LATINO | 2 - White Skin | No | No |
| 302-008 | 52 | Female | WHITE | HISPANIC OR LATINO | 3 - Light Brown Skin | No | No |
| 302-009 | 39 | Male | BLACK OR AFRICAN AMERICAN | NOT HISPANIC OR LATINO | 6 - Deeply Pigmented Dark Brown to<br>Black Skin | No | Yes |
| 302-010 | 43 | Male | NATIVE HAWAIIAN OR OTHER PACIFIC ISLANDER | NOT HISPANIC OR LATINO | 6 - Deeply Pigmented Dark Brown to<br>Black Skin | Yes | Yes |
| 302-011 | 22 | Female | BLACK OR AFRICAN AMERICAN | NOT HISPANIC OR LATINO | 5 - Dark Brown Skin | No | No |
| 302-012 | 44 | Male | WHITE | NOT HISPANIC OR LATINO | 2 - White Skin | No | Yes |
| 302-013 | 68 | Female | WHITE | NOT HISPANIC OR LATINO | 1 - Pale White Skin | No | No |
| 302-014 | 48 | Female | WHITE | NOT HISPANIC OR LATINO | 2 - White Skin | No | No |

ITC = Intent-to-Capture.

Mindset Medical, LLC IVC-400-006


Listing 16.2.4.1

Demographic and Other Baseline Characteristics

ITC Population

| Subject<br>ID | Age<br>(years) | Sex | Race | Ethnicity | Fitzpatrick Scale<br>Assignment | Is the subject wearing Glasses ? | |
|---|---|---|---|---|---|---|---|
| 302-015 | 44 | Male | BLACK OR AFRICAN AMERICAN | NOT HISPANIC OR LATINO | 5 - Dark Brown Skin | No | Yes |
| 302-016 | 22 | Male | BLACK OR AFRICAN AMERICAN | NOT HISPANIC OR LATINO | 6 - Deeply Pigmented Dark Brown to<br>Black Skin | No | No |
| 302-017 | 57 | Male | WHITE | NOT HISPANIC OR LATINO | 2 - White Skin | No | Yes |
| 302-018 | 32 | Female | ASIAN | NOT HISPANIC OR LATINO | 3 - Light Brown Skin | No | No |
| 302-019 | 42 | Male | WHITE | NOT HISPANIC OR LATINO | 2 - White Skin | No | Yes |
| 302-020 | 62 | Male | WHITE | NOT HISPANIC OR LATINO | 2 - White Skin | No | Yes |
| 302-021 | 44 | Female | WHITE | NOT HISPANIC OR LATINO | 2 - White Skin | No | No |
| 304-001 | 60 | Male | BLACK OR AFRICAN AMERICAN | NOT HISPANIC OR LATINO | 5 - Dark Brown Skin | No | Yes |
| 304-003 | 38 | Female | BLACK OR AFRICAN AMERICAN | NOT HISPANIC OR LATINO | 5 - Dark Brown Skin | No | No |
| 304-004 | 33 | Female | BLACK OR AFRICAN AMERICAN | NOT HISPANIC OR LATINO | 5 - Dark Brown Skin | No | No |
| 304-005 | 61 | Male | WHITE | NOT HISPANIC OR LATINO | 2 - White Skin | Yes | No |
| 304-006 | 69 | Female | WHITE | NOT HISPANIC OR LATINO | 2 - White Skin | No | No |
| 304-007 | 77 | Female | WHITE | NOT HISPANIC OR LATINO | 1 - Pale White Skin | Yes | No |
| 304-008 | 63 | Male | BLACK OR AFRICAN AMERICAN | NOT HISPANIC OR LATINO | 4 - Moderate Brown Skin | No | No |
| 304-009 | 55 | Male | WHITE | NOT HISPANIC OR LATINO | 2 - White Skin | No | Yes |
| 304-010 | 33 | Male | ASIAN | NOT HISPANIC OR LATINO | 2 - White Skin | No | No |
| 304-011 | 34 | Female | WHITE | NOT HISPANIC OR LATINO | 2 - White Skin | No | No |
| 304-012 | 53 | Female | WHITE | NOT HISPANIC OR LATINO | 3 - Light Brown Skin | No | No |

ITC = Intent-to-Capture.

Mindset Medical, LLC IVC-400-006


Listing 16.2.4.1

Demographic and Other Baseline Characteristics

ITC Population

| Subject ID | Age<br>(years) | Sex | Race | Ethnicity | Fitzpatrick Scale<br>Assignment | Is the subject wearing Glasses ? | |
|---|---|---|---|---|---|---|---|
| 304-013 | 27 | Male | WHITE | NOT HISPANIC OR LATINO | 2 - White Skin | No | Yes |
| 305-001 | 49 | Male | BLACK OR AFRICAN AMERICAN | NOT HISPANIC OR LATINO | 6 - Deeply Pigmented Dark Brown to<br>Black Skin | No | Yes |
| 305-002 | 51 | Female | BLACK OR AFRICAN AMERICAN | NOT HISPANIC OR LATINO | 6 - Deeply Pigmented Dark Brown to<br>Black Skin | No | No |
| 305-003 | 69 | Female | BLACK OR AFRICAN AMERICAN | NOT HISPANIC OR LATINO | 6 - Deeply Pigmented Dark Brown to Black Skin | No | No |
| 305-004 | 31 | Female | OTHER | HISPANIC OR LATINO | 2 - White Skin | No | No |
| 305-005 | 74 | Female | BLACK OR AFRICAN AMERICAN | NOT HISPANIC OR LATINO | 5 - Dark Brown Skin | No | No |
| 305-006 | 52 | Male | BLACK OR AFRICAN AMERICAN | NOT HISPANIC OR LATINO | 6 - Deeply Pigmented Dark Brown to<br>Black Skin | No | Yes |
| 305-007 | 46 | Female | BLACK OR AFRICAN AMERICAN | NOT HISPANIC OR LATINO | 5 - Dark Brown Skin | No | No |
| 305-008 | 38 | Male | BLACK OR AFRICAN AMERICAN | NOT HISPANIC OR LATINO | 5 - Dark Brown Skin | No | Yes |
| 305-009 | 62 | Female | WHITE | NOT HISPANIC OR LATINO | 2 - White Skin | Yes | No |
| 305-010 | 73 | Male | BLACK OR AFRICAN AMERICAN | NOT HISPANIC OR LATINO | 5 - Dark Brown Skin | Yes | Yes |
| 305-012 | 69 | Female | ASIAN | NOT HISPANIC OR LATINO | 3 - Light Brown Skin | Yes | No |
| 306-001 | 22 | Male | BLACK OR AFRICAN AMERICAN | NOT HISPANIC OR LATINO | 5 - Dark Brown Skin | No | Yes |
| 306-002 | 23 | Male | BLACK OR AFRICAN AMERICAN | NOT HISPANIC OR LATINO | 5 - Dark Brown Skin | No | Yes |
| 306-003 | 37 | Female | BLACK OR AFRICAN AMERICAN | NOT HISPANIC OR LATINO | 4 - Moderate Brown Skin | No | No |
| 306-004 | 38 | Male | BLACK OR AFRICAN AMERICAN | NOT HISPANIC OR LATINO | 6 - Deeply Pigmented Dark Brown to<br>Black Skin | No | Yes |
| 306-005 | 70 | Female | BLACK OR AFRICAN AMERICAN | NOT HISPANIC OR LATINO | 5 - Dark Brown Skin | No | No |
| 306-006 | 30 | Female | WHITE | NOT HISPANIC OR LATINO | 2 - White Skin | No | No |

ITC = Intent-to-Capture.

Mindset Medical, LLC IVC-400-006


Listing 16.2.4.1

Demographic and Other Baseline Characteristics

ITC Population

| Subject<br>ID | Age<br>(years) | Sex | Race | Ethnicity | Fitzpatrick Scale<br>Assignment | Is the subject wearing Glasses ? | |
|---|---|---|---|---|---|---|---|
| 306-007 | 36 | Female | WHITE | NOT HISPANIC OR LATINO | 2 - White Skin | No | No |
| 307-001 | 66 | Female | WHITE | NOT HISPANIC OR LATINO | 3 - Light Brown Skin | No | No |
| 307-002 | 66 | Male | AMERICAN INDIAN OR ALASKA<br>NATIVE/BLACK OR AFRICAN<br>AMERICAN | NOT HISPANIC OR LATINO | 5 - Dark Brown Skin | No | Yes |
| 307-003 | 24 | Male | WHITE | HISPANIC OR LATINO | 4 - Moderate Brown Skin | No | No |
| 307-004 | 34 | Male | WHITE | NOT HISPANIC OR LATINO | 3 - Light Brown Skin | No | Yes |
| 307-005 | 59 | Male | WHITE | NOT HISPANIC OR LATINO | 2 - White Skin | No | Yes |
| 307-006 | 23 | Male | AMERICAN INDIAN OR ALASKA<br>NATIVE | HISPANIC OR LATINO | 3 - Light Brown Skin | No | Yes |
| 307-008 | 44 | Male | WHITE | HISPANIC OR LATINO | 4 - Moderate Brown Skin | No | Yes |
| 307-009 | 63 | Male | BLACK OR AFRICAN AMERICAN | NOT HISPANIC OR LATINO | 5 - Dark Brown Skin | No | No |
| 307-010 | 44 | Male | BLACK OR AFRICAN AMERICAN | NOT HISPANIC OR LATINO | 5 - Dark Brown Skin | No | Yes |
| 307-011 | 58 | Male | WHITE | NOT HISPANIC OR LATINO | 2 - White Skin | No | Yes |

ITC = Intent-to-Capture.

Mindset Medical, LLC IVC-400-006
Page 1 of 2

 $\begin{tabular}{ll} Table 14.1.2.1 \\ Summary of Subject Demographic and Other Baseline Characteristics \\ ITC Population \\ \end{tabular}$ 

| | | Total |
|---|---|---|
| | | (N=82) |
| Characteristic | Statistic or Category | n (%) |
| Sex, n (%) | Male | 40 (48.8) |
| , , , | Female | 42 (51.2) |
| Ethnic Group, n (%) | Hispanic or Latino | 7 ( 8.5) |
| | Not Hispanic or Latino | 75 (91.5) |
| Race, n (%) | American Indian or Alaska Native/Black or African American | 1 (1.2) |
| | American Indian or Alaska Native | 1 (1.2) |
| | Asian | 5 ( 6.1) |
| | Black or African American | 32 (39.0) |
| | Native Hawaiian or Other Pacific Islander | 1 (1.2) |
| | White | 41 (50.0) |
| | Other | 1 ( 1.2) |
| Fitzpatrick Scale, n (%) | 1 - Pale White Skin | 6 (7.3) |
| - | 2 - White Skin | 26 (31.7) |
| | 3 - Light Brown Skin | 13 (15.9) |
| | 4 - Moderate Brown Skin | 5 ( 6.1) |
| | 5 - Dark Brown Skin | 20 (24.4) |
| | 6 - Deeply Pigmented Dark Brown to Black Skin | 12 (14.6) |
| Fitzpatrick Scale Group, n (%) [a] | Light | 32 (39.0) |
| | Medium | 18 (22.0) |
| | Dark | 32 (39.0) |

Program name: t 14 1 2 1.sas Run Date: 21NOV2023

 $<sup>% = 100 \</sup>times n/N.$  ITC = Intent-to-Capture.

<sup>[</sup>a] Fitzpatrick scale skin tones are grouped into light (Fitzpatrick 1 and 2), medium (Fitzpatrick 3 and 4) and dark (Fitzpatrick 5 and 6).

See Listing 16.2.4.1

Mindset Medical, LLC IVC-400-006
Page 2 of 2

 $\begin{tabular}{ll} Table 14.1.2.1 \\ Summary of Subject Demographic and Other Baseline Characteristics \\ ITC Population \\ \end{tabular}$ 

| Characteristic | Statistic or Category | Total<br>(N=82)<br>n (%) |
|----------------|-----------------------|--------------------------|
| Age (years) | n | 82 |
| nge (years) | Mean | 48.7 |
| | Standard deviation | 15.40 |
| | Median | 48.5 |
| | Minimum | 22 |
| | Maximum | 77 |

See Listing 16.2.4.1

Program name: t 14 1 2 1.sas Run Date: 21NOV2023

 $<sup>% = 100 \</sup>times n/N.$  ITC = Intent-to-Capture.

<sup>[</sup>a] Fitzpatrick scale skin tones are grouped into light (Fitzpatrick 1 and 2), medium (Fitzpatrick 3 and 4) and dark (Fitzpatrick 5 and 6).

Mindset Medical, LLC IVC-400-006


Listing 16.2.6.1

IVC App Pulse Rate and ECG Reference Device Heart Rate

ITC Population

| Subject ID | Session | Was the pulse rate taken by IVC? | Reason Pulse<br>was Not Taken | | Reason ECG<br>was Not<br>performed | Was ECG<br>Strip<br>Uploaded? | Reason ECG<br>Strip Was<br>Not Uploaded | Reason not<br>able to<br>Analyze | Pulse<br>Rate (BPM)<br>by IVC app | ECG<br>Reference<br>Device<br>Heart<br>Rate (BPM) |
|---|---|---|---|---|---|---|---|---|---|---|
| 301-001 | 1 | No | App not able to measure vitals | Yes | | Yes | | Null IVC<br>solution | | |
| | 2 | No | App not able to measure vitals | Yes | | Yes | | Null IVC solution | | |
| 301-002 | 1 | Yes | | Yes | | Yes | | | 60 | 60 |
| | 2 | Yes | | Yes | | Yes | | | 66 | 62 |
| 301-003 | 1 | No | App was not able to measure vitals | No | | Yes | | | | |
| | 2 | No | App was not able to measure vitals | No | | Yes | | | | |
| 301-004 | 1 | Yes | | Yes | | Yes | | | 69 | 69 |
| | 2 | Yes | | Yes | | Yes | | | 67 | 68 |
| 301-005 | 1 | Yes | | Yes | | Yes | | | 57 | 58 |
| | 2 | Yes | | Yes | | Yes | | | 57 | 57 |
| 301-006 | 1 | Yes | | Yes | | Yes | | | 69 | 69 |
| | 2 | Yes | | Yes | | Yes | | | 66 | 66 |

ITC = Intent-to-Capture.

Mindset Medical, LLC IVC-400-006


Listing 16.2.6.1

IVC App Pulse Rate and ECG Reference Device Heart Rate

ITC Population

| Subject<br>ID | Session | Was the pulse rate take by IVC? | n Reason Pulse Was ECG<br>was Not Taken performed? | Reason ECG<br>was Not<br>performed | Was ECG<br>Strip<br>Uploaded? | Reason ECG<br>Strip Was<br>Not Uploaded | Reason not able to Analyze | Pulse<br>Rate (BPM) | |
|---|---|---|---|---|---|---|---|---|---|
| 301-008 | 1 | | <del>-</del> | perrormed | - | Not opioaded | Allalyze | | Rate (BPM) |
| 301-008 | 1 | Yes | Yes | | Yes | | | 67 | 67 |
| | 2 | Yes | Yes | | Yes | | | 68 | 69 |
| 301-009 | 1 | Yes | Yes | | Yes | | | 71 | 70 |
| | 2 | Yes | Yes | | Yes | | | 71 | 71 |
| 301-010 | 1 | Yes | Yes | | Yes | | | 81 | 81 |
| | 2 | Yes | Yes | | Yes | | | 79 | 78 |
| 301-011 | 1 | Yes | Yes | | Yes | | | 64 | 65 |
| | 2 | Yes | Yes | | Yes | | | 60 | 61 |
| 301-012 | 1 | Yes | Yes | | Yes | | | 76 | 77 |
| | 2 | Yes | Yes | | Yes | | | 78 | 78 |
| 301-013 | 1 | Yes | Yes | | Yes | | | 72 | 72 |
| | 2 | Yes | Yes | | Yes | | | 73 | 74 |
| 301-014 | 1 | Yes | Yes | | Yes | | | 67 | 67 |

ITC = Intent-to-Capture.

Mindset Medical, LLC IVC-400-006


Listing 16.2.6.1

IVC App Pulse Rate and ECG Reference Device Heart Rate

ITC Population

| Subject | | Was the pulse | n Reason Pulse | Mag. ECC | Reason ECG<br>was Not | Was ECG<br>Strip | Reason ECG<br>Strip Was | Reason not able to | Pulse<br>Rate (BPM) | ECG<br>Reference<br>Device |
|---|---|---|---|---|---|---|---|---|---|---|
| ID | Session | by IVC? | was Not Taken | | performed | Uploaded? | Not Uploaded | | | Rate (BPM) |
| 301-014 | 2 | Yes | | Yes | • | Yes | * | | 68 | 69 |
| 301-015 | 1 | Yes | | No | | Yes | | | 70 | |
| | 2 | Yes | | Yes | | Yes | | | 67 | 66 |
| 301-016 | 1 | Yes | | Yes | | Yes | | | 73 | 73 |
| | 2 | Yes | | Yes | | Yes | | | 73 | 73 |
| 301-017 | 1 | Yes | | Yes | | Yes | | | 84 | 83 |
| | 2 | Yes | | Yes | | Yes | | | 83 | 83 |
| 301-018 | 1 | Yes | | Yes | | Yes | | | 67 | 67 |
| | 2 | Yes | | Yes | | Yes | | | 67 | 67 |
| 301-019 | 1 | Yes | | Yes | | Yes | | | 60 | 60 |
| | 2 | Yes | | Yes | | Yes | | | 60 | 60 |
| 301-020 | 1 | No | App not able | Yes | | Yes | | Null IVC | | |
| | | | to measure<br>vitals | | | | | solution | | |
| | 2 | No | App not able | Yes | | Yes | | Null IVC | | |
| | | | to measure<br>vitals | | | | | solution | | |
| 301-021 | 1 | Yes | | Yes | | Yes | | | 54 | 53 |

ITC = Intent-to-Capture.

Mindset Medical, LLC

IVC-400-006


Listing 16.2.6.1

IVC App Pulse Rate and ECG Reference Device Heart Rate

ITC Population

| Subject<br>ID | Session | Was the pulse rate take by IVC? | n Reason Pulse Was ECG<br>was Not Taken performed? | Reason ECG<br>was Not<br>performed | Was ECG<br>Strip<br>Uploaded? | Reason ECG<br>Strip Was<br>Not Uploaded | Reason not<br>able to<br>Analyze | Pulse<br>Rate (BPM)<br>by IVC app | ECG<br>Reference<br>Device<br>Heart<br>Rate (BPM) |
|---|---|---|---|---|---|---|---|---|---|
| 301-021 | 2 | Yes | Yes | | Yes | | | 53 | 53 |
| 301-022 | 1 | Yes | Yes | | Yes | | | 61 | 61 |
| | 2 | Yes | Yes | | Yes | | | 64 | 63 |
| 302-001 | 1 | Yes | Yes | | Yes | | | 80 | 80 |
| | 2 | Yes | Yes | | Yes | | | 79 | 79 |
| 302-002 | 1 | Yes | Yes | | Yes | | | 81 | 80 |
| | 2 | Yes | Yes | | Yes | | | 80 | 79 |
| 302-003 | 1 | Yes | Yes | | Yes | | | 65 | 67 |
| | 2 | Yes | Yes | | Yes | | | 68 | 68 |
| 302-004 | 1 | Yes | Yes | | Yes | | | 60 | 61 |
| | 2 | Yes | Yes | | Yes | | | 61 | 62 |
| 302-005 | 1 | Yes | Yes | | Yes | | | 69 | 69 |
| | 2 | Yes | Yes | | Yes | | | 69 | 69 |
| 302-006 | 1 | Yes | Yes | | Yes | | | 78 | 79 |

ITC = Intent-to-Capture.

Mindset Medical, LLC IVC-400-006


Listing 16.2.6.1

IVC App Pulse Rate and ECG Reference Device Heart Rate

ITC Population

| Subject<br>ID | Session | Was the pulse rate taker by IVC? | n Reason Pulse Was ECG<br>was Not Taken performed? | Reason ECG<br>was Not<br>performed | Was ECG<br>Strip<br>Uploaded? | Reason ECG<br>Strip Was<br>Not Uploaded | Reason not<br>able to<br>Analyze | Pulse<br>Rate (BPM)<br>by IVC app | ECG<br>Reference<br>Device<br>Heart<br>Rate (BPM) |
|---|---|---|---|---|---|---|---|---|---|
| 302-006 | 2 | Yes | Yes | | Yes | | | 78 | 78 |
| 302-007 | 1 | Yes | Yes | | Yes | | | 64 | 64 |
| | 2 | Yes | Yes | | Yes | | | 64 | 64 |
| 302-008 | 1 | Yes | Yes | | Yes | | | 53 | 54 |
| | 2 | Yes | Yes | | Yes | | | 55 | 55 |
| 302-009 | 1 | Yes | Yes | | Yes | | | 53 | 53 |
| | 2 | Yes | Yes | | Yes | | | 53 | 53 |
| 302-010 | 1 | Yes | Yes | | Yes | | | 57 | 57 |
| | 2 | Yes | Yes | | Yes | | | 54 | 55 |
| 302-011 | 1 | Yes | Yes | | Yes | | | 67 | 68 |
| | 2 | Yes | Yes | | Yes | | | 71 | 70 |
| 302-012 | 1 | Yes | Yes | | Yes | | | 64 | 64 |
| | 2 | Yes | Yes | | Yes | | | 64 | 64 |
| 302-013 | 1 | Yes | Yes | | Yes | | | 75 | 75 |

ITC = Intent-to-Capture.

Mindset Medical, LLC IVC-400-006


Listing 16.2.6.1

IVC App Pulse Rate and ECG Reference Device Heart Rate

ITC Population

| Subject<br>ID | Session | Was the pulse rate taken by IVC? | Reason Pulse<br>was Not Taken | | Reason ECG<br>was Not<br>performed | Was ECG<br>Strip<br>Uploaded? | Reason ECG<br>Strip Was<br>Not Uploaded | Reason not<br>able to<br>Analyze | Pulse<br>Rate (BPM)<br>by IVC app | ECG<br>Reference<br>Device<br>Heart<br>Rate (BPM) |
|---|---|---|---|---|---|---|---|---|---|---|
| 302-013 | 2 | Yes | | Yes | | Yes | | | 75 | 75 |
| 302-014 | 1 | Yes | | Yes | | Yes | | | 76 | 76 |
| | 2 | Yes | | Yes | | Yes | | | 78 | 78 |
| 302-015 | 1 | No | App not able to measure vitals | Yes | | Yes | | null IVC<br>solution | | |
| | 2 | No | App not able<br>to measure<br>vitals | Yes | | Yes | | null IVC<br>solution | | |
| 302-016 | 1 | Yes | | Yes | | Yes | | | 60 | 60 |
| | 2 | Yes | | Yes | | Yes | | | 61 | 61 |
| 302-017 | 1 | Yes | | Yes | | Yes | | | 86 | 87 |
| | 2 | Yes | | Yes | | Yes | | | 87 | 87 |
| 302-018 | 1 | Yes | | Yes | | Yes | | | 103 | 103 |
| | 2 | Yes | | No | | Yes | | | 105 | |
| 302-019 | 1 | Yes | | Yes | | Yes | | | 50 | 50 |
| | 2 | Yes | | Yes | | Yes | | | 50 | 50 |
| 302-020 | 1 | Yes | | Yes | | Yes | | | 85 | 84 |

ITC = Intent-to-Capture.

Mindset Medical, LLC IVC-400-006


Listing 16.2.6.1

IVC App Pulse Rate and ECG Reference Device Heart Rate

ITC Population

| | | Was the | | | | Reason ECG | | | ECG<br>Reference |
|---|---|---|---|---|---|---|---|---|---|
| Subject | | pulse<br>rate take | n Reason Pulse Was ECG | Reason ECG<br>was Not | Was ECG<br>Strip | Reason ECG<br>Strip Was | Reason not able to | Pulse<br>Rate (BPM) | Device<br>Heart |
| ID | Session | by IVC? | was Not Taken performed? | performed | Uploaded? | Not Uploaded | Analyze | by IVC app | Rate (BPM) |
| 302-020 | 2 | Yes | Yes | | Yes | | | 82 | 83 |
| 302-021 | 1 | Yes | Yes | | Yes | | | 74 | 75 |
| | 2 | Yes | Yes | | Yes | | | 78 | 79 |
| 304-001 | 1 | Yes | Yes | | Yes | | | 67 | 68 |
| | 2 | Yes | Yes | | Yes | | | 71 | 70 |
| 304-003 | 1 | Yes | Yes | | Yes | | | 53 | 53 |
| | 2 | Yes | Yes | | Yes | | | 53 | 52 |
| 304-004 | 1 | Yes | Yes | | Yes | | | 96 | 95 |
| | 2 | Yes | Yes | | Yes | | | 96 | 96 |
| 304-005 | 1 | Yes | Yes | | Yes | | | 71 | 70 |
| | 2 | Yes | Yes | | Yes | | | 71 | 70 |
| 304-006 | 1 | Yes | Yes | | Yes | | | 78 | 79 |

ITC = Intent-to-Capture.

Mindset Medical, LLC IVC-400-006


Listing 16.2.6.1

IVC App Pulse Rate and ECG Reference Device Heart Rate

ITC Population

| Subject<br>ID | Session | Was the pulse rate taker by IVC? | n Reason Pulse Was ECG<br>was Not Taken performed? | Reason ECG<br>was Not<br>performed | Was ECG<br>Strip<br>Uploaded? | Reason ECG<br>Strip Was<br>Not Uploaded | Reason not<br>able to<br>Analyze | Pulse<br>Rate (BPM)<br>by IVC app | ECG Reference Device Heart Rate (BPM) |
|---|---|---|---|---|---|---|---|---|---|
| 304-006 | 2 | Yes | Yes | | Yes | - | - | 78 | 78 |
| 304-007 | 1 | Yes | Yes | | Yes | | | 68 | 69 |
| | 2 | Yes | Yes | | Yes | | | 74 | 73 |
| 304-008 | 1 | Yes | Yes | | Yes | | | 74 | 73 |
| | 2 | Yes | Yes | | Yes | | | 75 | 75 |
| 304-009 | 1 | Yes | Yes | | Yes | | | 78 | 79 |
| | 2 | Yes | Yes | | Yes | | | 78 | 77 |
| 304-010 | 1 | Yes | Yes | | Yes | | | 67 | 67 |
| | 2 | Yes | Yes | | Yes | | | 67 | 67 |
| 304-011 | 1 | Yes | Yes | | Yes | | | 75 | 74 |
| | 2 | Yes | Yes | | Yes | | | 74 | 74 |
| 304-012 | 1 | Yes | Yes | | Yes | | | 71 | 70 |
| | 2 | Yes | Yes | | Yes | | | 68 | 69 |
| 304-013 | 1 | Yes | Yes | | Yes | | | 71 | 70 |

ITC = Intent-to-Capture.

Mindset Medical, LLC IVC-400-006


Listing 16.2.6.1

IVC App Pulse Rate and ECG Reference Device Heart Rate

ITC Population

| Subject<br>ID | Session | Was the pulse rate taken by IVC? | Reason Pulse Was ECG<br>was Not Taken performed? | Reason ECG<br>was Not<br>performed | Was ECG<br>Strip<br>Uploaded? | Reason ECG<br>Strip Was<br>Not Uploaded | Reason not<br>able to<br>Analyze | Pulse<br>Rate (BPM)<br>by IVC app | | е |
|---|---|---|---|---|---|---|---|---|---|---|
| 304-013 | 2 | Yes | Yes | | Yes | | | 73 | 72 | |
| 305-001 | 1 | No | app unable to Yes measure | | Yes | | Null IVC solution | | | |
| | 2 | No | app unable to No measure | | Yes | | | | | |
| 305-002 | 1 | No | app not able Yes<br>to measure | | Yes | | Null IVC solution | | | |
| | 2 | No | The second PRONo assessment was not completed per protocol per PM instruction. | | Yes | | | | | |
| 305-003 | 1 | No | App not able No to measure vitals. | | Yes | | | | | |
| | 2 | No | App not able No to measure vitals. | | Yes | | | | | |

ITC = Intent-to-Capture.

Mindset Medical, LLC IVC-400-006 

Listing 16.2.6.1

IVC App Pulse Rate and ECG Reference Device Heart Rate

ITC Population

| Subject<br>ID | Session | Was the pulse rate take by IVC? | n Reason Pulse Was ECG<br>was Not Taken perform | | Was ECG<br>Strip<br>Uploaded? | Reason ECG<br>Strip Was<br>Not Uploaded | Reason not<br>able to<br>Analyze | Pulse<br>Rate (BPM)<br>by IVC app | ECG<br>Reference<br>Device<br>Heart<br>Rate (BPM) |
|---|---|---|---|---|---|---|---|---|---|
| 305-004 | 1 | Yes | Yes | - | Yes | <del></del> | <del>-</del> | 64 | 65 |
| | 2 | Yes | Yes | | Yes | | | 64 | 64 |
| 305-005 | 1 | Yes | Yes | | Yes | | | 50 | 49 |
| | 2 | Yes | Yes | | Yes | | | 50 | 49 |
| 305-006 | 1 | No | App unable to Yes measure | | Yes | | Null IVC solution | | |
| | 2 | No | App unable to Yes measure | | Yes | | Null IVC solution | | |
| 305-007 | 1 | No | App unable to Yes measure | | Yes | | Null IVC solution | | |
| | 2 | No | App unable to Yes measure | | Yes | | Null IVC solution | | |
| 305-008 | 1 | No | App unable to Yes measure | | Yes | | Null IVC solution | | |
| | 2 | No | App unable to Yes measure | | Yes | | Null IVC solution | | |
| 305-009 | 1 | Yes | Yes | | Yes | | | 71 | 71 |
| | 2 | Yes | Yes | | Yes | | | 73 | 73 |
| 305-010 | 1 | Yes | Yes | | Yes | | | 53 | 53 |
| | 2 | Yes | Yes | | Yes | | | 52 | 53 |
| 305-012 | 1 | Yes | Yes | | Yes | | | 68 | 68 |
| | 2 | Yes | Yes | | Yes | | | 73 | 72 |
| 306-001 | 1 | No | App not able Yes<br>to measure<br>vitals | | Yes | | Null IVC<br>solution | | |
| | 2 | No | App not able No<br>to measure<br>vitals | | Yes | | | | |
| 306-002 | 1 | No | App not able No<br>to measure<br>vitals | | Yes | | | | |

ITC = Intent-to-Capture.

Mindset Medical, LLC IVC-400-006 

Listing 16.2.6.1

IVC App Pulse Rate and ECG Reference Device Heart Rate

ITC Population

| Subject ID | Session | Was the pulse rate taken by IVC? | Reason Pulse<br>was Not Taken | | Reason ECG<br>was Not<br>performed | Was ECG<br>Strip<br>Uploaded? | Reason ECG<br>Strip Was<br>Not Uploaded | Reason not<br>able to<br>Analyze | Pulse<br>Rate (BPM)<br>by IVC app | ECG<br>Reference<br>Device<br>Heart<br>Rate (BPM) |
|---|---|---|---|---|---|---|---|---|---|---|
| 306-002 | 2 | No | App not able to measure vitals | No | | Yes | | | | |
| 306-003 | 1 | Yes | | No | | Yes | | | 95 | |
| | 2 | Yes | | Yes | | Yes | | | 93 | 94 |
| 306-004 | 1 | No | <pre>app not able to measure vitals</pre> | Yes | | Yes | | Null IVC<br>solution | | |
| | 2 | Yes | | No | | Yes | | | 60 | |
| 306-005 | 1 | Yes | | Yes | | Yes | | | 63 | 62 |
| | 2 | Yes | | Yes | | Yes | | | 60 | 61 |
| 306-006 | 1 | Yes | | Yes | | Yes | | | 87 | 88 |
| | 2 | Yes | | Yes | | Yes | | | 87 | 87 |
| 306-007 | 1 | Yes | | Yes | | Yes | | | 77 | 77 |
| | 2 | Yes | | Yes | | Yes | | | 75 | 75 |
| 307-001 | 1 | Yes | | Yes | | Yes | | | 73 | 73 |
| | 2 | Yes | | Yes | | Yes | | | 75 | 74 |
| 307-002 | 1 | Yes | | Yes | | Yes | | | 84 | 83 |

ITC = Intent-to-Capture.

Mindset Medical, LLC IVC-400-006 

Listing 16.2.6.1

IVC App Pulse Rate and ECG Reference Device Heart Rate

ITC Population

| Subject<br>ID | Session | Was the pulse rate taken by IVC? | Reason Pulso | e Was ECG<br>en performed? | Reason ECG<br>was Not<br>performed | Was ECG<br>Strip<br>Uploaded? | Reason ECG<br>Strip Was<br>Not Uploaded | Reason not<br>able to<br>Analyze | Pulse<br>Rate (BPM)<br>by IVC app | ECG<br>Reference<br>Device<br>Heart<br>Rate (BPM) |
|---|---|---|---|---|---|---|---|---|---|---|
| 307-002 | 2 | Yes | | Yes | | Yes | | | 82 | 83 |
| 307-003 | 1 | Yes | | Yes | | Yes | | | 62 | 63 |
| | 2 | Yes | | Yes | | Yes | | | 62 | 62 |
| 307-004 | 1 | Yes | | Yes | | Yes | | | 64 | 65 |
| | 2 | Yes | | Yes | | Yes | | | 61 | 61 |
| 307-005 | 1 | Yes | | No | | Yes | | | 92 | |
| | 2 | Yes | | No | | Yes | | | 92 | |
| 307-006 | 1 | Yes | | Yes | | Yes | | | 77 | 76 |
| | 2 | Yes | | Yes | | Yes | | | 80 | 80 |
| 307-008 | 1 | No | app unable | to Yes | | Yes | | Null IVC | | |
| | | | measure | | | | | solution | | |
| | 2 | Yes | | Yes | | Yes | | | 79 | 79 |
| 307-009 | 1 | No | unable to | Yes | | Yes | | Null IVC | | |
| | | | measure<br>vitals | | | | | solution | | |

ITC = Intent-to-Capture.

Mindset Medical, LLC IVC-400-006 

Listing 16.2.6.1

IVC App Pulse Rate and ECG Reference Device Heart Rate

ITC Population

| Subject ID | Session | Was the pulse rate taker by IVC? | n Reason Pulse Was ECG<br>was Not Taken performed? | Reason ECG<br>was Not<br>performed | Was ECG<br>Strip<br>Uploaded? | Reason ECG<br>Strip Was<br>Not Uploaded | Reason not<br>able to<br>Analyze | Pulse<br>Rate (BPM)<br>by IVC app | |
|---|---|---|---|---|---|---|---|---|---|
| 307-009 | 2 | Yes | Yes | | Yes | | | 75 | 74 |
| 307-010 | 1 | No | no Pulse Rate No<br>obtained- App<br>not able to<br>measure<br>vitals | | No | Thumb drive not recognized by pixel phone. USB was sent back to sponsor for review on 7/20/23 | | | |
| | 2 | No | no Pulse Rate No<br>obtained- App<br>not able to<br>measure<br>vitals | | No | Thumb drive not recognized by pixel phone. USB was sent back to sponsor for review on 7/20/23 | , | | |
| 307-011 | 1 | Yes | Yes | | Yes | | | 60 | 59 |
| | 2 | Yes | Yes | | Yes | | | 57 | 58 |

ITC = Intent-to-Capture.

Mindset Medical, LLC IVC-400-006 Page 1 of 1

Listing 16.2.7.1 Adverse Events ITC Population

Relatio Any nship Unanticipated Caused MedDRA System Organ Class/ Adverse Study Subject Preferred Term/ SAE Study Device Discontinu Investigator AE Term Start Date End Date Ongoing? SAE? Criteria Severity Process Effect Outcome ation

No Data To Report

ITC = Intent-to-Capture. SAE = Serious Adverse Events.